

#### 1. RCT Details

This section provides a high-level overview of the RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes (DECLARE-TIMI 58)

### 1.2 Intended aim(s)

The primary objective will be evaluated in 2 steps. The first step will determine if dapagliflozin is noninferior to placebo for the incidence of MACE assessed with a noninferiority margin of 1.3. If noninferiority is statistically confirmed, the second step will be to determine if dapagliflozin reduces the incidence of the co-primary efficacy end points.

## 1.3 Primary endpoints for replication and RCT finding

- Major Adverse Cardiovascular Events, Including CV Death, Nonfatal Myocardial Infarction (MI), and Nonfatal Stroke
- · Cardiovascular death (CVD) or hospitalization for heart failure (HHF)

### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

A total of 1,390 subjects with MACE events will be required to have 85% power to demonstrate superiority of dapagliflozin to placebo if the true HR is 0.85. The trial was not formally powered for the second of the co-primary end points, CVD or HHF. However, we anticipate 87% power to detect an HR of 0.80 with a 1-sided  $\alpha$  of .0231.

## 1.5 Trial estimate

- MACE- HR, 0.93 (0.84 to 1.03) comparing dapagliflozin to placebo (Wiviott et al.)
- Cardiovascular death or hospitalization for heart failure- HR, 0.83 (0.73 to 0.95) comparing dapagliflozin to placebo

### 2. Person responsible for implementation of replication in Aetion

Ajinkya Pawar, Ph.D. implemented the study design in the Aetion Evidence Platform. S/he is not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform.

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

# 3. Data Source(s)

United/Optum, MarketScan, Medicare

# 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

Disenrollment

## Design Diagram - DECLARE TRIAL REPLICATION

Cohort Entry Date (Day 0)
[Dispensation of Dapagliflozin OR
Individual Non-Gliflozin Antidiabetic Class]



#### 5. Cohort Identification

## 5.1 Cohort Summary

This study will involve a new user, parallel group, cohort study design comparing dapagliflozin to the DPP-4 inhibitor (DPP4i) antidiabetic class. DPP4is serve as a proxy for placebo, since this class of antidiabetic drugs is not known to have an impact on the outcome of interest. The comparison against DPP4 inhibitors is the primary comparison. The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of canagliflozin or a comparator drug (cohort entry date). Follow-up for the outcomes (a. 3P-MACE and b. composite of heart failure hospitalization/all-cause mortality), begins the day after drug initiation. As in the trial, patients are allowed to take other antidiabetic medications during the study.

## 5.2 Important steps for cohort formation

### 5.2.1 Eligible cohort entry dates

Market availability of dapagliflozin in the U.S. started on January 8, 2014.

- For Marketscan and Medicare: Jan 8, 2014-Dec 31, 2017 (end of data availability).
- For Optum: Jan 8, 2014-Mar 31, 2019 (end of data availability).

# 5.2.2 Specify inclusion/exclusion criteria for cohort entry and define the index date

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

# 5.3 <u>Flowchart of the study cohort assembly</u> For dapagliflozin vs. DPP4i

| | Optum | | Marketscan | | Medicare* | |
|---|---|---|---|---|---|---|
| | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 74,864,884 | | 191,990,035 | | 23,466,175 |

| Patients who used exposure or a reference<br>between January 8, 2014 to Dec 2017 (for<br>Marketscan/Medicare)/March 2019 (for Optum) | -74,319,657 | 545,227 | -191,316,290 | 673,745 | -21,925,514 | 1,540,661 |
|---|---|---|---|---|---|---|
| Patients who have continuous 6 months registration in the database | -76,221 | 469,006 | -55,637 | 618,108 | -415,687 | 1,124,974 |
| Excluded due to prior use of referent | -351,484 | 117,522 | -416,417 | 201,691 | -784,720 | 340,254 |
| Excluded due to prior use of exposure | -15,355 | 102,167 | -58,415 | 143,276 | -19,316 | 320,938 |
| Excluded because patient qualified in >1 exposure category | -39 | 102,128 | -166 | 143,110 | -96 | 320,842 |
| Excluded based on missing Age | -3 | 102,125 | 0 | 143,110 | 0 | 320,842 |
| Excluded based on missing Gender | -9 | 102,116 | 0 | 143,110 | 0 | 320,842 |
| Excluded based on Inclusion 1- Age >= 40 | -2,873 | 99,243 | -6,212 | 136,898 | 0 | 320,842 |
| Excluded based on Inclusion 2- DM Type 2 | -4,077 | 95,166 | -6,581 | 130,317 | -3,494 | 317,348 |
| Excluded based on Inclusion 4- High Risk for CV event defined as having either established CV disease and/or multiple risk factors | -34,224 | 60,942 | -30,651 | 99,666 | -260 | 317,088 |
| Excluded based on Exclusion 1a- Current or recent (within 24 months) treatment with pioglitazone | -2,241 | 58,701 | -2,798 | 96,868 | -11,793 | 305,295 |
| Excluded based on Exclusion 1b- Current or recent (within 12 months) treatment with rosiglitazone | -3 | 58,698 | -6 | 96,862 | -13 | 305,282 |
| Excluded based on Exclusion 1c- Previous treatment with any SGLT2 inhibitor (Empagliflozin, ertugliflozin, or canagliflozin) in prior 6 months | -1,292 | 57,406 | -2,269 | 94,593 | -4,526 | 300,756 |
| Excluded based on Exclusion 1d- Any patient currently receiving chronic (>30 consecutive days) treatment with an oral steroid | -965 | 56,441 | -1,000 | 93,593 | -7,968 | 292,788 |
| Excluded based on Exclusion 2- Acute<br>cardiovascular event (in prior 60 days) | -660 | 55,781 | -1,528 | 92,065 | -9,725 | 283,063 |
| Excluded based on Exclusion 4- DM Type 1 OR<br>Secondary DM | -1,900 | 53,881 | -2,091 | 89,974 | -10,363 | 272,700 |
| Excluded based on Exclusion 5 - History of<br>Malignant Neoplasm (prior 5 years) | -2,587 | 51,294 | -2,869 | 87,105 | -19,117 | 253,583 |
| Excluded based on Exclusion 6- History of Bladder cancer (malignant and situ) anytime prior | -2 | 51,292 | -1 | 87,104 | -21 | 253,562 |

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

| Excluded based on Exclusion 7- Chronic cystitis<br>and/or recurrent urinary tract infections (prior<br>year) | -2,023 | 49,269 | -1,761 | 85,343 | -12,690 | 240,872 |
|---|---|---|---|---|---|---|
| Excluded based on Exclusion 8- CCI (180 days)- >= 10 | -235 | 49,034 | -61 | 85,282 | -665 | 240,207 |
| Excluded based on Exclusion 9-Pregnancy | -1 | 49,033 | -3 | 85,279 | 0 | 240,207 |
| Excluded based on Exclusion 15- Liver disease | -187 | 48,846 | -691 | 84,588 | -2,261 | 237,946 |
| Excluded based on Exclusion 16- CKD stage 3 and above | -1,479 | 47,367 | -809 | 83,779 | -6,680 | 231,266 |
| Excluded based on Exclusion 17- Hematuria | -129 | 47,238 | -173 | 83,606 | -630 | 230,636 |
| Excluded based on Exclusion 18- Non-compliance | -4 | 47,234 | -103 | 83,503 | -642 | 229,994 |
| Final cohort | | 47,234 | | 83,503 | | 229,994 |

<sup>\*</sup> Medicare database includes only patients with at least one diagnosis for diabetes, heart failure, or cerebrovascular disease.

#### 6. Variables

## 6.1 Exposure-related variables:

### Study drug:

The study exposure of interest is initiation of dapagliflozin. Initiation will be defined by no use of dapagliflozin or a comparator in the prior 6 months before treatment initiation (washout period).

## Comparator agents-

- · Initiators of dapagliflozin will be compared to initiators of
  - o DPP4i

We will also run feasibility numbers for these antidiabetic classes separately to identify the most appropriate comparator. Because dapagliflozin and comparators are frequently used as second or third line treatments of T2DM, we expect it to be unlikely that dapagliflozin and comparators are initiated in patients with substantially different baseline risk for proposed outcomes.

### 6.2 Covariates:

Age

- Sex
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (**Appendix B**). These covariates are based on those used by Patorno et al. (2019).

### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcomes of interest (definitions provided in **Appendix A**):

- <u>Co-primary outcome</u>: 3-point major adverse cardiovascular events (MACE), i.e., non-fatal myocardial infarction, non-fatal stroke, or CV mortality
- Co-primary outcome: Hospitalization for heart failure (HHF)/All-cause mortality
- · Secondary outcomes: Individual components:
  - Hospital admission for MI (for purposes of this individual component, fatal MI is included)
  - Hospital admission for stroke (for purposes of this individual component, fatal stroke is included)
  - o Hospital admission for heart failure
  - All-cause mortality/CV mortality:
    - All-cause inpatient mortality identified using discharge status codes will be used as a proxy for "CV mortality" in commercial databases
    - Information on CV mortality through data linkage with the National Death Index (NDI) will only become
      available at a later date for Medicare and will be used in secondary analyses.

Control outcome of interest (control outcome only serve to assess aspects of study validity but are not further interpreted):

1. Diabetic Ketoacidosis (we expect to see a positive association; Neal et al., 2017)

#### Control outcome definition

| Outcome | Definition | Comments |
|---|---|---|
| Control Outcomes | | |
| Diabetic Ketoacidosis | Inpatient ICD-9 diagnosis: 250.1x | Note- The corresponding ICD-10 codes will also be used |

### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of dapagliflozin and comparator and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (dapagliflozin and comparator) plus a defined grace period (i.e., 30 days after the end of the last prescription's days' supply in main analyses).
- The date of augmentation or switching from an exposure to a comparator or any other agent in the comparator class and vice versa (e.g. switching from saxagliptin to linagliptin would be a censoring event);
  - A dosage change on the index treatment does not fulfill this criterion
  - An added treatment that is not part of the exposure or comparator group does not fulfill this criterion (e.g. if a dapagliflozin user adds insulin, he or she does not get censored at the time of insulin augmentation)

Effectiveness research with Real World Data to support FDA's regulatory decision making

For the ITT analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

# 7. Initial Feasibility Analysis

#### Aetion report name:

For Dapagliflozin vs. DPP4i

Optum- https://bwh-dope.aetion.com/projects/details/664/results/42809/result/0

Marketscan- https://bwh-dope.aetion.com/projects/details/665/results/42810/result/0

Medicare- https://bwh-dope.aetion.com/projects/details/666/results/42811/result/0

## Date conducted: 10/15/2019

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

- Report patient characteristics by treatment group
- Report summary parameters of the overall study population
- · Report median follow-up time by treatment group
- Report reasons for censoring in the overall study population

#### 8. Initial Power Assessment

### Aetion report name:

For Dapagliflozin vs. DPP4i

Optum- https://bwh-dope.aetion.com/projects/details/664/results/42812/result/0

Marketscan- https://bwh-dope.aetion.com/projects/details/665/results/42813/result/0

Medicare- https://bwh-dope.aetion.com/projects/details/666/results/42814/result/0

Date conducted: 10/15/2019

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 11/4/2019 |
|-------------------------|------------------|----------------|-----------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 11/6/2019 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

### 9. Balance Assessment after PS matching

### Aetion report name:

Optum- https://bwh-dope.aetion.com/projects/details/664/results/45428/result/0

Marketscan- https://bwh-dope.aetion.com/projects/details/665/results/45429/result/0

Medicare- https://bwh-dope.aetion.com/projects/details/666/results/45430/result/0

Date conducted: 11/30/2019

After review of initial feasibility and power analyses, complete creation of the remaining covariates (see Table 1 below for list of covariates). Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates (excluding laboratory values, which are missing in some patients).

· Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

Report covariate balance after matching.

Note- For Table 1, please refer to Appendix B.

· Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy Outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| Death | 116 (0.23%) | 67 (0.27%) | 49 (0.20%) |
| Start of an additional exposure | 1,724 (3.46%) | 411 (1.65%) | 1,313 (5.27%) |
| End of index exposure | 29,607 (59.46%) | 14,752 (59.26%) | 14,855 (59.67%) |
| Specified date reached | 11,094 (22.28%) | 5,670 (22.78%) | 5,424 (21.79%) |
| End of patient enrollment | 6,215 (12.48%) | 3,125 (12.55%) | 3,090 (12.41%) |
| Switch to other DPP4i (for censoring) + nursing home admission | 1,034 (2.08%) | 870 (3.49%) | 164 (0.66%) |

· Report follow-up time by treatment group.

| | Median Follow-Up Time (Days) [IQR] | | |
|---|---|---|---|
| Patient Group | Optum | Marketscan | Medicare |
| Overall Patient Population | 119 [58-267] | 139 [61-310] | 118 [58-250] |
| Referent | 119 [58-286] | 120 [67-261] | 120 [67-261] |
| Exposure | 120 [58-251] | 118 [58-240] | 118 [58-240] |

· Report overall risk of the primary outcome.

| | Optum | Marketscan | Medicare |
|---|---|---|---|
| Risk per 1,000 patients (MACE) | 14.24 | 8.74 | 21.83 |
| Risk per 1,000 patients (composite of Heart failure hospitalization-any diagnosis position)/All-cause mortality | 22.46 | 13.19 | 37.16 |

### 10. Final Power Assessment

Date conducted: 12/1/2019

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9.

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

All other parameters in the table should be the same as in Section 8. If the study is to be implemented in more than one database, copy and paste excel sheet to report power for each database separately and for the pooled analysis that uses data from all databases together. Power calculations are based on the formulas from Chow et al. (2008).

o Pooled

For dapagliflozin vs. DPP4i (Primary outcome- MACE)

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 24,895 | Reference | 24,895 |
| Exposed | 24,895 | Exposed | 24,895 |
| Risk per 1,000 patients | 14.94 | Risk per 1,000 patients | 14.94 |
| Desired HR from RCT | 0.85 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 743.8626 | Number of events expected | 743.8626 |
| Power | 0.601152916 | Power | 0.947155457 |

<sup>•</sup> For dapagliflozin vs. DPP4i (Co-primary outcome- Heart failure (any position)/all-cause mortality)

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 24,895 | Reference | 24,895 |
| Exposed | 24,895 | Exposed | 24,895 |
| Risk per 1,000 patients | 24.27 | Risk per 1,000 patients | 24.27 |
| Desired HR from RCT | 0.8 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 1208.4033 | Number of events expected | 1208.4033 |
| Power | 0.972476483 | Power | 0.995341553 |

# o Optum

For dapagliflozin vs. DPP4i (Primary outcome- MACE)

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 3,316 | Reference | 3,316 |
| Exposed | 3,316 | Exposed | 3,316 |
| Risk per 1,000 patients | 14.24 | Risk per 1,000 patients | 14.24 |
| Desired HR from RCT | 0.85 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 94.43968 | Number of events expected | 94.43968 |
| Power | 0.12392638 | Power | 0.246629377 |

For dapagliflozin vs. DPP4i (Co-primary outcome- Heart failure (any position)/all-cause mortality)

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 3,316 | Reference | 3,316 |
| Exposed | 3,316 | Exposed | 3,316 |
| Risk per 1,000 patients | 22.46 | Risk per 1,000 patients | 22.46 |
| Desired HR from RCT | 0.8 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 148.95472 | Number of events expected | 148.95472 |
| Power | 0.275279358 | Power | 0.359825479 |

# o Marketscan

For dapagliflozin vs. DPP4i (Primary outcome- MACE)

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 12,415 | Reference | 12,415 |
| Exposed | 12,415 | Exposed | 12,415 |
| Risk per 1,000 patients | 8.74 | Risk per 1,000 patients | 8.74 |
| Desired HR from RCT | 0.85 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| North and a second and | 247.0442 | North and account account of | 247.0442 |
| Number of events expected | 217.0142 | Number of events expected | 217.0142 |
| Power | 0.223558993 | Power | 0.489043518 |

• For dapagliflozin vs. DPP4i (Co-primary outcome- Heart failure (any position)/all-cause mortality)

| | | The printer outcome | |
|---|---|---|---|
| Superiority Analysis | | Non-inferiority Analysis | |
| Number of patients matched | | Number of patients matched | |
| Reference | 12,415 | Reference | 12,415 |
| Exposed | 12,415 | Exposed | 12,415 |
| Risk per 1,000 patients | 13.19 | Risk per 1,000 patients | 13.19 |
| Desired HR from RCT | 0.8 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 327.5077 | Number of events expected | 327.5077 |
| Power | 0.52362617 | Power | 0.660585599 |

# o Medicare

• For dapagliflozin vs. DPP4i (Primary outcome- MACE)

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 9,164 | Reference | 9,164 |
| Exposed | 9,164 | Exposed | 9,164 |
| Risk per 1,000 patients | 21.83 | Risk per 1,000 patients | 21.83 |
| Desired HR from RCT | 0.85 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 400.10024 | Number of events expected | 400.10024 |
| Power | 0.369142646 | Power | 0.746657207 |

For dapagliflozin vs. DPP4i (Co-primary outcome- Heart failure (any position)/all-cause mortality)

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 9,164 | Reference | 9,164 |
| Exposed | 9,164 | Exposed | 9,164 |
| Risk per 1,000 patients | 37.16 | Risk per 1,000 patients | 37.16 |
| Desired HR from RCT | 0.8 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 681.06848 | Number of events expected | 681.06848 |
| Power | 0.829390401 | Power | 0.928339341 |

Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of
advisory board. Reviewers evaluate the results of the analyses described above in Sections 9 and 10, including numbers of
patients, balance in patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates
of outcomes and study power.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 12/5/2019 |
|-------------------------|------------------|----------------|------------|
| Reviewed by FDA: | David Martin | Date reviewed: | 12/20/2019 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

# 11. Study Confidence and Concerns

Deadline for voting on study confidence and listing concerns: 12/20/19

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- · All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the

success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the individual respondent.

### 12. Register study protocol on clinicalTrials.gov

### Date conducted:

· Register the study on clinicalTrials.gov and upload this document.

### 13. Comparative Analyses

### Aetion report name:

Date conducted:

# 13.1 For primary analysis:

 In the PS-matched cohort from Section 9, calculate the HR for each outcome for dapagliflozin versus referent patients using a Cox proportional hazards model.

### 13.2 For secondary analyses:

 In the pre-matched cohort, perform asymmetrical trimming to remove patients with PS values below the 2.5<sup>th</sup> percentile of treated patients and above the 97.5<sup>th</sup> percentile of untreated patients. In the trimmed cohort, calculate the HR for dapagliflozin versus referent patients using a Cox proportional hazards model, adjusting for deciles of the PS.

# 14. Requested Results

## 14.1 Results from primary and secondary analyses:

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

Separately for each endpoint:

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Primary analysis | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

### 15. References

American Diabetes Association. 8. Pharmacologic Approaches to Glycemic Treatment: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018;41(Suppl 1):S73-S85. doi:10.2337/dc18-S008.

Chow S, Shao J, Wang H. 2008. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177

Patorno E, Pawar A, Franklin JM, et al. Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study. Circulation. 2019;139: :2822-30.

Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, et al. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. The New England Journal of Medicine. 2019;380(4):347-57.

| # | DECLARE-TIMI 58 trial definitions | Implementation in routine care | References/Rationale | Color coding |
|---|---|---|---|---|
| $\vdash$ | Titlel details- Extimated Study Completion Date : July 18, 2018. | Actual Enrollment : 17,276 participants | Please see the following Google Drive for further details or any mixing in formation:<br>https://drive.aco.ele.com/span/Hdr4 WD41 benear/HB/D41 Tout/-VCcsb/D-d4/ | Criteria |
| | EXPOSURE vs. COMPARI | SCN | EC-50 codes are not little d in this document because of exact call side finitations and exace whe<br>number of EC-50 codes. Full EC-50 code little will be evaluate in the above Google Order Golder<br>(bits above). For it is EC-50 code coverances were completed using a SSA mace that<br>largetiments forward? bechard mapping based on the CMS EC-50 to EC-50 mapping.<br>Date of the exact side is a second or a second or a second or a second or a second or a<br>parameter of the exact side of the coverage of the exact of th | Adequate mapping in claims |
| Г | dapagifforin 10 mg/day vs. placebo | New use of depayificate vs. Individual non-gliffooth antidiabetic class (i.e., a DFP-61, a GCP-51M, and a sulfonylums) | | Intermediate mapping in claims |
| | Safety and co-primary of | facy | | Poor mapping or cannot be measured<br>in claims |
| | 8P-MACS:— CY dwells, noo-fatal Mi, noo-fatal inchensis stroke | Measured 1 days after drug initiation in dilagnosis position specified below and impatient care setting: impatient neutrality[Mit/Doubs — For Mit Any disposition in impatient care setting ECO+ diagnosis of ECX (paste represented inferrotion) excluding 610.22 (subsequent episode of care) For stroke Primary diagnosis position in impatient care setting ECO+ discharge diagnosis; EC | For Mil: #PPYFM his Medicare claims data (Clysta Y, Schamewrik S, Glynn RJ, Cannuacio CC, Avom J, Solomo DL. Accuracy of Medicare claims claim of diagnosis of acute reporantial inforction: estimating positive predictive rules on the hades of review of hospital records. American heart journal 2005;16:199-1091. #PPYFER 5th commercially-bound diagnostic and procedure rooted for cardiovecoder and generalistic Polymer of Commercial Privated population. Pharmacoopidemiology and Drug Schley. 2005;18:198-600. #PPY Length go non-section - commercially-bound-population. Pharmacoopidemiology and Drug Schley. 2005;18:598-600. #PPY Length go no SCh to 18th Sch Homoritagis struke #PPV Length go not obtained to returnish to Michael catalous loss and polymers of the PPY Length of the Schole of the Totalous Commercial Privated PPV Length of the Schole of the Totalous Homoritagis struke #PPV Length of the Schole of Totalous Homoritagis struke #PPV Length of Length of the Schole of Totalous Homoritagis struke #Plendude SJ, Harnold LH, 1913, et al. A systematic network of validated methods for identifying overlow-socked another or transverte Homoritagis and policy and policy and commercial recording to 1005;18:136-156-7-101. #Plendude SJ, Harnold LH, 1914, et al. A systematic network of the Schole of the Sch | Can't be removed in claims but not important for the analysis |
| | Co-primary efficacy | | | |
| | - CV death, hospitalization due to heart failure | Measured 1 days after drug initiation in any diagnosis position and inpetient care as titing:<br>Mear failure requiring beapsilusation: CD-0 diagnosis<br>4732, 365.81, 400.21, 400.21, 400.21, 400.41, 400.11, 400.41, 404.02, 404.12, 404.93<br>CV de atth-Dependent on data source, see mortality sheet | | |
| $\vdash$ | INCLUSION CRITERIA | | | |
| 1 | Provision of informed consent prior to any study specific procedures (including run-in) | N/A | | 1 |
| 2 | 2. Female or male aged a 40 years | Age >10 years at drug initiation Measured 1.00 days prior to and including day of drug initiation in any diagnosis position and the impatient or | | |
| 1 | 3. Diagnosed with T2DM | outpatient care setting | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagifficativeness other non- | 1 |
| 1 | Diagnosis of T2DM can be based on the following: | Total 2 Diabetes ICD-9 diagnosis: 250.x0, 250.x2 | gil floats antidiabetic drugs: population based cohort study." 8MJ 2018;160:k119<br>http://dx.doi.org/10.1186/bmj.k129 | |
| , | - Pior documentation of tree 2 disheter. AMOVOR - Treatment with anti-honomiscensis medications and/or det AMOVOR - ADA criteria; planta a radion skurzae > 200 mariel 11.1.1 monol(1) or facility > 126 majol (7.0 monol(1) or 2-b planta glacose > 200 mg/dl (7.0 monol(1) during an oral glacose tolerance test or IPAAC & 65%). | | Patomo, Bisabetta et al. "Singagifficain and the Höd of Heart Fallure Hospitalization in Routine<br>Clinical Case A Rist Analysis from the Empagifficain Comparative Effectiveness and Safety<br>(SMPHSS) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAMA.118.039177 | |
| 4 | 4. High likk for CV event defined as having either established CV disease and/or multiple risk factors: | Measured anytime prior to and including day of drag hit ation in any procedure position and inputient care setting Stable angion, 41 i.k.s. Unstable angion, 45 i.k.s. Unstable angion, 45 i.k.s. | | |
| | - Established CV Disease (See below for details) | | | l |
| | 4.1 Established Vascular Disease inchemic heart disease (any of the following): | • | | l |
| | - Documented Myscardial infaction | Measured anytime prior to and including day of drug hid at on in any diagnosis position and the inpatient or<br>outputient care acting<br><u>house MI</u> CCP+ diagnosis: 430 cm, (2st 6d) CCP+ diagnosis: 432 cm | Patorno, Blashetta et al. "Cardiovascular outcomes associated with canagifficatio versus other non-<br>gif Sods as intilizients drugs: population based cohort study." IRIJ 2013;160:0119<br>https://dx.doi.org/10.1116/bmj.3139 Patorno, Blashetta et al. "Imagelficatio and the Rid of Heart Fallure Hospitalization in Noutine<br>Clinical Care. A First Analysis from the Empaglificatio Comparative Effectioness and Safety<br>(BAPRES) Study." Chrosiston. 2013 April. doi:10.1156/CHCLL.NICHARALTI.030177 | |
| | Percutaneous Coronary Intervention | Measured anytime prior to and including day of drag biddedon in any procedure position and impatient care wetting—CPT-1:32973, 92982, 92964, 92965, 92969, 92920—92923, 92924—92925, 92987, 92983, 92981, 92983, 92984, 92982—92925, 92987, 92983, 92981, 92983, 92984, 92982—92925, 9 | Patoros, Sisabetta et al. "Cardiovascular outcomes associated with canagilificativ ownse other non-<br>giff four an estilabettic drugs population based cohort study." BMJ 2018;160:8519<br>Patoros, Silabetta et al. "Empagification and the Risk of Heart Fallure Hospitalization in Noutine<br>Clinical Care, A Pirat Analysis from the Empagificatic Comparative Silectionous and Safety<br>(SARPESS) Study." Circularison, 2019 Apr 8, doi:10.1161/CIRCULATIONAMA.118.039377 | |

| - Coronary Artery Bypass Graffing | CASC Measured surptions prior to and including day of drug initiation in any procedure position and inpetient care setting-CPT-4: 85500 – 88566, 88545, 88572 OR Measured surptions prior to and including day of drug initiation in any procedure position and inpetient or outpathent care withing - KCO-0 procedure, id. 12, 86.2x | |
|---|---|---|
| - Objective Findings of Coronary Stenools (> 50%) in at least 2 coronary arteries | Measured anytime prior to and including day of drug habitation in any diagnost position and inputient or<br>outputient care withing. Consert afficient fends and other forms of characteristic beautifuses. VCD-9 diagnosis 454.as. | Patorno, Shaketta et al. "Cardiovenular outcomes associated with caseglifusion versus other nor<br>gli Saria antibilisetti drugo population based orbitor duals," SMJ 2013;3603419<br>https://do.doi.org/10.1146/epu/1319<br>Patorno, Shaketta et al. "Singaglifusio and the Risk of Heart Fallure Hospitalization in Soutine<br>Clinical Case A First Analysis have the Engaglifusion Comparation Effect twees and Safety<br>SMP Hill Disable; "Considerio, 2013 day 6. doi:10.1145/SMP.CH.J.DRSMPAS.EL.2013737 |
| Combinuscular disease (any of the following): Documented lichemic Stroke | Measured surptime prior to and including day of drug initiation in any diagnoss position and inputient or<br>subpation care writing. Submits divide he and with mention of our dead industriand, VCD-0 diagnosis: 43 ft. xx, 43 ft. xx, 44 ft. xx | Patorno, Shalletta et al. "Cardiovenolar outcomes associated with cangificatio versus other nor<br>giffod a antidiabetic drugs population hased orbort study." BMJ 2019;16:03:119<br>https://do.doi.org/10.1146/bmj.1219<br>Patorno, Shalletta et al. "Singuigificatio and the Rhd of Heart Fallure Hospitalization in Soutine<br>Clinical Case A Rivet Analysis from the Singuigification Comparative Sinctheres and Safety<br>BMPHSI(Shallet). "Conclusion. 2019 art. doi:10.1145/SCICELARIOMANIATE.09917" |
| Known translated ischemic attack, primary intracerebral hernormage or subarachnoid hernormage do not qualify. - Carolid stenting or endarterectomy | NA. Measured supplies prior to and including day of drug initiation in any procedure position and in patient or<br>subjection care withing—<br>South describe or endorterations.<br>EXP procedure 28.23, 00.65, 00.68<br>CP14.165.001 | ICD-9 procedure code 90.62 is regarding intracranial vessel and was not included. |
| Peripheral Arterial Disease Jany of the followings: | | |
| - peripheral arierial stenting or surgical revascularization | Measured anytime prior to and including day of drug hibitation in any procedure position and the inpatient or<br>outparties care withing<br>the hibber of arterial destrictor outploal reasonal action. ICD-9 procedure; 29.25, 29.50, 29.99 | Pationia, Blushetta et al. "Cardiovascular outcomes associated with casagiffusin versus other nor<br>giff Suria antifoliatric drugs population based cohort exalp." BMJ 2013;160:X119<br>https://dx.dai.org/10.1146/bmj.1219<br>Pationia, Blushetta et al. "Empagiffusin and the Role of Heart Fallure Hospitalization in Routine<br>Clinical Case A Rivat Analysis burn the Empagiffusin Comparative Effectiveness and Safety<br>BMPHES(State)." Coloration. 2018 987. doi:10.1145/SCPCECEA/EMPMHA18.09917 |
| - lower extremity amputation as a result of pelipheral arterial obstructive disease | Measured anytime prior to and including day of drug liabilation in any diagnosis/procedure position and the impacts of or output out one setting places and remains and setting and anything and anything and anything and anything and anything and anything anything and anything anything and anything an | Paterno, Shahetta et al. "Cardiovecular outcome associated with caseglifusin versus other nor<br>giffusin antidiabetic drugs population based onbort study." IRIA 2018;160:1619<br>https://dw.doi.org/10.1146/bm/s1219<br>Paterno, Shahetta et al. "Empaglifusin and the Rida of Heart Falture Hospitalization in Noutine<br>Clinical Case A Rivet Analysis born the Empaglifusin Comparative Sinctimere and Safety<br>(AMPHSS) Case). "Consistan. 2018 part. doi:10.1145/JCRUSA.00044412.09817." |
| - Current symptoms of Intermittent claudication AND antisyltrachial Index (ABI) < 0.90 documented within last 12 months | Measure danytime prior to and including day of drug initiation in any diagnosis position and the inpatient or<br>subpatient can set the control of the control | |
| OR | • | |
| Sb. No known cardiovacular disease AND at least two cardiovacular risk factors in addition to TXDM, defined as: | • | |
| 6b. No known certiforwarder disease AND at least two certiforwarder disk factors in addition to TXDM, defined as: - App 2 55 years in mass and 2 60 is women. | -Age >55 years in nees and > 60 in women at drog industries | Note: This in the first risk factor. |
| 4b. No known cardiovascular duesse AND at least two cardiovascular risk factors in addition to TXDM, defined as: | -Age 255 years in mee and 260 in women at druginistation Measured supplies prior to and including day of druginistation in any diagnosis position and the inpatient or output including a CD-9 diagnosis 272.0x-272.4x | Patorno, Shabetta et al. "Cardiovescular outcome sescritared with canagifficativ were other nor<br>giff fouts ambilishetic druge population based cohort study." IRIU 2013;160:1519<br>http://dx.doi.org/10.1116/bmj.k119<br>Patorno, Shabetta et al. "Snoggifficatio and the Roi of Heart Failure Hospitalization in Nostine<br>Citizat Cana Roi To Analysis how the Tomorafficatic Consequent to Differentees and Galaxy. |
| B. No boxen cardiovacular disease AND at least two cardiovascular risk factors in addition to TZDM, defined as: — App > 25 years in main and > 60 is woman AND presence of at least 1 of the following additional risk factors (use below for details) | Measure d'amptine prior to and including day of drug initiation in any diagnosis position and the inputient or<br>infrariant care writing<br>Except initiation in CD+ diagnosis: 272.0x-372.4x | Paterns, Shahetta et al. "Cardiovasodar outcomes associated with canagificativ owns other no<br>gli floria antidiabetic drugs propoletica is based colourt multy." PMJ 2013;86:03119<br>http://dx.doi.org/10.1116/j.muj.3119<br>Paterns, Shahetta et al. "Smoothificatio and the Role of Heart Failure Hospitalization in Northe |
| No known cardiovacular disease AND at least two cardiovacular risk factors in addition to T2DM, defined as: Age 2 55 years in man and 2, 60 in women AND presence of at least 1 of the following additional risk factors (see below for details) - Dyslipidemia (at least one of the following) | Measured supplies prior to and including day of drug indication in any diagnosis position and the inputient or output incidents of the inputient or output incidents of the inputient of the input incidents of the input input incidents of the input incid | Patorno, Shabetta et al. "Cardiovenciar outcome associated with canagifficativ weren other nor<br>gifficute ambilishetic druge: population based cohort study." BMJ 2013;860:6139<br>http://dx.doi.org/10.1186/bmj.k119<br>Patorno, Shabetta et al. "Snapagificute and the Rol of Heart Faller Applications in Norther<br>Citical Cana & Fall Analysis from the Tomosofficial Company the Districtures and Galax." |
| B. No brown coefficeworder disease AND at least two coefficeworder disk factors in addition to T20M, defined as: - Age 2 50 years in man and 2, 60 in secones AND passence of at least 1 of the following additional risk factors (see below for details) - Dyslipidemia (at least one of the following) - Low-density lipoprotein cholesterol (LDL-C) > LBO mg/d (3.36 mms/r), within last 12 months - On lipid lowering therapy prescribed by a physician for dyslipidemia - Hypertension (at least one of the following) | Maximum d singilizer prior to and including day of drug inhibition in any diagnosis position and the inpution or subjection care writing. **The diagnosis 272.0x-372.4x** **The diagnosis 272.0x-372.4x** **Maximum diagnosis 272.0x-372.4x** **Maximum diagnosis prior to and including day of drug inhibition as a diagnosis group of one of the following maximum diagnosis into in the highlight group indication in an adaps and group of one of the following maximum diagnosis prior to and including day of drug inhibition in any diagnosis position and the inpution or uniquation care writing threat tension (CD-9 diagnosis 401.x 401.x) | Patorno, Shabetta et al. "Cardiovenciar outcome associated with cangliff oils we un other nor<br>giff foots and dubetic drugs: population based cohort et alsy." 8842 2013;160:6119<br>http://dx.doi.org/10.1186/kmj.k119<br>Patorno, Shabetta et al. "Snapagiffoots and the Not of Heart Failure Hospitalization in Routine<br>Citizad Case. 8 for Analysis from the Consulficial Community of Determinant and Galaxy. |
| No known cardiovacular disease AND at least two cardiovascular risk factors in addition to T20M, defined as: – Age 2 55 years in men and 2, 60 in women AND presence of at least 1 of the following additional risk factors (see below for details) - Dyslipidemia (at least one of the following) - Low-density lipoprotein cholesterol (LDL-C) >130 mg/d (3.36 mmol/L) within last 12 months - On lipid lowering therapy prescribed by a physician for dyslipidemia | Measured angline prior to and including day of drug inhibition in any diagnosis position and the inputient or unquitation care setting. Measured angline prior to and including day of drug inhibition is a dispending of one of the blowing medications into in the <u>Vasionse limit lovering SC</u> , deep . Measured angline prior to and including day of drug inhibition is a dispending of one of the blowing medications into in the <u>Vasionse limit lovering SC</u> , deep . Measured angline prior to and including day of drug inhibition in any diagnosis position and the inputient or unity attention care within SC and SC and Including day of drug inhibition in any diagnosis position and the inputient or unity attention. Also because of the SC angle of the SC and SC angline in the SC angle of the SC ang | Patornio, Disubetto et al. "Carolivoscodar outcomes associated with canagifficitiv sevan other nor giff forte an fidal-hetic drugs population based cohort code," Biol 2013/8606118 https://do.doi.org/10.1116/jmj.2159 |
| B. No brown coefficeworder disease AND at least two coefficeworder disk factors in addition to T20M, defined as: - Age 2 50 years in man and 2, 60 in secones AND passence of at least 1 of the following additional risk factors (see below for details) - Dyslipidemia (at least one of the following) - Low-density lipoprotein cholesterol (LDL-C) > LBO mg/d (3.36 mms/r), within last 12 months - On lipid lowering therapy prescribed by a physician for dyslipidemia - Hypertension (at least one of the following) | Maximum of singiline prior to and including day of drug inhibition in any diagnosis position and the inpution or subjection care writing. **Trace limitarial, K.D-9 diagnosis: 272.0x-372.4x **Measured surptime prior to and including day of drug inhibition as a dispending of one of the following test distribution in the highlighted limitarial prior to and including day of drug inhibition in any diagnosis position and the inpution or unique distribution in any diagnosis position and the inpution or unique tension (CD-9 diagnosis: 401.x - 405.x **Measured surptime prior to and including day of drug inhibition in any diagnosis position and the inpution or unique tension (CD-9 diagnosis: 401.x - 405.x) **Measured surptime prior to and including day of drug inhibition as a dispending of one of the following medications into in the ***Legithpurchasile** disert.** | Paterno, Disubetto et al. "Carolovamodar outcomes associated with cassagificatio sevan other nor gift forts as richishetic drugs; population hased cohort sculp," BMJ 2013;160:bill 9 Dispojich, dulong (20.1114/m)a 12.99 Dispojich dulong (20.1114/m)a 12.99 Dispojich (20.1114/m)a 12.99 Dispoji |
| B. No brown coefficenceder disease AND at least two coefficenceder disk factors in addition to T20M, defined as: - Age 2 50 years in man and 2, 60 in secones AND passence of at least 1 of the following additional risk factors (see below for details) - Dyslipidemia (at least one of the following) - Low-density lipoprotein cholesterol (LDL-C) > LBO mg/d (3.36 mms/r), within last 12 months - On lipid lowering therapy prescribed by a physician for dyslipidemia - Hypertension (at least one of the following) | Maximum d singition prior to and including day of drug inhibition in any diagnosis position and the inpution or subjection care writing. **Trace limitarial, K.D-9 diagnosis: 272.0x-372.4x **Measured singition prior to and including day of drug inhibition as a dispending of one of the following the diagnosis into the highlighted limitarians as a dispending of one of the following the diagnosis into in the highlighted limit into the diagnosis prior to and including day of drug inhibition in any diagnosis profit on and the impatient or uniquation care writing three transions (CD-9 diagnosis: 401.x –401.x) **Measured singition prior to and including day of drug inhibition in any diagnosis position and the impatient or uniquation care writing. **Measured singition prior to and including day of drug inhibition in any diagnosis position and the impatient or uniquation care. **Measured singition prior to and including day of drug inhibition in an adapsending of one of the following day of drug inhibition in an adapsending of one of the following. | Paterno, Disubetto et al. "Carolovamodar outcomes associated with cassagificatio sevan other nor gift forts as richishetic drugs; population hased cohort sculp," BMJ 2013;160:bill 9 Dispojich, dulong (20.1114/m)a 12.99 Dispojich dulong (20.1114/m)a 12.99 Dispojich (20.1114/m)a 12.99 Dispoji |

| ⊢ | EXCLUSION CRITERIA | | |
|---|---|---|---|
| $\vdash$ | Patients should not meet any exclusion criteria at the time of randomization. If at the time of enrollment, it is known that the | N/A | |
| L | patient will not meet criteria after a successful run-in period he/she should not be entered into run in. | | |
| | 1. Use of the following excluded medications: | • | |
| | Current or recent (within 24 months) treatment with ploglitzzone and/or use of ploglitzzone for 2 years or more at any time. | Measured 730 days prior to and including day of drug initiation as a dispensing of plugitazione | |
| | | Measured 100 days prior to and including day of drug initiation as a dispensing of resigitzance | |
| 1b | Current or recent (within 12 months) treatment with rosigilizatione | Measure 2305 days prior to and including day of drug instation as a dispensing of resigificance.<br>Measure 2300 days prior to and including day of drug instation as a dispensing of resigificance empagificatin, | |
| ic | Previous treatment with any SG(T2 inhibitor | arting fines, or count fines | |
| sd | <ul> <li>Any patient currently excelling chronic (&gt;30 consecutive days) treatment with an oral steroid at a dose equivalent to oral<br/>predistrione &gt;10 mg (e.g., betamethasone &gt;1.2 mg, desamethasone &gt;1.5 mg, hydrocordisone &gt;40 mg) per day</li> </ul> | Measured 180 days prior to and including day of drug institution as a dispensing of an onal continuous with<br>days cuply-100 days.<br>Cast continuous days of the continuous predictions, prediction on the continuous days and continuous predictions, prediction on the continuous days and continuous days are days and continuous days and continuous days are days and continuous days and continuous days are days and continuous days and continuous days are days and continuous days and continuous days are days are days and continuous days are days and continuous days are days and continuous days are days and continuous days are days are days and continuous days are days and continuous days are days are days are days are days and continuous days are days | Patomo, Bisaletta et d. "Cardiovascular outcome associated with canagificatio versus other nor<br>gif fluids ambitulents drugs copoulation based outcome study." Biol 2019;16:00119 https://dw.doi.org/10.1116/biol.1159 https://dw.doi.org |
| ⊢ | | Measured 60 days prior to and including day of drug initiation in any diagnosis/procedure position and the care | - Secretario de Secretario del Secretario de Secretario de Considera |
| 2 | 2. Anale cardiovascular event (e.g., ande coronary syndrome (ACS), transient inchemic attack (TIA), stroke, any revascularization, decomposated (if), sustained trachycards of weeks prior to randomization. Patients with acute cardiovascular events can be excelled in the nur-in period as long as randomization does not occur within it weeks of the event. | article budies bud below Mi (hapterine) Chapterine; CCD-0-diagnosis 410.xx Mi (hapterine) Chapterine; CCD-0-diagnosis 410.xx Caretar resounds foreign This chapterine; CCD-0-diagnosis 410.xx Caretar resounds foreign RD 49, 829-84, 929-84 (1994-00; CP-0-4, 929-8), 929-84, 929-85, 929-86, 929-83-929-82-13, 929-84-929-85, 929-83, 929-84, 929-94, 929-94, 929-94, 929-94, 929-94, 929-94, | Patorios, Shaletta et al. "Cardiovascular outcomes associated with canagifficatio versus other non-<br>giff fluid as intilulents of use proposition based robust study." BMJ 2013;160:5119 Patorios, Disabetta et al. "Impedification and the fills of Shart Tailiure Mosphillastics in its Northine<br>Clickat Care. A Taix tudgets from the ingragificatio comparative Sifectimes and Safety<br>(SMP 9555) Study." Circularios. 2018 Apr S. doi: 30.3163/CIRCULATIONAMAL18.0389377 |
| 3 | 3. Systolic BP > LBO or disastolic BP > 300 mmilig at randomization | Measured 180 days prior to and including day of drug instation in any diagnosis position and the inpatient or | |
| ٠ | 4. Diagnosis of Type 1 diabetes mellitus, Maturity onset diabetes of the young (MCOY), or secondary diabetes mellitus | Measured 150 day petro in our including day of drug instantion in any diagnosis position and the Impatient or<br>outpublished can settling<br>(https://tibediagnosis/56xx1, 250x2<br>Secondary diabetes KD-9 procedures 269.xx | Patoms, Disabetta et al. "Varidovenciar outcome associated with casagiffusion wests other non-<br>glift forts and blahetic drugs: population based cohort study." SMJ 2018;160:b119<br>http://dx.doi.org/10.1146/bmj.1319<br>Patomo, Sikaletta et al. "Impagiffusion and the Role of Heart Fallure Hospitalization in Routine<br>Clinical Care A Pinz Analysis town the Impagiffusion Comparathe (Efficiences and Safety<br>SMJ HSS) SMJ 25; Consistano. 2018 pp. doi:10.1145/SCPCLURICHMENT.10.09177 |
| s | S. Hillstony of bladder cancer or history of radiation therapy to the lower abdomen or palels at any time | Measured from that start all available data prior to drug held after in any diagnosis position and the inpatient or<br>outputient care artifug<br>Bladder cancer (maligness) and sho! KD-9 diagnosis: 233.7s | Patorno, Bisaletta et al. "Cardiovascular outcomes associated with canagifficatio versus other non-<br>igificatio antifoliatric drugs population based cohort study." BMJ 2018;160:h119<br>https://dx.dub.org/10.1116/bioys1319 Patorno, Bisaletta et al. "Empagificatio and the Risk of Heart Fallure Hospitalization in Noutine<br>Clinical Cana A Pirst Analysis hour the Empagification Comparathe diffectiveness and Safety<br>BMPRSS (Sust). Circulation. 2018 pt. doi:10.1116/JCPCLRICHOMANLIS.09177 |
| 6 | 6. History of any other malignancy within 5 years (with the exception of successfully treated non-melanoma skin cancers) | Measured 1815 days prior to drug initiation in any diagnode position and the impatient or outpatient care acting Mixtury of muligrant neoplasm KD-9 diagnosis 140.x=205.xx (except 173.xx, non-medianoma skin cancer) | |
| , | 7. Chronic cyttliss and/or recurrent urinary tract infections (3 or more in the last year) | Measure 5:50 days prior to and including the day of drug initiation in any diagnosis position and the inputient or<br>outputient care setting<br>Preferensivities or unknown treat infection (UTE) CC+4 diagnosis: 590.4, 599.0 | |
| | 8. Any conditions that, in the opinion of the insectigator, may render the patient unable to complete the study including but not limited to confidence (NYNA class NY CNF, securent ventricular arrhythmized) or non-cardionscular disease (e.g., active muligrancy with the exception of basel oil carcinoma, cirrhosis, choosic long disease, severe autoinsmuse disease) and/or a libely fatal outcome within 5 years | Measured 180 days prior to and including the day of drug indication - CC1 >= 10 | Sages, Josh J. et. al. "Examinised convorted thy wore predicted mortality in elderly patients better than existing wore." J. Dis Spidenius. 2011. Jul (64/7): 744-58. doi: 10.1016/j.) July 2-200. 10.004. Sau, Jersey W. et. al. "Validation of the Combined Convorted try Index of Charlson and Bibbauser to Predict 3-Cup Martality. According to the Combined Convorted try. 2018 Sep. 54(9): 812. doi: 10.109/July 2000.000000000000000000000000000000000 |
| | 9. Pregnant or breast-feeding patients | Measure £180 days prior to and including day of drug inhibition in any diagnosis position and inpatie at or subjection came withing<br>Englasmix—fee "Pregnancy" for ICD-9 diagnosis and procedure codes. | Enumon, Alexica, et. al. "Etndy protocol for the-dahlgatran, aphaban, riverceaban, edocaban, earfield comparative effectiveness research etndy." J. Comp. 58. Rec. (2018) 7(3), 57–66. doi: 10.2217/joe-3817-0053. |

| 11 | is 15. AST or ALT > lix ULN or Total billioubin > 2.5 x ULN 5. S. CrCl < 60 mil/min (based on the Cockroft-Gaudt equation) | <u>Liber disease</u><br>EC-9 diagnosis (17thus, 57thus-57thus, 456.thu-456.2x, 576.ftx, 782.4x, 789.5x<br>EC-9 procedure codes 88.3x, 42.41 | Patorios, Blashetta et al. "Cardiovascular outcomes associated with canagificatis versus other non-<br>gli floris antifildentic drugs population based cohort study." 860: 2013;860:5119<br>http://dx.doi.org/10.1186/kmjl.3119<br>Patorios, Blashetta et al. "Sinpagificatio and the Rids of Heart Fallure Hospitalizatios in Routine<br>Clinical Cane. A First Analysis Issue the Finpagificatio Comparative Effectiveness and Gelety<br>3869/850] Study." Circulation. 2019 Apr 8. doi:10.1161/CIRCULATIOMMALIS.038127 |
|---|---|---|---|
| 13 | 16. CrCl < 60 mi/min (based on the Cockroft-Gault equation) 17. Hematuria (confirmed by microscopy at Visit 1) with no explanation as judged by the investigator up to randomization. If bladder cancer is identified, patients are not eligible to participate. | outpatient care setting | |

| Trial ID | sNDA21 |
|---|---|
| Trial Name (with web links) | DECLARE-TIMI 58 |
| Trial Name (with pdf links) | |
| NCT_ | NCT01730534 |
| Trial category | Secondary indication |
| Run-in period Description | |
| Run-in period? | |
| Therapeutic Area | Endocrinology |
| Study batch | Diabetes medications |
| RCT Category | 4a- Unintended S with label change |
| Brand Name | Fanxiga |
| Generic Name | Dapagliflozin |
| Sponsor | |
| <u>Year</u> | 2019 |
| | Cardiovascular death (CVD) or hospitalization for heart failure (HHF) |
| | <ul> <li>Major Adverse Cardiovascular Events, Including CV Death, Nonfatal Myocardial Infarction (MI), and Nonfatal Stroke</li> </ul> |
| Measurable endpoint | |
| Exposure | Dapagliflozin |
| <u>Comparator</u> | Placebo |
| <u>Population</u> | Patients with type 2 diabetes who had or were at risk for atherosclerotic cardiovascular disease |
| Trial finding | HR, 0.83 (0.73 to 0.95) for Cardiovascular death or hospitalization for heart failure comparing dapagliflozin to placebo |
| Notes | |
| No. of Patients | 17160 |
| Non-inferiority margin | HR = 1.30 |
| Assav Sens. Outcome | |
| Assay Sens. Endpoint (from trial) | |
| | A total of 1,390 subjects with MACE events will be required to have 85% power to demonstrate superiority of dapagliflozin to placebo if the |
| <u>Power</u> | true HR is 0.85. The trial was not formally powered for the second of the co-primary end points, CVD or HHF. However, we anticipate 87% |
| | power to detect an HR of 0.80 with a 1-sided α of .0231. |
| Blinding | Double-blinded |
| Statistical Method | |
| Approval indication | |

# Mortality-Dependent on data source. 1. All-cause mortality / inpatient mortality Identified using the vital status file-Medicare Identified using the discharge status codes-Optum-20 = EXPIRED • 21 = EXPIRED TO BE DEFINED AT STATE LEVEL 22 = EXPIRED TO BE DEFINED AT STATE LEVEL 23 = EXPIRED TO BE DEFINED AT STATE LEVEL 24 = EXPIRED TO BE DEFINED AT STATE LEVEL 25 = EXPIRED TO BE DEFINED AT STATE LEVEL 26 = EXPIRED TO BE DEFINED AT STATE LEVEL 27 = EXPIRED TO BE DEFINED AT STATE LEVEL • 28 = EXPIRED TO BE DEFINED AT STATE LEVEL • 29 = EXPIRED TO BE DEFINED AT STATE LEVEL 40 = EXPIRED AT HOME (HOSPICE) 41 = EXPIRED IN A MEDICAL FACILITY (HOSPICE) 42 = EXPIRED - PLACE UNKNOWN (HOSPICE) Truven- 20 - Died 22 - Died • 23 - Died • 24 - Died 25 - Died 26 - Died 27 - Died 28 - Died 29 - Died

• 40 - Other died status or Expired at home (Hospice claims only) (depends on year)

- 41 Other died status or Expired in medical facility (Hospice claims only) (depends on year)
- 42 Other died status or Expired place unknown (Hospice claims only) (depends on year)
- 21 Died or Disch./Transf. to court/law enforcement (depends on year)

## 2. CV mortality

Information on CV mortality through data linkage with the National Death Index (NDI) will be available for Medicare at a later date. We will conduct secondary analyses using CV mortality at that time.

| Antidiabetic class | Specific agent | Notes |
|---|---|---|
| | Canagliflozin | Approved 3/29/2013 |
| SGLT2-inhibitors | Dapagliflozin | |
| SGL12-minonors | Empagliflozin | |
| | Ertugliflozin | Approved Dec 21, 2017 |
| | Glimepiride | |
| 2 <sup>nd</sup> generation sulfonylureas | Glipizide | |
| | Glyburide | |
| | Alogliptin | |
| DPP-4 inhibitors | Linagliptin | |
| DPP-4 inhibitors | Saxagliptin | |
| | Sitagliptin | |
| | Exenatide | |
| | Liraglutide | |
| GLP-1 receptor agonist (GLP1-RA) | Albiglutide | Approved April 15, 2014 and discontinued July 26, 2017 |
| | Dulaglutide | Approved Sep 18, 2014 |
| | Lixisenatide | Approved July 28, 2016 |
| | Semaglutide | Approved Dec 5, 2017 |
| | Insulin Aspart | |
| | Insulin Aspart/Insulin Aspart Protamine | |
| | Insulin Degludec | |
| | Insulin Detemir | |
| | Insulin Glargine | |
| | Insulin Glulisine | |
| Insulin | Insulin human isophane (NPH) | |
| | Insulin human regular (search with NPH, | |
| | don't want bf-pk) | |
| | Insulin human regular/ Insulin human isophane (NPH) | |
| | Insulin Lispro | |
| | Insulin Lispro/Insulin Lispro Protamine | |
| Glitzzones | Pioglitazone | |

| Опиадопея | Rosiglitazone |
|------------------------------------------|----------------|
| Meglitinides | Nateglinide |
| | Repaglinide |
| Alpha-glucosidase inhibitors | Acarbose |
| | Miglitol |
| Pramlintide | Pramlintide |
| 1 <sup>st</sup> generation sulfonylureas | Acetohexamide |
| | Chlorpropamide |
| | Tolazamide |
| | Tolbutamide |

| Statins and Other Lipid Lowering Medications |
|--------------------------------------------------------------|
| AMLODIPINE BESYLATE/ATORVASTATIN CALCIUM |
| ARGININE/NIACIN/YOHIMBE BARK/GINSENG/GNK/DAMIANA/SCHISANDRA |
| ATORVASTATIN CALCIUM |
| CERAMIDES 1,3,6-11/NIACINAMIDE |
| CERAMIDES 1,3,6-11/NIACINAMIDE/HYALURONIC ACID |
| CHOLESTYRAMINE |
| CHOLESTYRAMINE (WITH SUGAR) |
| CHOLESTYRAMINE/ASPARTAME |
| COLESEVELAM HCL |
| COLESTIPOL HCL |
| EZETIMIBE |
| EZETIMIBE/ATORVASTATIN CALCIUM |
| EZETIMIBE/SIMVASTATIN |
| FENOFIBRATE |
| FENOFIBRATE NANOCRYSTALLIZED |
| FENOFIBRATE, MICRONIZED |
| FLUVASTATIN SODIUM |
| FOLIC ACID/NIACINAMIDE/CUPRIC OXIDE/ZINC OXIDE |
| FOLIC ACID/NIACINAMIDE/ZINC |
| GEMFIBROZIL |
| INOSITOL NIACINATE |
| IRON PYROPHOSPHATE/CYANOCOBALAMIN/FA/NIACIN/PYRIDOXINE HCL |
| LECITHIN/SITOSTEROLS/NIACIN/BETAINE/CHITOSAN |
| LOVASTATIN |
| LYSINE HCL/NIACINAMIDE/THIAMINE |
| MELATONIN/TRYPTOPHAN/VALERIAN/CHAMOMILE/NIACIN/INOSITOL/B6 |
| NIACIN |
| NIACIN (INOSITOL NIACINATE) |
| NIACIN/CAPSAICIN/YOHIMBE BARK/GINSENG/GNK BI EX/DAMIANA/OATS |
| NIACIN/LOVASTATIN |
| NIACIN/SIMVASTATIN |
| NIACINAMIDE |

| NIACINAMIDE ASCORBATE |
|--------------------------------------------------------------|
| NIACINAMIDE/AZELAIC ACID/ZINC OXIDE/VIT B6/COPPER/FA |
| PECTIN/INOSITOL/BIOFLAVONOIDS/NIACIN/SOYBEAN |
| PITAVASTATIN CALCIUM |
| POLICOSANOL/INOSITOL NIACINATE/GARLIC |
| PRAVASTATIN SODIUM |
| ROSUVASTATIN CALCIUM |
| SIMVASTATIN |
| SITAGLIPTIN PHOSPHATE/SIMVASTATIN |
| THIAMINE HCL/RIBOFLAVIN/NIACINAMIDE/CYANOCOBALAMIN/PROTEASE |
| THIAMINE HCL/RIBOFLAVIN/NIACINAMIDE/DEXPANTHENOL/PYRIDOXINE |
| THIAMINE M.NIT/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/B6/B12/C/FA |
| THIAMINE/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/B6/B12/VIT C/FA |
| THIAMINE/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/VIT B6/B12/IRON |
| THIAMINE/RIBOFLAVIN/NIACIN/PANT ACID/B6/IRON/METHION/CHOLINE |
| VITAMIN B COMPLEX/NIACINAMIDE/PANTOTHENIC ACID/HERBAL DRUGS |

| Antihypertensive Medications |
|-------------------------------------------------------|
| ACEBUTOLOL HCL |
| ALISKIREN HEMIFUMARATE/AMLODIPINE BESYLATE |
| ALISKIREN HEMIFUMARATE/AMLODIPINE/HYDROCHLOROTHIAZIDE |
| AMLODIPINE BESYLATE |
| AMLODIPINE BESYLATE/ATORVASTATIN CALCIUM |
| AMLODIPINE BESYLATE/BENAZEPRIL HCL |
| AMLODIPINE BESYLATE/OLMESARTAN MEDOXOMIL |
| AMLODIPINE BESYLATE/VALSARTAN |
| AMLODIPINE BESYLATE/VALSARTAN/HYDROCHLOROTHIAZIDE |
| APRACLONIDINE HCL |
| ATENOLOL |
| ATENOLOL/CHLORTHALIDONE |
| AZILSARTAN MEDOXOMIL |
| AZILSARTAN MEDOXOMIL/CHLORTHALIDONE |
| BENAZEPRIL HCL |
| BENAZEPRIL HCL/HYDROCHLOROTHIAZIDE |
| BENDROFLUMETHIAZIDE |
| BEPRIDIL HCL |
| BETAXOLOL HCL |
| BISOPROLOL FUMARATE |
| BISOPROLOL FUMARATE/HYDROCHLOROTHIAZIDE |
| BRIMONIDINE TARTRATE/TIMOLOL MALEATE |
| BUMETANIDE |
| CANDESARTAN CILEXETIL |
| CANDESARTAN CILEXETIL/HYDROCHLOROTHIAZIDE |
| CAPTOPRIL |
| CAPTOPRIL/HYDROCHLOROTHIAZIDE |
| CARTEOLOL HCL |
| CARVEDILOL |
| CARVEDILOL PHOSPHATE |
| CHLOROTHIAZIDE |
| CHLORTHALIDONE |

| CLEVIDIPINE BUTYRATE |
|-----------------------------------------------|
| CLONIDINE |
| CLONIDINE HCL |
| CLONIDINE HCL/CHLORTHALIDONE |
| CLONIDINE HCL/PF |
| DILTIAZEM HCL |
| DILTIAZEM HCL IN 0.9 % SODIUM CHLORIDE |
| DILTIAZEM HCL/DEXTROSE 5 % IN WATER |
| DILTIAZEM MALATE |
| DORZOLAMIDE HCL/TIMOLOL MALEATE |
| DORZOLAMIDE HCL/TIMOLOL MALEATE/PF |
| DOXAZOSIN MESYLATE |
| ENALAPRIL MALEATE |
| ENALAPRIL MALEATE/DILTIAZEM MALATE |
| ENALAPRIL MALEATE/FELODIPINE |
| ENALAPRIL MALEATE/HYDROCHLOROTHIAZIDE |
| ENALAPRILAT DIHYDRATE |
| EPLERENONE |
| EPROSARTAN MESYLATE |
| EPROSARTAN MESYLATE/HYDROCHLOROTHIAZIDE |
| ESMOLOL HCL |
| ETHACRYNIC ACID |
| FELODIPINE |
| FOSINOPRIL SODIUM |
| FOSINOPRIL SODIUM/HYDROCHLOROTHIAZIDE |
| FUROSEMIDE |
| GUANABENZ ACETATE |
| GUANADREL SULFATE |
| GUANETHIDINE SULFATE |
| GUANFACINE HCL |
| HYDRALAZINE HCL |
| HYDRALAZINE HCL/HYDROCHLOROTHIAZIDE |
| HYDRALAZINE HCL/RESERPINE/HYDROCHLOROTHIAZIDE |

| HYDROCHLOROTHIAZIDE |
|------------------------------------------|
| HYDROFLUMETHIAZIDE |
| INDAPAMIDE |
| IRBESARTAN |
| IRBESARTAN/HYDROCHLOROTHIAZIDE |
| ISOSORBIDE DINITRATE |
| ISOSORBIDE DINITRATE/HYDRALAZINE HCL |
| ISOSORBIDE MONONITRATE |
| ISRADIPINE |
| LABETALOL HCL |
| LISINOPRIL |
| LISINOPRIL/DIETARY SUPPLEMENT, COMB. 10 |
| LISINOPRIL/HYDROCHLOROTHIAZIDE |
| LOSARTAN POTASSIUM |
| LOSARTAN POTASSIUM/HYDROCHLOROTHIAZIDE |
| METHYCLOTHIAZIDE |
| METHYLDOPA |
| METHYLDOPA/CHLOROTHIAZIDE |
| METHYLDOPA/HYDROCHLOROTHIAZIDE |
| METHYLDOPATE HCL |
| METOLAZONE |
| METOPROLOL SUCCINATE |
| METOPROLOL SUCCINATE/HYDROCHLOROTHIAZIDE |
| METOPROLOL TARTRATE |
| METOPROLOL TARTRATE/HYDROCHLOROTHIAZIDE |
| METYROSINE |
| MIBEFRADIL DI-HCL |
| MINOXIDIL |
| MOEXIPRIL HCL |
| MOEXIPRIL HCL/HYDROCHLOROTHIAZIDE |
| NEBIVOLOL HCL |
| NICARDIPINE HCL |
| NIFEDIPINE |

| NIMODIPINE |
|--------------------------------------------------------------|
| NISOLDIPINE |
| NITROGLYCERIN |
| OLMESARTAN MEDOXOMIL |
| OLMESARTAN MEDOXOMIL/AMLODIPINE BESYLATE/HYDROCHLOROTHIAZIDE |
| OLMESARTAN MEDOXOMIL/HYDROCHLOROTHIAZIDE |
| PERINDOPRIL ARGININE/AMLODIPINE BESYLATE |
| PERINDOPRIL ERBUMINE |
| POLYTHIAZIDE |
| PRAZOSIN HCL |
| PRAZOSIN HCL/POLYTHIAZIDE |
| QUINAPRIL HCL |
| QUINAPRIL HCL/HYDROCHLOROTHIAZIDE |
| RAMIPRIL |
| RANOLAZINE |
| RESERPINE |
| RESERPINE/CHLOROTHIAZIDE |
| RESERPINE/HYDROCHLOROTHIAZIDE |
| RESERPINE/HYDROFLUMETHIAZIDE |
| RESERPINE/METHYCLOTHIAZIDE |
| RESERPINE/POLYTHIAZIDE |
| SOTALOL HCL |
| SPIRONOLACTONE |
| TELMISARTAN |
| TELMISARTAN/AMLODIPINE BESYLATE |
| TELMISARTAN/HYDROCHLOROTHIAZIDE |
| TERAZOSIN HCL |
| TIMOLOL |
| TIMOLOL MALEATE |
| TIMOLOL MALEATE/HYDROCHLOROTHIAZIDE |
| TIMOLOL MALEATE/PF |
| TORSEMIDE |
| TRANDOLAPRIL |

| TRANDOLAPRIL/VERAPAMIL HCL |
|-------------------------------|
| TRIAMTERENE |
| TRICHLORMETHIAZIDE |
| VALSARTAN |
| VALSARTAN/HYDROCHLOROTHIAZIDE |
| VERAPAMIL HCL |

# Pregnancy Dx codes 650 NORMAL DELIVERY 660 OBSTRUCTED LABOR 661 ABNORMALITY OF FORCES OF LABOR 662 LONG LABOR 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY 665 OTHER OBSTETRICAL TRAUMA 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND DELIVERY 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR COMPLICATION V24 POSTPARTUM CARE AND EXAMINATION V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER V24.2 ROUTINE POSTPARTUM FOLLOW V27 OUTCOME OF DELIVERY V27.0 MOTHER WITH SINGLE LIVEBORN V27.1 MOTHER WITH SINGLE STILLBORN V27.2 MOTHER WITH TWINS BOTH LIVEBORN V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN V27.4 MOTHER WITH TWINS BOTH STILLBORN V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY Procedure codes 72.0 LOW FORCEPS OPERATION 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY 72.2 MID FORCEPS OPERATION 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY 72.29 OTHER MID FORCEPS OPERATION 72.3 HIGH FORCEPS OPERATION 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY 72.39 OTHER HIGH FORCEPS OPERATION
#### Appendix A

- 72.4 FORCEPS ROTATION OF FETAL HEAD
  72.5 BREECH EXTRACTION
  72.51 PARTIAL BREECH EXTRACTION WIT
- 72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.52 OTHER PARTIAL BREECH EXTRACTION
- 72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.54 OTHER TOTAL BREECH EXTRACTION
- 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD
- 72.7 VACUUM EXTRACTION
- 72.71 VACUUM EXTRACTION WITH EPISIOTOMY
- 72.79 OTHER VACUUM EXTRACTION
- 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY
- 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY
- 73.0 ARTIFICIAL RUPTURE OF MEMBRANES
- 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES
- 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES
- 73.1 OTHER SURGICAL INDUCTION OF LABOR
- 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION
- 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION
- 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION
- 73.3 FAILED FORCEPS
- 73.4 MEDICAL INDUCTION OF LABOR
- 73.5 MANUALLY ASSISTED DELIVERY
- 73.51 MANUAL ROTATION OF FETAL HEAD
- 73.59 OTHER MANUALLY ASSISTED DELIVERY
- 73.6 EPISIOTOMY
- 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY
- 73.9 OTHER OPERATIONS ASSISTING DELIVERY
- 73.91 EXTERNAL VERSION ASSISTING DELIVERY
- 73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD
- 73.93 INCISION OF CERVIX TO ASSIST DELIVERY
- 73.94 PUBIOTOMY TO ASSIST DELIVERY
- 73.99 OTHER OPERATIONS ASSISTING DELIVERY
- 74.0 CLASSICAL CESAREAN SECTION
- 74.1 LOW CERVICAL CESAREAN SECTION
- 74.2 EXTRAPERITONEAL CESAREAN SECTION

#### Appendix A

- 74.3 REMOVAL OF EXTRATUBAL ECTOPIC PREGNANCY
- 74.4 CESAREAN SECTION OF OTHER SPECIFIED TYPE
- 74.9 CESAREAN SECTION OF UNSPECIFIED TYPE
- 74.91 HYSTEROTOMY TO TERMINATE PREGNANCY
- 74.99 OTHER CESAREAN SECTION OF UNSPECIFIED TYPE
- 75.4 MANUAL REMOVAL OF RETAINED PLACENTA
- 75.5 REPAIR OF CURRENT OBSTETRIC LACERATION OF UTERUS
- 75.6 REPAIR OF OTHER CURRENT OBSTETRIC LACERATION
- 75.7 MANUAL EXPLORATION OF UTERINE CAVITY, POSTPARTUM
- 75.9 OTHER OBSTETRIC OPERATIONS

#### Appendix B



| C | Optu | m I | MarketS | can | Medicare | | | POOLED | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Reference-DPP4i v2 E | xposure - Dapaglifozin v2 | Reference-DPP4iv2 B | xposure - Dapaglifozin v2 | Reference-DPP4i v2 | Exposure -<br>Dapagirloan v2 | Reference-DPP4iv2 Exp | posure - Dapaglifozin v2 | St. Diff. |
| Number of patients | 43,710 | 3,481 | 70,087 | 13,292 | 220,061 | 9,217 | 333,858 | 25,990 | |
| Age | | | | | | | | | |
| mean (sd) | 64.48 (9.80) | 58.44 (6.69) | 61.12 (8.57) | 57.95 (5.83) | 73.25 (6.69) | 70.29 (4.93) | 69.56 (7.58) | 62.39 (5.66) | 1.07 |
| median (IQR) | 63.00 [57.00, 71.00] | 58.00 [54.00, 62.00] | 60.00 [36.00, 64.00] | 38.00 [35.00, 61.00] | 72.00 [68.00, 77.00] 9. | 00 [67.00, 73.00] | 68.30 (7.58) | 61.90 (5.66) | 0.96 |
| Age categories without zero category | | | | | | | | | |
| 18 - 34; n (%) | 6,388 (14.6%) | 907 (26.1%) | 12,884 (18.4%) | 3,220 (24.2%) | 0 (0.0%) | 0 (0.0%) | 19,272 (5.8%) | 4,127 (15.9%) | -0.33 |
| 55 -64; n (%) | 17,548 (40.1%) | 2,099 (60.3%) | 41,083 (58.6%) | 9,162 (68.9%) | 2,206 (1.0%) | 79 (0.9%) | 60,837 (18.2%) | 11,340 (43.6%) | -0.57 |
| 65 -74; n (%) | 12,125 (27.7%) | 390 (11.2%) | 9,946 (14.2%) | 754 (5.7%) | 138,975 (63.2%) | 7,545 (81.9%) | 161,046 (48.2%) | 8,689 (33.4%) | 0.30 |
| >=75; n (%) | 7,649 (17.5%) | 85 (2.4%) | 6,174 (8.8%) | 156 (1.2%) | 78,880 (35.8%) | 1,593 (17.3%) | 92,703 (27.8%) | 1,834 (7.1%) | 0.57 |
| Gender without zero category-United | | | | | | | | | |
| Maies; n (%) | 25,356 (58.0%) | 2,199 (63.2%) | 41,300 (58.9%) | 8,073 (60.7%) | 102,718 (46.7%) | 4,790 (52.0%) | 169,374 (50.7%) | 15,062 (58.0%) | -0.15 |
| Females; n (%) | 18,354 (42.0%) | 1,282 (36.8%) | 28,787 (41.1%) | 5,219 (39.3%) | 117,343 (53.3%) | 4,427 (48.0%) | 164,484 (49.3%) | 10,928 (42.0%) | 0.15 |
| Race | | | | | | | | | |
| White; n (%) | N/A | N/A | N/A | N/A | 165,288 (75.1%) | 7,433 (80.6%) | 165,288 (75.1%) | 7,433 (80.6%) | -0.13 |
| Black; n (%) | N/A | N/A | N/A | N/A | 24,910 (11.3%) | 760 (8.2%) | 24,910 (11.3%) | 760 (8.2%) | 0.10 |
| Asian; n (%) | N/A | N/A | N/A | N/A | 9,877 (4.5%) | 303 (3.3%) | 9,877 (4.5%) | 303 (3.3%) | 0.06 |
| Hispanic; n (%) | N/A | N/A | N/A | N/A | 9,330 (4.2%) | 298 (3.2%) | 9,330 (4.2%) | 298 (3.2%) | 0.05 |
| North American Native; n (%) | N/A | N/A | N/A | N/A | 1,273 (0.6%) | 25 (0.3%) | 1,273 (0.6%) | 25 (0.3%) | 0.04 |
| Other/Unknown; n (%) | N/A | N/A | N/A | N/A | 9,383 (4.3%) | 398 (4.3%) | 9,383 (4.3%) | 398 (4.3%) | 0.00 |
| Region without zero category-United v3 (lumping missings | Anther category with West | | | | | | | | |
| Northeast; n (%) | 5.438 (12.4%) | 223 (6.4%) | 14,081 (20.1%) | 1,756 (13.2%) | 43,499 (19.8%) | 1,537 (16.7%) | 63.018 (18.9%) | 3,516 (13.5%) | 0.15 |
| South; n (%) | 21,918 (50.1%) | 1,967 (56.5%) | 16,006 (22.8%) | 2,196 (16.5%) | 93,209 (42.4%) | 4.286 (46.5%) | 131.133 (39.3%) | 8,449 (32.5%) | 0.14 |
| Midwest; n (%) | 8,880 (20.3%) | 846 (24.3%) | 33,051 (47.2%) | 8,242 (62.0%) | 47,609 (21.6%) | 1,828 (19.8%) | 89,540 (26.8%) | 10,916 (42.0%) | -0.32 |
| West; n (%) | 7,474 (17.1%) | 445 (12.8%) | 6,248 (8.9%) | 1,033 (7.8%) | 35,744 (16.2%) | 1,366 (17.0%) | 49,466 (14.8%) | 3,044 (11.7%) | 0.09 |
| Unknown+missing; n (%) | N/A | N/A | 701 (1.0%) | 65 (0.5%) | N/A | N/A | 701 (1.0%) | 65 (0.5%) | 0.06 |
| CV Covariates | 140 | 140 | 702 [2.070] | p.ca) ca | inje. | 140 | 702 [2.076] | 05 (0.5/4) | 0.00 |
| Ischemic heart disease; n (%) | 12,863 (29,4%) | 666 (19.1%) | 13.724 (19.6%) | 2,236 (16.8%) | 52,757 (24.0%) | 2.042 (22.2%) | 79.344 (23.8%) | 4,944 (19.0%) | 0.12 |
| Acute MI; n (%) | 394 (1.4%) | 33 (0.9%) | 437 (0.6%) | 73 (0.5%) | 1,148 (0.5%) | 45 (0.5%) | 2,179 (0.7%) | 151 (0.6%) | 0.01 |
| ACS/unstable angina; n (%) | 773 (1.8%) | 39 (1.1%) | 590 (0.8%) | 104 (0.8%) | 1,486 (0.7%) | 52 (0.6%) | 2,849 (0.9%) | 195 (0.8%) | 0.01 |
| Old MI; n (%) | 1,758 (4.0%) | 80 (2.3%) | 1,031 (1.5%) | 149 (1.1%) | 5,358 (2.4%) | 190 (2.1%) | 8,147 (2.4%) | 419 (1.6%) | 0.06 |
| Stable angina; n (%) | 2,754 (6.3%) | 112 (3.2%) | 1,780 (2.5%) | 340 (2.6%) | 6,214 (2.8%) | 286 (3.1%) | 10,748 (3.2%) | 738 (2.8%) | 0.02 |
| 0 - (7 | | \ / | | 1 | . ( ) | | | , , | |
| Coronary atherosclerosis and other forms of chronic ischer | 11,791 (27.0%) | 621 (17.8%) | 12,885 (18.4%) | 2,047 (15.4%) | 50,482 (22.9%) | 1,958 (21.2%) | 75,158 (22.5%) | 4,626 (17.8%) | 0.12 |
| Other atherosclerosis with ICD10 v2 Copy; n (%) | 368 (0.8%) | 22 (0.6%) | 488 (0.7%) | 55 (0.4%) | 2,671 (1.2%) | 80 (0.9%) | 3,527 (1.1%) | 157 (0.6%) | 0.05 |
| Previous cardiac procedure (CABG or PTCA or Stent) v4; n (5 | 300 (0.7%) | 23 (0.7%) | 263 (0.4%) | 42 (0.3%) | 530 (0.2%) | 17 (0.2%) | 1,093 (0.3%) | 82 (0.3%) | 0.00 |
| History of CABG or PTCA; n (%) | 3,143 (7.2%) | 147 (4.2%) | 1,788 (2.6%) | 284 (2.1%) | 12,768 (5.8%) | 493 (5.3%) | 17,699 (5.3%) | 924 (3.6%) | 0.08 |
| Any stroke; n (%) | 3,268 (7.5%) | 119 (3.4%) | 3,412 (4.9%) | 441 (3.3%) | 15,616 (7.1%) | 343 (5.9%) | 22,296 (6.7%) | 1,105 (4.3%) | 0.11 |
| Ischemic stroke (w and w/o mention of cerebral infarction) | 3,222 (7.4%) | 115 (3.3%) | 3,384 (4.8%) | 441 (3.3%) | 15,455 (7.0%) | 344 (3.9%) | 22,061 (6.6%) | 1,100 (4.2%) | 0.11 |
| Hemorrhagic stroke; n (%) | 111 (0.3%) | 4 (0.1%) | 66 (0.1%) | 3 (0.0%) | | | | | |
| TIA; n (%) | 577 (1.3%) | 19 (0.5%) | 420 (0.6%) | 70 (0.5%) | 1,800 (0.8%) | 76 (0.8%) | 2,797 (0.8%) | 163 (0.6%) | 0.02 |
| Other cerebrovascular disease; n (%) | 797 (1.8%) | 22 (0.6%) | 688 (1.0%) | 82 (0.6%) | 3,866 (1.8%) | 113 (1.2%) | 5,351 (1.6%) | 217 (0.8%) | 0.07 |
| Late effects of cerebrovascular disease; n (%) | 825 (1.9%) | 14 (0.4%) | 481 (0.7%) | 52 (0.4%) | 3,254 (1.5%) | 79 (0.9%) | 4,560 (1.4%) | 143 (0.6%) | 0.08 |
| Cerebrovascular procedure; n (%) | 73 (0.2%) | 4 (0.1%) | 53 (0.1%) | 5 (0.0%) | 40.004 (0.004) | | 24 224 (2 28) | ana (n. 1911) | |
| Heart failure (CHF); n (%) | 3,344 (7.7%) | 147 (4.2%) | 2,486 (3.5%) | 300 (2.3%) | 15,991 (7.3%) | 311 (3.3%) | 21,821 (6.5%) | 958 (3.7%) | 0.13 |
| Peripheral Vascular Disease (PVD) or PVD Surgery v2; n (%) | 3,644 (8.3%) | 128 (3.7%) | 2,871 (4.1%) | 407 (3.1%) | 19,371 (8.8%) | 645 (7.0%) | 25,886 (7.8%) | 1,180 (4.5%) | 0.14 |
| Atrial fibrillation; n (%) | 3,088 (7.1%) | 121 (3.5%) | 3,280 (4.7%) | 384 (2.9%) | 20,557 (9.3%) | 684 (7.4%) | 26,925 (8.1%) | 1,180 (4.6%) | 0.14 |
| Other cardiac dysrhythmia; n (%) | 4,016 (9.2%) | 184 (5.3%) | 4,007 (5.7%) | 509 (3.8%) | 22,999 (10.5%) | 846 (9.2%) | 31,022 (9.3%) | 1,539 (5.9%) | 0.14 |
| Cardiac conduction disorders; n (%) | 1,154 (2.6%) | 55 (1.6%) | 1,065 (1.5%) | 152 (1.1%) | 6,593 (3.0%) | 234 (2.5%) | 8,812 (2.6%) | 441 (1.7%) | 0.06 |
| Other CVD; n (%) | 4,947 (11.3%) | 232 (6.7%) | 5,164 (7.4%) | 668 (5.0%) | 26,017 (11.8%) | 932 (10.1%) | 36,128 (10.8%) | 1,832 (7.0%) | 0.13 |
| Diabetes-related complications | | | -,(,) | 222 (2.274) | | () | , | -,(,,,-) | |
| Diabetic retinopathy; n (%) | 2,281 (5.2%) | 152 (4.4%) | 2,156 (3.1%) | 410 (3.1%) | 13,152 (6.0%) | 623 (6.8%) | 17,589 (5.3%) | 1,185 (4.6%) | 0.03 |
| | | | -,() | | ,[0.4] | ( | , | -,( | |
| Diabetes with other ophthalmic manifestations; n (%) | 270 (0.6%) | 3 (0.1%) | 1,356 (1.9%) | 223 (1.7%) | 5,038 (2.3%) | 194 (2.1%) | 6,664 (2.0%) | 420 (1.6%) | 0.03 |
| Retinal detachment, vitreous hemorrhage, vitrectomy; n (7 | 140 (0.3%) | 10 (0.3%) | 179 (0.3%) | 33 (0.2%) | 703 (0.3%) | 31 (0.3%) | 1,022 (0.3%) | 74 (0.3%) | 0.00 |
| Retinal laser coagulation therapy; n (%) | 189 (0.4%) | 8 (0.2%) | 305 (0.4%) | 58 (0.4%) | 1,041 (0.5%) | 60 (0.7%) | 1,535 (0.5%) | 126 (0.5%) | 0.00 |
| Occurrence of Diabetic Neuropathy v2 Copy; n (%) | 7,714 (17.6%) | 306 (14.5%) | 7,231 (10.3%) | 1,572 (11.8%) | 37,142 (16.9%) | 1,753 (19.0%) | 52,087 (15.6%) | 3,831 (14.7%) | 0.03 |

| Occurrence of diabetic nephropathy V3 with ICD10 Copy; r | 3,743 (8.6%) | 180 (5.2%) | 2,838 (4.0%) | 525 (3.9%) | 12,264 (5.6%) | 503 (5.5%) | 18,845 (5.6%) | 1,208 (4.6%) | 0.05 |
|---|---|---|---|---|---|---|---|---|---|
| Hypoglycemia v2; n (%) | 983 (2.2%) | 76 (2.2%) | 1,292 (1.8%) | 215 (1.6%) | 4,479 (2.0%) | 116 (1.3%) | 6,754 (2.0%) | 407 (1.6%) | 0.03 |
| Hyperglycemia; n (%) | 1,941 (4.4%) | 109 (3.1%) | 2,407 (3.4%) | 462 (3.5%) | 8,655 (3.9%) | 346 (3.8%) | 13,003 (3.9%) | 917 (3.5%) | 0.02 |
| 11-01 | | | | | | | | , , , | |
| Disorders of fluid electrolyte and acid-base balance; n (%) | 2,385 (5.5%) | 99 (2.8%) | 2,318 (3.3%) | 351 (2.6%) | 11,157 (5.1%) | 289 (3.1%) | 15,860 (4.8%) | 739 (2.8%) | 0.10 |
| Diabetic ketoacidosis; n (%) | 75 (0.2%) | 7 (0.2%) | 112 (0.2%) | 12 (0.1%) | 388 (0.2%) | 10 (0.1%) | 575 (0.2%) | 29 (0.1%) | 0.03 |
| District Income and Infra | 12 (5.274) | 7 (0.274) | 222 (0.234) | 22 (0.279) | 300 (0.234) | 20 (0.204) | 575 (5.274) | 25 (0.274) | 0.00 |
| December 1 | num (n mik) | 10 (0.3%) | 287 (0.4%) | 49 (0.4%) | 906 (0.4%) | 50 (0.5%) | 1,411 (0,4%) | 109 (0.4%) | 0.00 |
| Hyperosmolar hyperglycemic nonketotic syndrome (HONK | 218 (0.5%) | 10 (0.3%) | 287 (0.4%) | 49 (0.476) | 906 (0.476) | 30 (0.3%) | 1,411 (0.4%) | 109 (0.4%) | 0.00 |
| Diabetes with peripheral circulatory disorders with ICD-10 | 3,048 (7.0%) | 122 (3.5%) | 2,146 (3.1%) | 302 (2.3%) | 13,823 (6.3%) | 524 (5.7%) | 19,017 (5.7%) | 948 (3.6%) | 0.10 |
| Diabetic Foot; n (%) | 998 (2.3%) | 69 (2.0%) | 1,020 (1.5%) | 196 (1.5%) | 4,442 (2.0%) | 169 (1.8%) | 6,460 (1.9%) | 434 (1.7%) | 0.02 |
| Gangrenev2; n (%) | 143 (0.3%) | 6 (0.2%) | 127 (0.2%) | 19 (0.1%) | | | | | ** |
| Lower extremity amputation; n (%) | 413 (0.9%) | 22 (0.6%) | 223 (0.3%) | 43 (0.3%) | 922 (0.4%) | 29 (0.3%) | 1,558 (0.5%) | 094 (0.4%) | 0.01 |
| Osteomyelitis; n (%) | 326 (0.7%) | 21 (0.6%) | 270 (0.4%) | 56 (0.4%) | 862 (0.4%) | 28 (0.3%) | 1,458 (0.4%) | 105 (0.4%) | 0.00 |
| Skin infections v2; n (%) | 2,389 (5.5%) | 200 (5.7%) | 3,272 (4.7%) | 634 (4.9%) | 12,212 (5.5%) | 521 (5.7%) | 17,873 (5.4%) | 1,375 (5.3%) | 0.00 |
| Brectile dysfunction; n (%) | 1,344 (3.1%) | 148 (4.3%) | 1,904 (2.7%) | 416 (3.1%) | 4,876 (2.2%) | 268 (2.9%) | 8,124 (2.4%) | 832 (3.2%) | -0.05 |
| 1 | | \ <i>\</i> | | , , | | | | , , | |
| Diabetes with unspecified complication; n (%) | 2,256 (5.2%) | 139 (4.0%) | 3,047 (4.3%) | 724 (5.4%) | 9,808 (4.5%) | 520 (5.6%) | 15,111 (4.5%) | 1,383 (5.3%) | -0.04 |
| Diabetes mellitus without mention of complications; n [%] | 38,070 (87.1%) | 3,082 (88.5%) | 63,750 (91.0%) | 11,623 (87.4%) | 203,187 (92.3%) | 8,184 (88.8%) | 305,007 (91.4%) | 22,889 (88.1%) | 0.11 |
| Hypertension: 1 inpatient or 2 outpatient claims within 36 | 35,414 (81.0%) | 2,709 (77.8%) | 50,237 (71.7%) | 9,739 (73.3%) | 191,800 (87.2%) | 7,981 (86.6%) | 277,451 (83.1%) | 20,429 (78.6%) | 0.11 |
| Hyperlipidemia v2; n (%) | 31,957 (73.1%) | 2,632 (75.6%) | 47,756 (68.1%) | 9,565 (72.0%) | 167,881 (76.3%) | 7,097 (77.0%) | 247,594 (74.2%) | 19,294 (74.2%) | 0.00 |
| Edema; n (%) | 2,298 (5.3%) | 153 (4.4%) | 2,224 (3.2%) | 370 (2.8%) | 14,695 (6.7%) | 559 (6.1%) | 19,217 (5.8%) | 1,082 (4.2%) | 0.07 |
| Renal Dysfunction (non-diabetic) v2; n (%) | 4,552 (10.4%) | 148 (4.3%) | 3,654 (5.2%) | 420 (3.2%) | 21,679 (9.9%) | 525 (5.7%) | 29,885 (9.0%) | 1,093 (4.2%) | 0.19 |
| Occurrence of acute renal disease v2; n (%) | 817 (1.9%) | 15 (0.4%) | 736 (1.1%) | 53 (0.4%) | 3.193 (1.5%) | 51 (0.6%) | 4,746 (1.4%) | 119 (0.5%) | 0.09 |
| Occurrence of chronic renal insufficiency; n (%) | 2,889 (6.6%) | 96 (2.8%) | 1,885 (2.7%) | 225 (1.7%) | 14,526 (6.6%) | 330 (3.6%) | 19,300 (5.8%) | 651 (2.5%) | 0.17 |
| Chronic kidney diseasev2; n (%) | 2,594 (5.9%) | 79 (2.3%) | 1,599 (2.3%) | 184 (1.4%) | 12,582 (5.7%) | 285 (3.1%) | 16,775 (5.0%) | 548 (2.1%) | 0.16 |
| | | | | , , | | | | | |
| OXD Stage 3-4; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #VALUE! | 000 (0.0%) | #VALUE! |
| Occurrence of hypertensive nephropathy; n (%) | 1,135 (2.6%) | 41 (1.2%) | 811 (1.2%) | 103 (0.8%) | 4,671 (2.1%) | 137 (1.5%) | 6,617 (2.0%) | 281 (1.1%) | 0.07 |
| Occurrence of miscellaneous renal insufficiency v2; n (%) | 1,450 (3.3%) | 55 (1.6%) | 1,386 (2.0%) | 149 (1.1%) | 8,794 (4.0%) | 238 (2.6%) | 11,630 (3.5%) | 442 (1.7%) | 0.11 |
| Glaucoma or cataracts v2; n (%) | 7,468 (17.1%) | 424 (12.2%) | 9,759 (13.9%) | 1,525 (11.5%) | 57,293 (26,0%) | 2,348 (25.5%) | 74,520 (22.3%) | 4,297 (16.5%) | 0.15 |
| Cellulitis or abscess of toe; n (%) | 574 (1.3%) | 32 (0.9%) | 616 (0.9%) | 128 (1.0%) | 2,388 (1.1%) | 119 (1.3%) | 3,578 (1.1%) | 279 (1.1%) | 0.00 |
| Footuicer; n (%) | 961 (2.2%) | 64 (1.8%) | 1,012 (1,4%) | 196 (1.5%) | 4,383 (2.0%) | 164 (1.8%) | 6,356 (1.9%) | 424 (1.6%) | 0.02 |
| | 32 (0.1%) | 0 (0.0%) | 34 (0.0%) | | 4,363 [2.076] | 104 [1.0/0] | 0,330 (1.376) | 424 [1.0/0] | 0.02 |
| Bladder stones; n (%) | | | | 6 (0.0%) | | | | | |
| Kidney stones; n (%) | 652 (1.5%) | 49 (1.4%) | 971 (1.4%) | 164 (1.2%) | 3,229 (1.5%) | 135 (1.5%) | 4,852 (1.5%) | 348 (1.3%) | 0.02 |
| Uninary tract infections (UTIs); n (%) | 310 (0.7%) | 6 (0.2%) | 322 (0.5%) | 39 (0.4%) | 1,604 (0.7%) | 63 (0.7%) | 2,236 (0.7%) | 128 (0.5%) | 0.03 |
| Dipstick urinalysis; n (%) | 13,140 (30.1%) | 896 (25.7%) | 19,643 (28.0%) | 3,866 (29.1%) | 66,715 (30.3%) | 2,706 (29.4%) | 99,498 (29.8%) | 7,468 (28.7%) | 0.02 |
| Non-dipstick urinalysis; n (%) | 17,924 (41.0%) | 1,446 (41.5%) | 24,807 (35.4%) | 5,524 (41.6%) | 88,718 (40.3%) | 3,834 (41.6%) | 131,449 (39.4%) | 10,804 (41.6%) | -0.04 |
| Urine function test; n (%) | 597 (1.4%) | 27 (0.8%) | 986 (1.4%) | 118 (0.9%) | 4,593 (2.1%) | 171 (1.9%) | 6,176 (1.8%) | 316 (1.2%) | 0.05 |
| Cytology; n (%) | 149 (0.3%) | 6 (0.2%) | 185 (0.3%) | 21 (0.2%) | 627 (0.3%) | 30 (0.3%) | #VALUE! | 57 (0.2%) | #VALUE! |
| Cystoscopy; n (%) | 148 (0.3%) | 10 (0.3%) | 281 (0.4%) | 38 (0.3%) | 883 (0.4%) | 34 (0.4%) | 1,312 (0.4%) | 082 (0.3%) | 0.02 |
| Other Covariates | 240 (0.374) | 20(0.3/4) | 202 (0.475) | 30 (0.374) | 203 (0.474) | 24 (0.474) | 2,522 (6.474) | 002 (0.3/9) | 0.02 |
| | a nen in alki | | a fa alk l | o in offil | a in alt | a in air l | a nen in alti | ene (e elle) | |
| Liver disease; n (%) | 1,363 (3.1%) | 75 (2.2%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 1,363 (0.4%) | 075 (0.3%) | 0.02 |
| Osteoarthritis; n (%) | 6,248 (14.3%) | 369 (10.6%) | 7,550 (10.8%) | 1,251 (9.4%) | 44,989 (20.4%) | 1,818 (19.7%) | 58,787 (17.6%) | 3,438 (13.2%) | 0.12 |
| Other arthritis, arthropathies and musculoskeletal pain; n | 15,128 (34.6%) | 1,076 (30.9%) | 20,490 (29.2%) | 3,770 (28.4%) | 87,318 (39.7%) | 3,527 (38.3%) | 122,936 (36.8%) | 8,373 (32.2%) | 0.10 |
| Dorsopathies; n (%) | 9,446 (21.6%) | 711 (20.4%) | 12,419 (17.7%) | 2,401 (18.1%) | 52,738 (24.0%) | 2,297 (24.9%) | 74,603 (22.3%) | 5,409 (20.8%) | 0.04 |
| Fractures; n (%) | 1,033 (2.4%) | 39 (1.7%) | 1,335 (1.9%) | 174 (1.3%) | 6,400 (2.9%) | 204 (2.2%) | 8,768 (2.6%) | 437 (1.7%) | 0.06 |
| Fallsv2; n (%) | 1,217 (2.8%) | 42 (1.2%) | 730 (1.0%) | 65 (0.5%) | 7,186 (3.3%) | 202 (2.2%) | 9,133 (2.7%) | 309 (1.2%) | 0.11 |
| Osteoporosis; n (%) | 1,611 (3.7%) | 57 (1.6%) | 1,263 (1.8%) | 144 (1.1%) | 15,514 (7.0%) | 485 (5.3%) | 18,388 (5.5%) | 686 (2.6%) | 0.15 |
| Hyperthyroidism; n (%) | 283 (0.6%) | 20 (0.6%) | 373 (0.5%) | 73 (0.5%) | 1.823 (0.8%) | 71 (0.8%) | 2,479 (0.7%) | 164 (0.6%) | 0.01 |
| Hypothyroidism v2; n (%) | 6,367 (14.6%) | 492 (14.1%) | 8,029 (11.5%) | 1,618 (12.2%) | 26,926 (12.2%) | 966 (10.5%) | 41,322 (12.4%) | 3,076 (11.8%) | 0.02 |
| Other disorders of thyroid gland V2; n (%) | 1,621 (3.7%) | 146 (4.2%) | 2,343 (3.3%) | 512 (3.9%) | 8,530 (3.9%) | 426 (4.6%) | 12,494 (3.7%) | 1,084 (4.2%) | -0.03 |
| | | · · | | | | | | | |
| Depression; n (%) | 3,619 (8.3%) | 251 (7.2%) | 4,285 (6.1%) | 852 (6.4%) | 19,362 (8.8%) | 702 (7.6%) | 27,266 (8.2%) | 1,805 (6.9%) | 0.05 |
| Anxiety; n (%) | 3,526 (8.1%) | 223 (6.4%) | 3,861 (5.5%) | 795 (6.0%) | 16,485 (7.5%) | 657 (7.1%) | 23,872 (7.2%) | 1,675 (6.4%) | 0.03 |
| Sleep_Disorder; n (%) | 2,998 (6.9%) | 348 (10.0%) | 5,787 (8.3%) | 1,097 (8.3%) | 14,646 (6.7%) | 530 (5.8%) | 23,431 (7.0%) | 1,975 (7.6%) | -0.02 |
| Dementia; n (%) | 1,413 (3.2%) | 24 (0.7%) | 1,007 (1.4%) | 62 (0.5%) | 11,942 (5.4%) | 218 (2.4%) | 14,362 (4.3%) | 304 (1.2%) | 0.19 |
| Delirium; n (%) | 381 (0.9%) | 12 (0.3%) | 317 (0.5%) | 25 (0.2%) | 2,125 (1.0%) | 38 (0.4%) | 2,823 (0.8%) | 75 (0.3%) | 0.07 |
| Psychosis; n (%) | 463 (1.1%) | 12 (0.3%) | 337 (0.5%) | 37 (0.3%) | 3,030 (1,4%) | 62 (0.7%) | 3,830 (1.1%) | 111 (0.4%) | 0.08 |
| Obesity; n (%) | 8,934 (20.4%) | 909 (26.1%) | 10,456 (14.9%) | 2,628 (19.8%) | 28,022 (12.7%) | 1,534 (16.6%) | 47,412 (14.2%) | 5,071 (19.5%) | -0.14 |
| Overweight; n (%) | 2,478 (5.7%) | 148 (4.3%) | 1,974 (2.8%) | 371 (2.8%) | 8,173 (3.7%) | 369 (4.0%) | 12,625 (3.8%) | 888 (3.4%) | 0.02 |
| Smoking; n (%) | 5,327 (12.2%) | 326 (9.4%) | 4,014 (5.7%) | 706 (5.3%) | 23,022 (10.5%) | 981 (10.6%) | 32,363 (9.7%) | 2,013 (7.7%) | 0.02 |
| Alcohol abuse or dependence; n (%) | 393 (0.9%) | 27 (0.8%) | 340 (0.5%) | 46 (0.3%) | 1,034 (0.5%) | 41 (0.4%) | 1,767 (0.5%) | 114 (0.4%) | 0.01 |
| Drug abuse or dependence; n (%) | 631 (1.4%) | 31 (0.9%) | 415 (0.6%) | 73 (0.5%) | 1,673 (0.8%) | 78 (0.8%) | 2,719 (0.8%) | 182 (0.7%) | 0.01 |
| COPD; n (%) | 3,746 (8.6%) | 138 (4.0%) | 3,000 (4.3%) | 386 (2.9%) | 19,590 (8.9%) | 752 (8.2%) | 26,336 (7.9%) | 1,276 (4.9%) | 0.12 |

| Asthma; n (%) | 2,352 (5.4%) | 162 (4.7%) | 2,922 (4.2%) | 479 (3.6%) | 11,824 (5.4%) | 496 (5.4%) | 17,098 (5.1%) | 1,137 (4.4%) | 0.03 |
|---|---|---|---|---|---|---|---|---|---|
| Obstructive sleep apnea; n (%) | 4,416 (10.1%) | 410 (11.8%) | 7,088 (10.1%) | 1,623 (12.2%) | 13,492 (6.1%) | 847 (9.2%) | 24,996 (7.5%) | 2,880 (11.1%) | -0.12 |
| Pneumonia; n (%) | 860 (2.0%) | 43 (1.2%) | 998 (1.4%) | 121 (0.9%) | 4,495 (2.0%) | 134 (1.5%) | 6,353 (1.9%) | 298 (1.1%) | 0.07 |
| Imaging; n (%) | 66 (0.2%) | 1 (0.0%) | 24 (0.0%) | 3 (0.0%) | • | • | • | | •• |
| Diabetes Medications | complex of the | -1 | | | | | () | | |
| DM Medications - AGIs; n (%) | 187 (0.4%) | 7 (0.2%) | 203 (0.3%) | 35 (0.3%) | 1,130 (0.5%) | 57 (0.6%) | 1,520 (0.5%) | 99 (0.4%) | 0.01 |
| DM Medications - Glitazones; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #VALUE! | 000 (0.0%) | #VALUE! |
| DM Medications - GLP-1 RA; n (%) | 1,549 (3.5%) | 754 (21.7%) | 2,487 (3.5%) | 2,764 (20.8%) | 4,959 (2.3%) | 1,316 (16.4%) | 8,995 (2.7%) | 5,034 (19.4%) | -0.55 |
| DM Medications - Insulin; n (%) | 6,845 (15.7%) | 933 (26.8%) | 8,963 (12.8%) | 3,433 (25.8%) | 33,577 (15.3%) | 2,551 (27.7%) | 49,385 (14.8%) | 6,917 (26.6%) | -0.29 |
| DM Medications - Meglitinides; n (%) | 407 (0.9%) | 21 (0.6%) | 761 (1.1%) | 117 (0.9%) | 3,328 (1.5%) | 154 (1.7%) | 4,496 (1.3%) | 292 (1.1%) | 0.02 |
| DM Medications - Metformin; n (%) | 33,521 (76.7%) | 2,635 (75.7%) | 56,594 (80.7%) | 10,496 (79.0%) | 163,913 (74.5%) | 6,881 (74.7%) | 254,028 (76.1%) | 20,012 (77.0%) | -0.02 |
| Concomitant initiation or current use of 2nd Generation S | 13,270 (30.4%) | 919 (26.4%) | 20,051 (28.6%) | 3,167 (23.8%) | 77,226 (35.1%) | 2,975 (32.3%) | 110,547 (33.1%) | 7,061 (27.2%) | 0.13 |
| Concomitant initiation or current use of AGIs; n (%) | 131 (0.3%) | 3 (0.1%) | 138 (0.2%) | 23 (0.2%) | 829 (0.4%) | 40 (0.4%) | 1,098 (0.3%) | 66 (0.3%) | 0.00 |
| Concomitant initiation or current use of Glitazones; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #VALUE! | 000 (0.0%) | #VALUE! |
| Concomitant initiation or current use of GLP-1 RA; n (%) | 901 (2.1%) | 531 (15.3%) | 1,451 (2.1%) | 1,985 (14.9%) | 2,539 (1.2%) | 1,128 (12.2%) | 4,891 (1.5%) | 3,644 (14.0%) | -0.48 |
| Concomitant initiation or current use of Insulin; n (%) | 5,120 (11.7%) | 687 (19.7%) | 6,746 (9.6%) | 2,633 (19.8%) | 25,867 (11.8%) | 2,042 (22.2%) | 37,733 (11.3%) | 5,362 (20.6%) | -0.26 |
| Concomitant initiation or current use of Meglitinides; n (% | 299 (0.7%) | 14 (0.4%) | 568 (0.8%) | 68 (0.5%) | 2,421 (1.1%) | 108 (1.2%) | 3,288 (1.0%) | 190 (0.7%) | 0.03 |
| Concomitant initiation or current use of Metformin; n (%) | 29,232 (66.9%) | 2,143 (61.6%) | 50,259 (71.7%) | 9,068 (68.2%) | 142,769 (64.9%) | 5,925 (64.3%) | 222,260 (66.6%) | 17,136 (65.9%) | 0.01 |
| Past use of 2nd Generation SUs Copy; n (%) | 3,105 (7.1%) | 280 (8.0%) | 4,603 (6.6%) | 855 (6.4%) | 15,787 (7.2%) | 632 (6.9%) | 23,495 (7.0%) | 1,767 (6.8%) | 0.01 |
| Past use of AGIs Copy; n (%) | 56 (0.1%) | 4 (0.1%) | 65 (0.1%) | 12 (0.1%) | 301 (0.1%) | 17 (0.2%) | 422 (0.1%) | 33 (0.1%) | 0.00 |
| Past use of Glitazones Copy; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #VALUE! | 000 (0.0%) | #VALUE! |
| Past use of GLP-1 RA Copy; n (%) | 705 (1.6%) | 254 (7.3%) | 1,101 (1.6%) | 839 (6.3%) | 2,421 (1.1%) | 388 (4.2%) | 4,227 (1.3%) | 1,481 (5.7%) | -0.24 |
| Past use of Insulin Copy; n (%) | 1,725 (3.9%) | 246 (7.1%) | 2,218 (3.2%) | 800 (6.0%) | 7,713 (3.5%) | 509 (5.5%) | 11,656 (3.5%) | 1,555 (6.0%) | -0.12 |
| Past use of Meglitinides Copy; n (%) | 108 (0.2%) | 7 (0.2%) | 193 (0.3%) | 49 (0.4%) | 907 (0.4%) | 46 (0.5%) | 1,208 (0.4%) | 102 (0.4%) | 0.00 |
| Past use of metiformin (final) Copy; n (%) | 4,289 (9.8%) | 492 (14.1%) | 6,335 (9.0%) | 1,428 (10.7%) | 21,144 (9.6%) | 956 (10.4%) | 31,768 (9.5%) | 2,876 (11.1%) | -0.05 |
| Other Medications | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 19,467 (44.5%) | 1,538 (44.2%) | 30,496 (43.5%) | 5,845 (44.0%) | 97,611 (44.4%) | 3,934 (42.7%) | 147,574 (44.2%) | 11,317 (43.5%) | 0.01 |
| Use of ARBs; n (%) | 12,584 (28.8%) | 999 (28.7%) | 20,278 (28.9%) | 4,039 (30.4%) | 69,754 (31.7%) | 3,122 (33.9%) | 102,616 (30.7%) | 8,160 (31.4%) | -0.02 |
| Use of Loop Diuretics - United; n (%) | 5,037 (11.5%) | 242 (7.0%) | 5,607 (8.0%) | 892 (6.7%) | 31,180 (14.2%) | 1,117 (12.1%) | 41,824 (12.5%) | 2,251 (8.7%) | 0.12 |
| Use of other diuretics- United; n (%) | 1,343 (3.1%) | 74 (2.1%) | 1,784 (2.5%) | 307 (2.3%) | 6,652 (3.0%) | 278 (3.0%) | 9,779 (2.9%) | 659 (2.5%) | 0.02 |
| Use of nitrates-United; n (%) | 3,045 (7.0%) | 137 (3.9%) | 3,294 (4.7%) | 474 (3.6%) | 13,835 (6.3%) | 474 (5.1%) | 20,174 (6.0%) | 1,085 (4.2%) | 0.08 |
| Use of other hypertension drugs; n (%) | 2,609 (6.0%) | 134 (3.8%) | 3,205 (4.6%) | 489 (3.7%) | 15,257 (6.9%) | 550 (6.0%) | 21,071 (6.3%) | 1,173 (4.5%) | 0.08 |
| Use of digoxin-United; n (%) | 757 (1.7%) | 33 (0.9%) | 977 (1.4%) | 91 (0.7%) | 5,889 (2.7%) | 198 (2.1%) | 7,623 (2.3%) | 322 (1.2%) | 0.08 |
| Use of Anti-errhythmics; n (%) | 613 (1.4%) | 28 (0.8%) | 807 (1.2%) | 110 (0.8%) | 3,689 (1.7%) | 122 (1.3%) | 5,109 (1.5%) | 260 (1.0%) | 0.05 |
| Use of COPD/asthma meds- United; n (%) | 6,650 (15.2%) | 414 (11.9%) | 10,129 (14.5%) | 1,811 (13.6%) | 36,341 (16.5%) | 1,501 (16.3%) | 53,120 (15.9%) | 3,726 (14.3%) | 0.04 |
| Use of statins; n (%) | 30,612 (70.0%) | 2,331 (67.0%) | 46,308 (66.1%) | 8,857 (66.6%) | 156,377 (71.1%) | 6,648 (72.1%) | 233,297 (69.9%) | 17,836 (68.6%) | 0.03 |
| Use of other lipid-lowering drugs; n (%) | 5,220 (11.9%) | 475 (13.6%) | 9,349 (13.3%) | 1,910 (14.4%) | 26,311 (12.0%) | 1,189 (12.9%) | 40,880 (12.2%) | 3,574 (13.8%) | -0.05 |
| Use of antiplatelet agents; n (%) | 7,356 (16.8%) | 404 (11.6%) | 9,660 (13.8%) | 1,637 (12.3%) | 30,271 (13.8%) | 1,179 (12.8%) | 47,287 (14.2%) | 3,220 (12.4%) | 0.05 |
| ose or an aprilia a apartit, in (14) | 7,250 (20.074) | 404 (22.074) | 3,000 [23.07] | 2,037 (22.374) | 30,272 (23.079) | 2,275 (22.079) | 47,207 (24.274) | 3,220 (22,470) | 0.03 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, Apixal | 2,845 (6.5%) | 148 (4.3%) | 3,431 (4.9%) | 440 (3.3%) | 18,185 (8.3%) | 672 (7.3%) | 24,461 (7.3%) | 1,260 (4.8%) | 0.11 |
| and a second and a second at the second at t | 2,515 (5.514) | 240(4.274) | 2,132 (1.314) | 4.0 (2.2.4) | 20,205 (0.5/4) | 572(7.2.4) | 24,102 (1.2.1) | 2,200 (1.074) | 0.22 |
| Use of heparin and other low-molecular weight heparins; n | 134 (0.3%) | 5 (0.1%) | 4 (0.0%) | 1 (0.0%) | 661 (0.3%) | 19 (0.2%) | 799 (0.2%) | 025 (0.1%) | 0.03 |
| Use of NSAIDs; n (%) | 7,110 (16.3%) | 579 (16.6%) | 11.464 (16.4%) | 2,469 (18.6%) | 36,034 (16.4%) | 1,610 (17.5%) | 34,608 (16.4%) | 4,658 (17.9%) | -0.04 |
| Use of oral corticosteroids; n (%) | 5,386 (12.3%) | 378 (10.9%) | 8,380 (12.0%) | 1,364 (11.8%) | 28,350 (12.9%) | 1,209 (13.1%) | 42,116 (12.6%) | 3,151 (12.1%) | 0.02 |
| Use of bisphosphonate (United); n (%) | 762 (1.7%) | 20 (0.6%) | 631 (0.9%) | 70 (0.5%) | 6,860 (3.1%) | 185 (2.0%) | 8,253 (2.5%) | 275 (1.1%) | 0.11 |
| Use of opioids-United; n (%) | 9.929 (22.7%) | 810 (23.3%) | 14.956 (21.3%) | 2,977 (22.4%) | 46,726 (21.2%) | 1,905 (20.7%) | 71,611 (21.4%) | 5,692 (21.9%) | -0.01 |
| Use of antidepressants; n (%) | 10,234 (23.4%) | 757 (21.7%) | 14,545 (20.8%) | 3,235 (24.3%) | 51,686 (23.5%) | 2,284 (24.8%) | 76,465 (22.9%) | 6,276 (24.1%) | -0.03 |
| Use of antipsychotics; n (%) | 1,102 (2.5%) | 53 (1.5%) | 1,152 (1.6%) | 211 (1.6%) | 6,028 (2.7%) | 188 (2.0%) | 8,282 (2.5%) | 452 (1.7%) | 0.06 |
| Use of anticonvulsants; n (%) | 7,085 (16.2%) | 484 (13.9%) | 8,267 (11.8%) | 1,618 (12.2%) | 34,448 (15.7%) | 1,475 (16.0%) | 49,800 (14.9%) | 3,577 (13.8%) | 0.03 |
| Use of lithium-United; n (%) | 89 (0.2%) | 2 (0.1%) | 78 (0.1%) | 17 (0.1%) | 246 (0.1%) | 12 (0.1%) | 413 (0.1%) | 031 (0.1%) | 0.00 |
| | 4,586 (10.5%) | 347 (10.0%) | 6,362 (9.1%) | 1,350 (10.2%) | 22,806 (10.4%) | 919 (10.0%) | 33,754 (10.1%) | 2,616 (10.1%) | 0.00 |
| Use of Benzos-United; n (%) | 2,481 (5.7%) | 222 (6.4%) | 3,970 (5.7%) | 858 (6.5%) | 11,456 (5.2%) | 516 (5.6%) | 17,907 (5.4%) | 1,396 (6.1%) | -0.03 |
| Use of anxiolytics/hypnotics-United; n (%) | 2,481 (5.7%)<br>832 (1.9%) | 13 (0.4%) | 3,970 (5.7%)<br>726 (1.0%) | 838 (6.3%)<br>30 (0.2%) | 11,436 (5.2%)<br>8,953 (4.1%) | 162 (1.8%) | 17,907 (5.4%) | 1,396 (6.1%)<br>205 (0.8%) | -0.03<br>0.17 |
| Use of dementia meds-United; n (%)<br>Use of antiparkinsonian meds-United; n (%) | 832 (1.9%)<br>962 (2.2%) | 49 (1.4%) | 1,279 (1.8%) | 235 (1.8%) | 6,237 (2.8%) | 267 (2.9%) | 10,513 (3.1%)<br>8,478 (2.5%) | | 0.17 |
| | 2 (0.0%) | 1 (0.0%) | | | 0,23/ (2.076) | 207 (2.370) | 0,470 (2.378) | 551 (2.1%) | 0.03 |
| Any use of praminitide; n (%) | 0 (0.0%) | 0 (0.0%) | 6 (0.0%)<br>6 (0.0%) | 11 (0.1%) | 20 (0.0%) | 0 (0.0%) | 026 (0.0%) | 000 (0.0%) | 0.00 |
| Any use of 1st generation sulfonylureas; n (%) | | | | 0 (0.0%) | | | | , , | |
| Entresto (sacubitril/valsartan); n (%) | 78 (0.2%) | 3 (0.1%) | 49 (0.1%) | 1 (0.0%) | 109 (0.0%) | 12 (0.1%) | 236 (0.1%) | 016 (0.1%) | 0.00 |
| Initiation as monotherapy v4 Copy; n (%) | 35,682 (81.6%) | 3,155 (90.6%) | 56,616 (80.8%) | 11,790 (88.7%) | 198,099 (90.0%) | 9,217 (100.0%) | 290,397 (87.0%) | 24,162 (93.0%) | -0.20 |
| | an ann ion of the | a none (on oth) | a man in whit | men in with | m. ** | andr. | 113,797 | 16,773 | |
| Lab values- HbA1c (%) v3; n (%) | 18,338 (42.0%) | 1,391 (40.0%) | 4,710 (6.7%) | 861 (6.5%) | N/A | N/A | 23,048 (20.3%) | 2,252 (13.4%) | 0.19<br>0.16 |
| Lab values- HbA1c (%) (within 3 months) v3; n (%) | 14,895 (34.1%) | 1,138 (32.7%) | 3,877 (5.5%) | 703 (5.3%) | N/A | N/A | 18,772 (16.5%) | 1,841 (11.0%) | 0.16 |

| Lab values- HbA1c (%) (within 6 months) v3; n (%) | 18,338 (42.0%) | 1,391 (40.0%) | 4,710 (6.7%) | 861 (6.5%) | N/A | N/A | 23,048 (20.3%) | 2,252 (13.4%) | 0.19 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values- BNP; n (%) | 353 (0.8%) | 8 (0.2%) | 62 (0.1%) | 4 (0.0%) | N/A | N/A | 413 (0.4%) | 012 (0.1%) | 0.06 |
| Lab values- BNP (within 3 months); n (%) | 218 (0.5%) | 7 (0.2%) | 40 (0.1%) | 4 (0.0%) | N/A | N/A | 258 (0.2%) | 011 (0.1%) | 0.03 |
| Lab values- BNP (within 6 months); n (%) | 353 (0.8%) | 8 (0.2%) | 62 (0.1%) | 4 (0.0%) | N/A | N/A | 415 (0.4%) | 012 (0.1%) | 0.06 |
| Lab values- BUN (mg/di); n (%) | 18,021 (41.2%) | 1,412 (40.6%) | 4,595 (6.6%) | 804 (6.0%) | N/A | N/A | 22,616 (19.9%) | 2,216 (13.2%) | 0.18 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 14,331 (32.8%) | 1,123 (32.3%) | 3,628 (5.2%) | 628 (4.7%) | N/A | N/A | 17,959 (15.8%) | 1,751 (10.4%) | 0.16 |
| | | | | , , | | N/A | - 1 | | |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 18,021 (41.2%) | 1,412 (40.6%) | 4,595 (6.6%) | 804 (6.0%) | N/A | | 22,616 (19.9%) | 2,216 (13.2%) | 0.18 |
| Lab values- Creatinine (mg/dl) v2; n (%) | 18,551 (42.4%) | 1,450 (41.7%) | 4,918 (7.0%) | 857 (6.4%) | N/A | N/A | 23,469 (20.6%) | 2,307 (13.8%) | 0.18 |
| Lab values- Creatinine (mg/dl) (within 3 months) v2; n (%) | 14,772 (33.8%) | 1,156 (33.2%) | 3,902 (5.6%) | 672 (5.1%) | N/A | N/A | 18,674 (16.4%) | 1,828 (10.9%) | 0.16 |
| totales and in the fall total and a second and the | 18,551 (42,4%) | 1,450 (41.7%) | a numbra of the | 857 (6.4%) | **** | N/A | 22 450 (20 5%) | 2 222 (42 281 | 0.18 |
| Lab values- Creatinine (mg/dl) (within 6 months) v2; n (%) | | | 4,918 (7.0%) | , , | N/A | | 23,469 (20.6%) | 2,307 (13.8%) | |
| Lab values- HDL level (mg/dl); n (%) | 15,811 (36.2%) | 1,242 (35.7%) | 4,322 (6.2%) | 822 (6.2%) | N/A | N/A | 20,133 (17.7%) | 2,064 (12.3%) | 0.15 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 12,021 (27.5%) | 941 (27.0%) | 3,317 (4.7%) | 615 (4.6%) | N/A | N/A | 15,338 (13.5%) | 1,556 (9.3%) | 0.13 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 15,811 (36.2%) | 1,242 (35.7%) | 4,322 (6.2%) | 822 (6.2%) | N/A | N/A | 20,133 (17.7%) | 2,064 (12.3%) | 0.15 |
| Lab values- LDL level (mg/dl) v2; n (%) | 16,269 (37.2%) | 1,262 (36.3%) | 4,427 (6.3%) | 797 (6.0%) | N/A | N/A | 20,696 (18.2%) | 2,059 (12.3%) | 0.16 |
| 22 13 13 23 23 14 | 20,200 (37.274) | 2,202 (30.374) | 4,427 (0.274) | 757 (0.074) | · · | | 20,000 (20.20) | 2,000 (22,000) | 0.20 |
| Lab values- LDL level (mg/dl) (within 3 months) v2; n (%) | 12,390 (28.3%) | 955 (27.4%) | 3,400 (4.9%) | 599 (4.5%) | N/A | N/A | 15,790 (13.9%) | 1,554 (9.3%) | 0.14 |
| Lab values controls (mg/di) (within 3 months) vz., ii (/a) | 12,390 (28.3/6) | 933 (27.474) | 3,400 [4.3/6] | J55 (4.5.4) | N/A | IN/A | 15,790 [13.976] | 1,334 (5.376) | 0.14 |
| Lab values-LDL level (mg/dl) (within 6 months) v2; n (%) | 16,269 (37.2%) | 1,262 (36.3%) | 4,427 (6.3%) | 797 (6.0%) | N/A | N/A | 20,696 (18.2%) | 2,059 (12.3%) | 0.16 |
| Lab values- NT-proBNP; n (%) | 46 (0.1%) | 5 (0.1%) | 12 (0.0%) | 1 (0.0%) | N/A | N/A | 58 (0.1%) | 6 (0.0%) | 0.04 |
| Lab values- NT-proBNP (within 3 months); n (%) | 26 (0.1%) | 3 (0.1%) | 8 (0.0%) | 0 (0.0%) | N/A | N/A | 34 (0.0%) | 3 (0.0%) | - |
| Lab values- NT-proBNP (within 6 months); n (%) | 46 (0.1%) | 5 (0.1%) | 12 (0.0%) | 1 (0.0%) | N/A | N/A | 58 (0.1%) | 6 (0.0%) | |
| Lab values-Total cholesterol (mg/dl) v2; n (%) | 16,044 (36.7%) | 1,274 (36.6%) | 4,327 (6.2%) | 827 (6.2%) | N/A | N/A | 20,371 (17.9%) | 2,101 (12.5%) | 0.15 |
| Lab values-Total cholesterol (mg/dl) (within 3 months) v2; | 12,207 (27.9%) | 964 (27.7%) | 3,321 (4.7%) | 619 (4.7%) | N/A | N/A | 15,528 (13.6%) | 1,583 (9.4%) | 0.13 |
| Lab values-Total cholesterol (mg/dl) (within 6 months) v2; | 16,044 (36.7%) | 1,274 (36.6%) | 4,327 (6.2%) | 827 (6.2%) | N/A | N/A | 20,371 (17.9%) | 2,101 (12.5%) | 0.15 |
| | | | | | N/A | N/A | | | 0.15 |
| Lab values-Triglyceride level (mg/d1); n (%) | 15,910 (36.4%) | 1,273 (36.6%) | 4,281 (6.1%) | 812 (6.1%) | NA | NYA | 20,191 (17.7%) | 2,085 (12.4%) | 0.13 |
| Lab values-Triglyceride level (mg/dl) (within 3 months); n (: | 12,111 (27.7%) | 965 (27.7%) | 3,287 (4.7%) | 609 (4.6%) | N/A | N/A | 15,398 (13.5%) | 1,574 (9.4%) | 0.13 |
| Lab values-Triglyceride level (mg/dl) (within 6 months); n (: | 15,910 (36.4%) | 1,273 (36.6%) | 4,281 (6.1%) | 812 (6.1%) | N/A | N/A | 20,191 (17.7%) | 2,085 (12,4%) | 0.15 |
| | | | | | - | | | | |
| Lab result number- HbA1c (%) mean (only 2 to 20 included | 40.335 | 4.707 | 4.628 | 854 | N/A | N/A | 22.863 | 2 222 | |
| | 18,235 | 1,383 | 4 | | _ | | , | 2,237 | |
| mean (sd) | 8.35 (1.78) | 8.60 (1.74) | 8.43 (1.87) | 8.50 (1.80) | N/A | N/A | 8.37 (1.80) | 8.56 (1.76) | -0.11 |
| median (IQR) | 8.00 [7.10, 9.20] | 8.20 [7.40, 9.50] | 8.00 [7.10, 9.30] | 8.00 [7.10, 9.55] | N/A | N/A | 8.00 (1.80) | 8.12 (1.76) | -0.07 |
| Missing; n (%) | 25,475 (58.3%) | 2,098 (60.3%) | 65,459 (93.4%) | 12,438 (93.6%) | N/A | N/A | 90,934 (79.9%) | 14,536 (86.7%) | -0.18 |
| Lab result number- BNP mean v2 | 353 | 2,050 (00.5.4) | 62 | 22,130 (33.034) | N/A | N/A | 415 | 12 | 0.20 |
| | | • | | | | | | | |
| mean (sd) | 154.08 (373.54) | 62.94 (82.60) | 526.58 (2,180.80) | 25.75 (28.92) | N/A | N/A | 209.73 (907.39) | 50.54 (74.74) | 0.25 |
| median [IQR] | 65.40 [27.20, 164.00] | 13.10 [1.23, 159.75] | 71.00 [26.75, 193.75] | 20.00 [1.50, 55.75] | N/A | N/A | #VALUE! | 15.40 (74.74) | #VALUE! |
| Missing; n (%) | 43,357 (99.2%) | 3,473 (99.8%) | 70,025 (99.9%) | 13,288 (100.0%) | N/A | N/A | 113,382 (99.6%) | 16,761 (99.9%) | -0.06 |
| | 18 021 | 1.412 | 4.595 | 13,200 (200.074) | N/A | N/A | 22.616 | 2.216 | 0.00 |
| Lab result number- BUN (mg/di) mean v2 | 20,022 | | 4 | 804 | | | , | -, | |
| mean (sd) | 16.92 (6.36) | 15.66 (4.60) | 1,098.70 (12,576.94) | 221.02 (5,818.55) | N/A | N/A | 236.71 (5668.81) | 90.17 (3504.95) | 0.03 |
| median [IQR] | 16.00 [13.00, 20.00] | 15.00 [12.50, 18.00] | 15.67 [13.00, 19.00] | 15.00 [13.00, 18.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing n (%) | 25,689 (58.8%) | 2,069 (59.4%) | 65,492 (93.4%) | 12,488 (94.0%) | N/A | N/A | 91,181 (80.1%) | 14,557 (86.8%) | -0.18 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 to 15 | 18.407 | 1,444 | 4,354 | 725 | N/A | N/A | 22,761 | 2.169 | |
| | 0.95 (0.27) | 0.88 (0.19) | 0.95 (0.25) | 0.90 (0.20) | N/A | N/A | 0.95 (0.27) | 0.89 (0.19) | 0.26 |
| mean (sd) | | | | | | | | | |
| median [IQR] | 0.91 [0.77, 1.08] | 0.88 [0.74, 1.00] | 0.92 [0.78, 1.05] | 0.90 [0.77, 1.00] | N/A | N/A | 0.91 (0.27) | 0.89 (0.19) | 0.09 |
| Missing; n (%) | 25,303 (57.9%) | 2,037 (58.5%) | 65,733 (93.8%) | 12,567 (94.5%) | N/A | N/A | 91,036 (80.0%) | 14,604 (87.1%) | -0.19 |
| Lab result number- HDL level (mg/dl) mean (only =:5000 in | 15.811 | 1.242 | 4,292 | 822 | N/A | N/A | 20.103 | 2.064 | |
| mean (sd) | 45.18 (13.27) | 43.30 (12.25) | 45.19 (45.80) | 43.92 (12.86) | N/A | N/A | 45.18 (24.21) | 43.55 (12.50) | 0.08 |
| | | | · · · | , , | | | \ <i>\</i> | | |
| median [IQR] | 43.00 [36.00, 52.00] | 41.50 [35.00, 50.25] | 43.00 [36.00, 52.00] | 42.00 [35.00, 51.00] | N/A | N/A | 43.00 (24.21) | 41.70 (12.50) | 0.07 |
| Missing; n (%) | 27,899 (63.8%) | 2,239 (64.3%) | 65,795 (93.9%) | 12,470 (93.8%) | N/A | N/A | 93,694 (82.3%) | 14,709 (87.7%) | -0.15 |
| | | | • | • | | | | - | |
| Lab result number- LDL level (mg/dl) mean (only = 5000 in | 15,877 | 1,250 | 3,990 | 713 | N/A | N/A | 19,867 | 1,963 | |
| mean (sd) | 86.40 (40.73) | 81.75 (39.30) | 89.57 (42.63) | 88.81 (43.09) | N/A | N/A | 87.04 (41.12) | 84.31 (40.73) | 0.07 |
| | | | | 87.00 (62.50, 112.50) | | | | | 0.01 |
| median (IQR) | 84.00 [62.00, 110.00] | 83.00 [60.00, 105.00] | 88.00 [64.00, 114.12] | | N/A | N/A | 84.80 (41.12) | 84.45 (40.73) | |
| Missing: n (%) | 27,833 (63.7%) | 2,231 (64.1%) | 66,097 (94.3%) | 12,579 (94.6%) | N/A | N/A | 93,930 (82.5%) | 14,810 (88.3%) | -0.16 |
| Lab result number-Total cholesterol (mg/dl) mean (only=c | 16,029 | 1,274 | 4,296 | 827 | N/A | N/A | 20,325 | 2,101 | |
| mean (sd) | 173.66 (47.24) | 172.86 (43.86) | 176.94 (50.12) | 176.61 (49.24) | N/A | N/A | 174.35 (47.86) | 174.34 (46.06) | 0.00 |
| median [IQR] | 167.00 [142.00, 198.50] | 168.00 [143.00, 195.00] | 172.45 [146.50, 204.00] | 170.00 [143.00, 203.00] | N/A | N/A | 168.15 (47.86) | 168.79 (46.06) | -0.01 |
| | | | | | | | , , | \ | -0.01 |
| Missing: n (%) | 27,681 (63.3%) | 2,207 (63.4%) | 65,791 (93.9%) | 12,465 (93.8%) | N/A | N/A | 93,472 (82.1%) | 14,672 (87.5%) | -0.13 |

| Les contactue—Triggerielate (my fill prime (my see ) 1.50 (1.50 ( | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Mailing (P) | | , | 1,273 | 4-1- | | N/A | N/A | 20,157 | -, | |
| Martin M | | | | | | | | , , , | | |
| Las mate number—remogation mane (only 40 included) 13.15.65 13.15.15.15.15.15.15.15.15.15.15.15.15.15. | | | | | | | | | | |
| | Missing n (%) | 27,802 (63.6%) | 2,208 (63.4%) | 65,838 (93.9%) | 12,480 (93.9%) | N/A | N/A | 93,640 (82.3%) | 14,688 (87.6%) | -0.15 |
| | Lab conditionable. Here and objection many facility of included | 43.004 | 040 | 3 300 | | N/A | N/A | 45 400 | 4.474 | |
| | | | | | | | | | | 0.05 |
| Maring Ph | | | | | | | | | | |
| Lat must furnise - function mane (poly y 90 and x 11 33 1,279 34 1,279 34 | | | | | | | | | | |
| | | 30,303 (70.774) | 2,363 (73.676) | 00,030(33.23) | 22,733 [33.079] | nya. | 140 | 37,007 (03.078) | 23,302 (32.270) | 0.27 |
| | Lab result number- Serum sodium mean (only > 90 and < 15 | 18,022 | 1,415 | 4,636 | 852 | N/A | N/A | 22,658 | 2,267 | |
| 1800 | | 139.31 (2.76) | 139.24 (2.48) | 138.90 (2.60) | 138.79 (2.34) | N/A | N/A | 139.23 (2.73) | 139.07 (2.43) | 0.06 |
| Let most incomer - Naturation mass (only-) of ord crit ordinot. 1.43 | | 139.50 [138.00, 141.00] | 139.00 [138.00, 141.00] | 139.00 [137.00, 141.00] | 139.00 [137.00, 140.00] | N/A | N/A | 139.40 (2.73) | 139.00 (2.43) | 0.15 |
| Let most incomer - Naturation mass (only-) of ord crit ordinot. 1.43 | Missing; n (%) | 25,688 (58.8%) | 2,066 (59.4%) | 65,451 (93.4%) | 12,440 (93.6%) | N/A | N/A | 91,139 (80.1%) | 14,506 (86.5%) | -0.17 |
| Mare | | | | | | | | | | |
| Maring (Fig) 4.39 (4.10) | | | | | | | | | | |
| Lab result number—Glucose Passing or random mean (mit) 1.0.2 | | | | | | | - | | | |
| Liber Preside number—Glucose (halling or random) memi (only)mem (orl)1.1.1.1.1.1.1.1.1.1.1.1.1.1.1.1.1.1 | | | | | | | | | | |
| | Missing n (%) | 26,759 (61.2%) | 2,136 (61.4%) | 66,140 (94.4%) | 12,561 (94.5%) | N/A | N/A | 92,899 (81.6%) | 14,697 (87.6%) | -0.17 |
| | Laboration and a Classical States and a laboration and a | 40.000 | | 4.777 | | 21/2 | n/a | 22.700 | | |
| | | | | | | | | | | 0.03 |
| Maintage Ph | | \ / | \ <i>\</i> | \ <i>\</i> | \ <i>\</i> | | | \ / | \ <i>\</i> | |
| Lib result number - Potassium mean [coty 1-7 included]mean [st]mean [st]mean [st]de [cot]de [c | | | | | | | | , , | | |
| mesimp(IQT) | <del></del> | ,, | 4 | | | | | | | |
| meni [pt] | Lab result number- Potassium mean (only 1-7 included) | 18,422 | 1,437 | 4,485 | 779 | N/A | N/A | 22,907 | 2,216 | |
| Marging n No | | 4.46 (0.41) | 4.42 (0.40) | 4.34 (0.44) | 4.29 (0.42) | N/A | N/A | 4.44 (0.42) | 4.37 (0.41) | 0.17 |
| Commontify Scores Comm | median [IQR] | 4.45 [4.20, 4.70] | 4.40 [4.20, 4.70] | 4.30 [4.00, 4.60] | 4.30 [4.00, 4.50] | N/A | N/A | 4.42 (0.42) | 4.36 (0.41) | 0.14 |
| CC Lid osph-(CD9 and ICD10 V2 men [pd] 2.24 [1.70] 1.70 [1.28] 1.36 [1.30] 1.52 [1.10] 2.28 [1.64] 2.10 [1.41] 2.13 [1.58] 1.75 [1.24] 0.31 men [pd] 2.00 [1.00, 3.00] 1.00 [1.00, 2.00] 1.00 [1.00, 2.00] 1.00 [1.00, 2.00] 2.00 [1.00, 3.00] 1.79 [1.38] 1.33 [1.24] 0.31 men [pd] 2.30 [1.00, 3.00] 1.00 [1.00, 2.00] 1.00 [1.00, 2.00] 2.00 [1.00, 3.00] 1.79 [1.38] 1.33 [1.24] 0.31 men [pd] 1.30 [1.30] 1.3 | Missing: n (%) | 25,288 (57.9%) | 2,044 (58.7%) | 65,602 (93.6%) | 12,513 (94.1%) | N/A | N/A | 90,890 (79.9%) | 14,557 (86.8%) | -0.19 |
| menip | | | | | | | | | | |
| -menip(pt) 2.00 [1.00, 3.00] 1.00 [1.00, 2.00] 1.00 [1.00, 2.00] 1.00 [1.00, 2.00] 2.00 [1.00, 3.00] 2.00 [1.00, 3.00] 1.79 [1.58] 1.33 [1.24] 0.33 Fraity Score: Qualitative Version 363 days as Categories, v1 | | | | | | | | | | |
| Pailty Some Qualitative Version 360 days as Categories, v.1 Or. [N] | | | | | | | | | | |
| or. [6] | median [IQR] | 2.00 [1.00, 3.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 1.79 (1.58) | 1.35 (1.24) | 0.31 |
| or. [6] | Series Series Series in Maria 258 de la Series Series de | | | | | | | | | |
| to 2: n Ph | | 22.256/52.28() | 4 003/53 5%) | 25 200/50 5%) | 7 024 (50 0%) | 02 540 (42 5%) | 5 C77 (C4 5%) | 152 174 (45 6%) | 15 300 (50 191) | -0.27 |
| -3 or more n (%) 6,590 (16.0%) 337 (11.4%) 9,323 (13.6%) 1.133 (8.7%) 51.617 (23.5%) 1.60 (12.6%) 68,130 (20.4%) 2.710 (10.4%) 0.28 Prailty Score Empirical Version 363 days as Categories, v3 | | | | | | | | | | |
| Prinity Score: Empirical Version 365 days, as: Categories, v3 | | | | | | | | | | |
| 0.12908; n/h) 11,507 (26.6 h) 1220 (31.0 h) 22,110 (31.5 h) 4,747 (31.7 h) 31,18 (16.0 h) 1811 (19.6 h) 68,907 (20.6 h) 7,778 (29.9 h) 0.22 (31.0 h) 13,002 (30.9 h) 12,007 (30.9 h) 12,007 (30.6 h) 23,005 (31.5 h) 4,844 (36.6 h) 64,307 (29.3 h) 10,194 (30.4 h) 9,103 (31.5 h) 0.12 (31.5 h) 0.1 | | 0,550 (20.0.4) | 227 (22777) | 2,525(25.0.4) | 2,222 (2.77) | 32,027 (23.574) | 2,200 (22.0.0) | 20,230 (20,111) | 2,720 (20.779) | 5.25 |
| 0.12908; n/h) 11,507 (26.6 h) 1220 (31.0 h) 22,110 (31.5 h) 4,747 (31.7 h) 31,18 (16.0 h) 1811 (19.6 h) 68,907 (20.6 h) 7,778 (29.9 h) 0.22 (31.0 h) 13,002 (30.9 h) 12,007 (30.9 h) 12,007 (30.6 h) 23,005 (31.5 h) 4,844 (36.6 h) 64,307 (29.3 h) 10,194 (30.4 h) 9,103 (31.5 h) 0.12 (31.5 h) 0.1 | Frailty Score: Empirical Version 365 days as Categories, v3 | | | | | | | | | |
| 0 1.523167; n [%] 13,02 [30.5%] 1,260 [36.2%] 23,355 [38.5%] 4,834 [36.4%] 64,373 [29.5%] 10,1594 [30.4%] 9,130 [35.1%] 0.10 | | 11,607 (26.6%) | 1,220 (35.0%) | 22,110 (31.5%) | 4,747 (35.7%) | 35,188 (16.0%) | 1,811 (19.6%) | 68,905 (20.6%) | 7,778 (29.9%) | -0.22 |
| Non-Frailty; (n / h) | | 13,502 (30.9%) | 1,260 (36.2%) | 23,555 (33.6%) | 4,834 (36.4%) | 64,537 (29.3%) | 3,036 (32.9%) | 101,594 (30.4%) | 9,130 (35.1%) | -0.10 |
| Prailty Score (mean): Qualitative Version 365 days, v1mean [xt]mean [xt] | >=0.1631167; n (%) | 18,601 (42.6%) | 1,001 (28.8%) | 24,422 (34.8%) | 3,711 (27.9%) | 120,336 (54.7%) | 4,370 (47.4%) | 163,359 (48.9%) | 9,082 (34.9%) | 0.29 |
| mean [cd] | Non-Frailty; n (%) | 24,902 (57.0%) | 1,839 (52.8%) | 36,675 (52.3%) | 6,921 (52.1%) | 10,548 (4.8%) | 381 (4.1%) | 72,125 (21.6%) | 9,141 (35.2%) | -0.31 |
| mean [cd] | | | | | | | | | | |
| median (iQR) | | | | | | | | | | |
| Fraity Score [mean]: Empirical Version 365 days, v2mean [x5]mean [x5]median [DQR]median [DQR] | | | | | | | | | | |
| mesin [23] 0.17 [0.05] 0.15 [0.04] 0.15 [0.04] 0.14 [0.04] 0.14 [0.04] 0.18 [0.06] 0.17 [0.05] 0.17 [0.06] 0.15 [0.04] 0.39 merian [DR] 0.15 [0.13, 0.19] 0.14 [0.12, 0.17] 0.14 [0.12, 0.17] 0.14 [0.12, 0.16] 0.17 [0.14, 0.21] 0.16 [0.13, 0.19] 0.16 [0.06] 0.17 [0.04] 0.20 Healthcare Utilization Any hospitalization within prior 30 days; n [%] 3,020 [6.9%] 138 [4.0%] 3,300 [4.7%] 397 [3.0%] 12,377 [5.6%] 313 [3.4%] 18,697 [5.6%] 848 [3.3%] 0.11 Any hospitalization within prior 30 days; n [%] 1,005 [2.3%] 23 [0.7%] 896 [1.3%] 52 [0.4%] 3,315 [1.5%] 48 [0.5%] 5,216 [1.6%] 123 [0.5%] 0.11 Any hospitalization during prior 31-180 days; n [%] 2,160 [4.9%] 17 [3.4%] 2,481 [3.5%] 312 [2.6%] 9,435 [4.3%] 273 [3.0%] 14,097 [4.2%] 741 [2.9%] 0.05 Endocrinologist Visit; n [%] 3,435 [1.0%] 719 [20.7%] 6,290 [9.0%] 2,264 [17.0%] 23,625 [10.7%] 1,457 [13.8%] 34,280 [10.3%] 34,280 | | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.66 (1.80) | 0.00 (1.31) | 0.42 |
| median (ICR) | | 0.47(0.00) | n and in nat | n an in nat | n a a local | a sala cel | 0.47 (0.05) | n and need | 0.48 (0.04) | 0.35 |
| Healthcare Utilization Any hospitalization; n (%) Any hospitalization within prior 30 days; n (%) 1,005 (2.3%) 1,005 (2.3% | | | | | | | | | | |
| Any hospitalization; n (%) 3,020 (6.9%) 138 (4.0%) 3,300 (4.7%) 397 (3.0%) 12,377 (5.6%) 313 (3.4%) 18,697 (5.6%) 848 (3.3%) 0.11 Any hospitalization within prior 30 days; n (%) 1,005 (2.3%) 23 (0.7%) 896 (1.3%) 52 (0.4%) 3,315 (1.5%) 48 (0.5%) 5,216 (1.6%) 123 (0.5%) 0.11 Any hospitalization during prior 31-180 days; n (%) 2,160 (4.9%) 117 (3.4%) 2,481 (3.5%) 351 (2.6%) 9,456 (4.3%) 273 (3.0%) 14,077 (4.2%) 741 (2.0%) 742 (2.0%) 742 (2.0%) 742 (2.0%) 742 (2.0%) 743 | | 0.15 (0.15, 0.15) | 0.14[0.11, 0.17] | 0.14 [0.11, 0.17] | 0.14(0.11, 0.10) | 0.17 (0.14, 0.11) | 0.10 [0.13, 0.13] | 0.10 (0.00) | 0.25(0.04) | 0.20 |
| Any hospitalization within prior 30 days; n (%) 1,005 (2.3%) 23 (0.7%) 896 (1.3%) 52 (0.4%) 3,313 (1.5%) 48 (0.5%) 5,216 (1.6%) 123 (0.5%) 0.11 Any hospitalization during prior 31-180 days; n (%) 2,160 (4.9%) 117 (3.4%) 2,481 (3.5%) 351 (2.6%) 9,456 (4.3%) 273 (3.0%) 14,097 (4.2%) 741 (2.9%) 0.07 Bridgerinologist Visit; n (%) 4,365 (10.0%) 719 (20.7%) 6,290 (9.0%) 2,264 (17.0%) 23,625 (10.7%) 1,457 (13.8%) 34,280 (10.3%) 4,440 (17.1%) 0.20 Bridgerinologist Visit; (30 days prior); n (%) 2,851 (6.5%) 548 (13.7%) 4,089 (3.8%) 1,488 (11.2%) 15,666 (7.6%) 970 (10.5%) 22,374 (6.7%) 3,271 (12.0%) 0.17 Internal medicine/hamily medicine visits; n (%) 33,818 (77.4%) 2,030 (58.3%) 61,331 (87.8%) 11,642 (87.6%) 178,740 (81.2%) 7,344 (79.7%) 274,089 (82.1%) 21,016 (80.9%) 0.03 Internal medicine/hamily medicine visits; (31 to 180 days prior) v2; 25,331 (58.0%) 1,697 (48.8%) 49,865 (71.1%) 9,603 (72.2%) 132,425 (69.8%) 230,967 (69.2%) 17,733 (68.2%) 0.02 Condiologist visit; n (%) 13,109 (30.0%) 740 (21.3%) 14,339 (20.5%) 2,488 (18.7%) 62,166 (28.2%) 2,290 (24.8%) 89,614 (26.8%) 5,518 (21.8%) 5,518 (21.2%) 5,518 (2 | | 3.020 (6.9%) | 138 (4.0%) | 3.300 (4.7%) | 397 (3.0%) | 12,377 (5.6%) | 313 (3.4%) | 18,697 (5.6%) | 848 (3.3%) | 0.11 |
| Any hospitalization during prior 31-180 days; n (%) 2,160 (4.9%) 117 (3.4%) 2,481 (3.5%) 331 (2.6%) 9,436 (4.3%) 273 (3.0%) 14,097 (4.2%) 741 (2.9%) 0.07 Bodocrinologist Visit; n (%) 4,365 (10.0%) 719 (20.7%) 6,290 (9.0%) 2,264 (17.0%) 23,625 (10.7%) 1,457 (13.8%) 34,280 (10.3%) 4,440 (17.1%) 0.20 Bodocrinologist Visit (30 days prior); n (%) 2,869 (6.6%) 348 (13.7%) 4,287 (6.0%) 1,733 (13.2%) 15,268 (6.9%) 970 (10.5%) 22,374 (6.7%) 3,271 (12.6%) 0.20 Bodocrinologist Visit (31 to 180 days prior); n (%) 2,851 (6.5%) 505 (14.5%) 4,089 (3.8%) 1,488 (11.2%) 16,666 (7.6%) 1,117 (12.1%) 23,606 (7.1%) 3,110 (12.0%) 0.17 Internal medicine/hamily medicine visits; n (%) 33,818 (77.4%) 2,030 (88.3%) 61,331 (87.8%) 11,642 (87.6%) 178,740 (81.2%) 7,344 (79.7%) 274,089 (82.1%) 21,016 (80.9%) 0.03 Internal medicine/hamily medicine visits (30 days prior) v2; 25,331 (58.0%) 1,353 (38.9%) 46,643 (66.6%) 8,792 (66.1%) 129,466 (58.8%) 5,186 (56.3%) 201,440 (60.3%) 15,331 (59.0%) 0.03 Internal medicine/hamily medicine visits (31 to 180 days prior) v2; 25,331 (58.0%) 1,697 (48.8%) 49,865 (71.1%) 9,603 (72.2%) 152,425 (69.3%) 6,433 (69.8%) 230,967 (69.2%) 17,733 (68.2%) 0.02 Cardiologist visit; n (%) 13,109 (30.0%) 740 (21.3%) 14,339 (20.3%) 2,488 (18.7%) 62,166 (28.2%) 2,290 (24.8%) 89,614 (26.8%) 5,518 (21.2%) 0.13 | | | | - 1 | | | | - 1 | | |
| Endocrinologist Visit; n (%) 4,365 (10.0%) 719 (20.7%) 6,290 (9.0%) 2,264 (17.0%) 23,625 (10.7%) 1,457 (13.8%) 34,280 (10.3%) 4,440 (17.1%) -0.20 Endocrinologist Visit (30 days prior); n (%) Endocrinologist Visit (31 to 180 days prior); n (%) 2,869 (6.6%) 3,271 (12.6%) 3,110 (12.0%) 3,110 ( | | | | | | | | | | |
| Endocrinologist Visit (30 days prior); n (%) 2,869 (6.6%) 348 (15.7%) 4,237 (6.0%) 1,733 (13.2%) 15,268 (6.9%) 970 (10.5%) 22,374 (6.7%) 3,271 (12.6%) -0.20 Endocrinologist Visit (31 to 180 days prior); n (%) 2,851 (6.5%) 305 (14.5%) 305 (14.5%) 4,089 (5.8%) 1,488 (11.2%) 16,666 (7.6%) 1,117 (12.1%) 23,606 (7.1%) 33,818 (77.4%) 2,030 (58.3%) 61,531 (87.8%) 11,642 (87.6%) 178,740 (81.2%) 7,344 (79.7%) 274,089 (82.1%) 21,016 (80.9%) 0.03 Internal medicine/family medicine visits (30 days prior) v2; 25,331 (38.0%) 1,333 (38.9%) 46,643 (66.6%) 8,792 (66.1%) 129,466 (38.8%) 5,186 (56.3%) 201,440 (60.3%) 13,331 (39.0%) 0.03 Internal medicine/family medicine visits (31 to 180 days prior) v2; 28,677 (65.6%) 1,697 (48.8%) 49,865 (71.1%) 9,603 (72.2%) 152,425 (69.3%) 6,433 (69.8%) 230,967 (69.2%) 3,518 (21.2%) 0.03 | | | | | | | | | | |
| Endocrinologist Visit (31 to 180 days prior); n (%) 2,851 (6.5%) 505 (14.5%) 4,089 (5.8%) 1,488 (11.2%) 16,666 (7.6%) 178,740 (81.2%) 7,344 (79.7%) 274,089 (82.1%) 21,016 (80.9%) 0.03 Internal medicine/family medicine visits (30 days prior) v2; 25,331 (38.0%) 1,353 (38.9%) 46,643 (66.6%) 8,792 (66.1%) 129,466 (38.8%) 5,186 (56.3%) 201,440 (60.3%) 15,331 (59.0%) 0.03 Internal medicine/family medicine visits (31 to 180 days prior) v2; 28,677 (65.6%) 1,697 (48.8%) 49,865 (71.1%) 9,603 (72.2%) 13,425 (69.3%) 62,166 (28.2%) 2,290 (24.8%) 89,614 (26.8%) 5,188 (26.8%) 5,181 (26.8%) 17,733 (68.2%) 0.02 Cardiologist visit; n (%) | | | 548 (15.7%) | 4,237 (6.0%) | | | | | 3,271 (12.6%) | -0.20 |
| Internal medicine/family medicine visits [31 days prior] v2; 25,331 [38.0%] 1,333 [38.9%] 46,643 [66.6%] 8,792 [66.1%] 129,466 [38.8%] 5,186 [36.3%] 201,440 [60.3%] 15,331 [39.0%] 0.03 Internal medicine/family medicine visits [31 to 180 days pr 28,677 [65.6%] 1,697 [48.8%] 49,865 [71.1%] 9,603 [72.2%] 132,425 [69.3%] 6,433 [69.8%] 230,967 [69.2%] 17,733 [68.2%] 0.02 Cardiologist visit; n [%] 13,109 [30.0%] 740 [21.3%] 14,339 [20.3%] 2,488 [18.7%] 62,166 [28.2%] 2,290 [24.8%] 89,614 [26.8%] 5,518 [21.2%] 0.13 | | | 505 (14.5%) | | | 16,666 (7.6%) | | | | -0.17 |
| Internal medicine/family medicine visits [31 days prior] v2; 25,331 [38.0%] 1,333 [38.9%] 46,643 [66.6%] 8,792 [66.1%] 129,466 [38.8%] 5,186 [36.3%] 201,440 [60.3%] 15,331 [39.0%] 0.03 Internal medicine/family medicine visits [31 to 180 days pr 28,677 [65.6%] 1,697 [48.8%] 49,865 [71.1%] 9,603 [72.2%] 132,425 [69.3%] 6,433 [69.8%] 230,967 [69.2%] 17,733 [68.2%] 0.02 Cardiologist visit; n [%] 13,109 [30.0%] 740 [21.3%] 14,339 [20.3%] 2,488 [18.7%] 62,166 [28.2%] 2,290 [24.8%] 89,614 [26.8%] 5,518 [21.2%] 0.13 | Internal medicine/family medicine visits; n (%) | 33,818 (77.4%) | 2,030 (58.3%) | 61,531 (87.8%) | 11,642 (87.6%) | 178,740 (81.2%) | 7,344 (79.7%) | 274,089 (82.1%) | 21,016 (80.9%) | 0.03 |
| Internal medicine/family medicine visits (31 to 180 days pr 28,677 (65.6%) 1,697 (48.8%) 49,865 (71.1%) 9,603 (72.2%) 152,425 (69.3%) 6,433 (69.8%) 230,967 (69.2%) 17,733 (68.2%) 0.02 Cardiologist visit; n (%) 13,109 (30.0%) 740 (21.3%) 14,339 (20.5%) 2,488 (18.7%) 62,166 (28.2%) 2,290 (24.8%) 89,614 (26.8%) 5,518 (21.2%) 0.13 | | | | | | | | | | |
| Cardiologist visit n (%) ' 13,109 (30.0%) 740 (21.3%) 14,339 (20.5%) 2,488 (18.7%) 62,166 (28.2%) 2,290 (24.8%) 89,614 (26.8%) 5,518 (21.2%) 0.13 | Internal medicine/family medicine visits (30 days prior) v2; | 25,331 (58.0%) | 1,353 (38.9%) | 46,643 (66.6%) | 8,792 (66.1%) | 129,466 (58.8%) | 5,186 (56.3%) | 201,440 (60.3%) | 15,331 (59.0%) | 0.03 |
| Cardiologist visit n (%) ' 13,109 (30.0%) 740 (21.3%) 14,339 (20.5%) 2,488 (18.7%) 62,166 (28.2%) 2,290 (24.8%) 89,614 (26.8%) 5,518 (21.2%) 0.13 | | an emple | 4 000 (45-) | an new less select | a con for -5-1 | ann ann ler -5-1 | e annien ent | 222 222 les -5-1 | 42 222 (ca -5-1 | |
| | | | | | | | | - 1 / | | |
| 1,676 (6.476) באבונים ביוברים ומיברים ביוברים | | | | | | | | - 1 | | |
| | manner or cardiologist visits (30 days prior); it (76) | 4,705 (10.8%) | 251(7.2%) | 4,808 (6.9%) | /33 (3.3%) | 20,600 [9.4%] | 090 (7.3%) | 30,113 (9.0%) | 1,6/6 [6.4%] | 0.10 |

| Number of Cardiologist visits (31 to 180 days prior); n (%) | 11,053 (25.3%) | 622 (17.9%) | 12,065 (17.2%) | 2,109 (15.9%) | 53,433 (24.3%) | 1,998 (21.7%) | 76,551 (22.9%) | 4,729 (18.2%) | 0.12 |
|---|---|---|---|---|---|---|---|---|---|
| Bectrocardiogram v2; n (%) | 13,667 (31.3%) | 812 (23.3%) | 19,434 (27.7%) | 3,190 (24.0%) | 64,105 (29.1%) | 2,449 (26.6%) | 97,206 (29.1%) | 6,451 (24.8%) | 0.10 |
| Use of glucose test strips; n (%) | 1,583 (3.6%) | 143 (4.1%) | 2,505 (3.6%) | 523 (3.9%) | 6,748 (3.1%) | 228 (2.5%) | 10,836 (3.2%) | 894 (3.4%) | -0.01<br>#DIV/0! |
| Dielysis; n (%) | 3 (0.0%) | 1 (0.0%) | 3 (0.0%) | 0 (0.0%) | 25 (0.0%) | 0 (0.0%) | 031 (0.0%) | 001 (0.0%) | |
| Naive new user v8 Copy; n (%) | 8,086 (18.5%) | 369 (10.6%) | 12,706 (18.1%) | 1,626 (12.2%) | 31,513 (14.3%) | 879 (9.5%) | 52,305 (15.7%) | 2,874 (11.1%) | 0.14 |
| Nantidiabetic drugs at index date v3 Copy | 2 42 (0.75) | 2.24 (0.00) | 2 42 (0 22) | 2.20(0.00) | 244/025 | 2 22 (0.05) | 2 44 (0 75) | 2 20 (0 00) | -0.19 |
| mean (sd)<br>median (IOR) | 2.12 (0.75)<br>2.00 [2.00, 3.00] | 2.24 (0.89)<br>2.00 [2.00, 3.00] | 2.13 (0.72)<br>2.00 (2.00, 3.00) | 2.28 (0.86)<br>2.00 [2.00, 3.00] | 2.14 (0.76) | 2.33 (0.86)<br>2.00 [2.00, 3.00] | 2.14 (0.75)<br>2.00 (0.75) | 2.29 (0.86)<br>2.00 (0.86) | 0.19 |
| median (I/Opt) | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 (0.73) | 2.00 (0.86) | 0.00 |
| number of different/distinct medication prescriptions | | | | | | | | | |
| mean (sd) | 9.83 (4.85) | 9.60 (4.67) | 8.91 (4.34) | 9.66 (4.53) | 9.38 (4.19) | 9.76 (4.29) | 9.34 (4.31) | 9.69 (4.47) | -0.08 |
| median (IQR) | 9.00 [6.00, 12.00] | 9.00 [6.00, 12.00] | 8.00 [6.00, 11.00] | 9.00 [6.00, 12.00] | 9.00 [6.00, 12.00] | 9.00 [7.00, 12.00] | 8.79 (4.31) | 9.00 (4.47) | -0.05 |
| Number of Hospitalizations | | | | | | | | | |
| mean (sd) | 0.08 (0.33) | 0.04 (0.22) | 0.05 (0.25) | 0.03 (0.19) | 0.07 (0.30) | 0.04 (0.23) | 0.07 (0.29) | 0.03 (0.21) | 0.16 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.29) | 0.00 (0.21) | 0.00 |
| Number of hospital days | | | | | | | | | |
| mean (sd) | 0.45 (2.50) | 0.19 (1.12) | 0.28 (1.87) | 0.15 (1.13) | 0.40 (2.56) | 0.21 (1.62) | 0.38 (2.42) | 0.18(1.32) | 0.10 |
| median (IQR) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (2.42) | 0.00 (1.32) | 0.00 |
| Number of Emergency Department (ED) visits v3 | | | | | | | | | |
| mean (sd) | 0.35 (1.12) | 0.20 (0.71) | 0.10 (1.08) | 0.06 (0.65) | 0.36 (1.08) | 0.28 (0.94) | 0.30 (1.09) | 0.16 (0.77) | 0.15 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (1.09) | 0.00 (0.77) | 0.00 |
| Number of Office visits | !! | | | | | | | | |
| mean (sd)<br>median (IOR) | 4.60 (3.62)<br>4.00 [2.00, 6.00] | 4.33 (3.24)<br>3.00 (2.00, 6.00) | 4.23 (3.37)<br>3.00 (2.00, 5.00) | 4.32 (3.23)<br>4.00 (2.00, 6.00) | 4.74 (3.65)<br>4.00 (2.00, 6.00) | 4.96 (3.55)<br>4.00 (2.00, 7.00) | 4.61 (3.59) | 4.55 (3.35) | 0.02<br>-0.02 |
| median (icip)<br>Number of Endocrinologist visits | 4.00 [2.00, 6.00] | 3.00 [2.00, 6.00] | 3.00 [2.00, 5.00] | 4.00 [2.00, 6.00] | 4.00 [2.00, 6.00] | 4.00 [2.00, 7.00] | 3.79 (3.59) | 3.87 (3.35) | -0.02 |
| mean (sd) | 0.46 (2.19) | 1.21 (3.74) | 0.39 (2.06) | 0.92 (3.24) | 0.59 (2.92) | 1.02 (4.01) | 0.53 (2.67) | 0.99 (3.60) | -0.15 |
| median (IQR) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (2.67) | 0.00 (3.60) | 0.00 |
| Number of internal medicine/family medicine visits | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00] | 0.50 [0.50, 0.50] | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.55 (2.57) | 0.55 (5.55) | 0.00 |
| mean (sd) | 8.04 (11.91) | 4.73 (8.01) | 6.69 (8.43) | 6.65 (7.61) | 7.09 (9.42) | 7.18 (10.03) | 7.13 (9.59) | 6.58 (8.60) | 0.06 |
| median [IQR] | 4.00 [1.00, 10.00] | 2.00 [0.00, 6.00] | 4.00 [2.00, 9.00] | 5.00 [2.00, 9.00] | | 4.00 [1.00, 10.00] | 4.00 (9.59) | 4.24 (8.60) | -0.03 |
| Number of Cardiologist visits | | | | | | | | ` ' | |
| mean (sd) | 1.44 (3.70) | 0.97 (2.93) | 0.84 (2.68) | 0.70 (2.14) | 1.37 (3.88) | 1.14 (3.20) | 1.27 (3.64) | 0.89 (2.67) | 0.12 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 (3.64) | 0.00 (2.67) | 0.00 |
| Number electrocardiograms received v2 | | | | | | | | | |
| mean (sd) | 0.60 (1.39) | 0.36 (0.93) | 0.47 (1.10) | 0.38 (0.89) | 0.53 (1.14) | 0.46 (1.03) | 0.53 (1.17) | 0.41 (0.95) | 0.11 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (1.17) | 0.00 (0.95) | 0.00 |
| Number of HbA1c tests ordered | | | | | | | | | |
| mean (sd) | 1.24 (0.88) | 1.28 (0.85) | 1.07 (0.85) | 1.32 (0.81) | 1.40 (0.82) | 1.49 (0.81) | 1.31 (0.83) | 1.37 (0.82) | -0.07 |
| median [IQR] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 (0.83) | 1.00 (0.82) | 0.00 |
| Number of glucose tests ordered | | | | | | 0.42 (0.00) | 0.00 (0.00) | | -0.01 |
| mean (sd)<br>median (ICR) | 0.52 (3.68)<br>0.00 (0.00, 0.00) | 0.38 (0.97)<br>0.00 (0.00, 0.00) | 0.36 (1.40)<br>0.00 (0.00, 0.00) | 0.41 (1.07)<br>0.00 [0.00, 0.00] | 0.39 (0.98)<br>0.00 (0.00, 0.00) | 0.42 (0.98)<br>0.00 (0.00, 0.00) | 0.40 (1.68)<br>0.00 (1.68) | 0.41 (1.03)<br>0.00 (1.03) | 0.01 |
| Number of lipid tests ordered | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 (1.00) | 0.00(1.03) | 0.00 |
| mean (sd) | 0.99 (0.93) | 1.06 (0.98) | 0.90 (1.15) | 1.11(1.15) | 1.01 (0.80) | 1.07 (0.83) | (0.90) | 1.09(1.02) | -0.11 |
| median (IOR) | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | | 1.00 [1.00, 2.00] | 1.00 (0.90) | 1.00(1.02) | 0.00 |
| Number of creatinine tests ordered | 2.52 [2.66, 2.66] | 2.52 (2.00, 2.00) | | | 2.22 (0.00, 2.00) | | 2.00 [0.50] | 200[202] | 0.00 |
| mean (sd) | 0.04 (0.28) | 0.04 (0.28) | 0.04 (0.29) | 0.03 (0.22) | 0.06 (0.31) | 0.06 (0.32) | 0.05 (0.30) | 0.04 (0.27) | 0.04 |
| median (IQR) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | | 0.00 (0.30) | 0.00 (0.27) | 0.00 |
| Number of BUN tests ordered | | | | | | | | | |
| mean (sd) | 0.02 (0.21) | 0.02 (0.18) | 0.03 (0.23) | 0.02 (0.16) | 0.04 (0.24) | 0.04 (0.24) | 0.04 (0.23) | 0.03 (0.19) | 0.05 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.23) | 0.00 (0.19) | 0.00 |
| Number of tests for microal burninuria | | | | | | | | | |
| mean (sd) | 0.75 (1.12) | 0.74 (1.11) | 0.61 (1.00) | 0.73 (1.09) | 0.45 (0.66) | 0.47 (0.68) | 0.52 (0.81) | 0.64 (0.97) | -0.13 |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.81) | 0.00 (0.97) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd digit level Cop | • | | | | | | | | |
| mean (sd) | PY<br>5.95 (7.69) | 3.93 (6.05) | 2.58 (4.25) | 2.81 (3.90) | 5.37 (7.03) | 6.34 (6.84) | 4.86 (6.64) | 4.28 (5.41) | 0.10 |
| median (IQR) | 4.00 [0.00, 9.00] | 0.00 [0.00, 6.00] | 0.00 [0.00, 4.00] | 0.00 [0.00, 5.00] | | 5.00 [0.00, 10.00] | 3.16 (6.64) | 1.77 (5.41) | 0.23 |
| - Party | -r.oc pr.oc, 5.00] | a.aa [a.aa, a.aa] | a.oo pr.oo, 4.00] | 0.00 [0.00, 0.00] | 4.00 (0.00, 0.00) | 2.22 [0.00, 20.00] | 3.20 (0.04) | 277 (3.42) | 0.23 |
| Use of thiazide; n (%) | 4,816 (11.0%) | 361 (10.4%) | 7,336 (10.5%) | 1,284 (9.7%) | 30,023 (13.6%) | 1,165 (12.6%) | 42,175 (12.6%) | 2,810 (10.8%) | 0.06 |
| Use of beta blockers; n (%) | 17,867 (40.9%) | 1,105 (31.7%) | 24,668 (35.2%) | 4,337 (32.6%) | 97,465 (44.3%) | 3,864 (41.9%) | 140,000 (41.9%) | 9,306 (35.8%) | 0.13 |
| Use of calcium channel blockers; n (%) | 11,695 (26.8%) | 766 (22.0%) | 17,484 (24.9%) | 3,114 (23.4%) | 70,925 (32.2%) | 2,700 (29.3%) | 100,104 (30.0%) | 6,580 (25.3%) | 0.11 |

| | | | | PS-matched | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Optur | m | MarketS | can | Medica | re | | POOLED | |
| Variable | Reference-DPP4i v2 E | oposure - Dapaglifozin v2 | Reference-DPP4i v2 E | oposure - Dapaglifozin v2 | Reference-DPP4iv2 B | xposure - Dapaglitozin v2 | Reference-DPP4i v2 | Exposure - Dapaglifozin v2 | St. Diff |
| Number of patients | 3316 | 3316 | 12415 | 12415 | 9164 | 9164 | 24,895 | 24,895 | |
| Age | | | | | | | | | |
| mean (sd) | 38.44 (7.64) | 58.61 (6.71) | 57.91 (6.56) | 58.10 (5.82) | 70.32 (4.86) | 70.31 (4.94) | 62.55 (6.16) | 62.66 (5.65) | -0.02 |
| median [IQR] | 58.00 [54.00, 62.00] | 58.00 [54.00, 62.00] | 58.00 [54.00, 61.00] | 58.00 [55.00, 61.00] | 69.00 [67.00, 73.00] | 69.00 [67.00, 73.00] | 62.05 (6.16) | 62.05 (5.65) | 0.00 |
| Age categories without zero category | | | | | | | | | |
| 18 - 34; n (%) | 1,019 (30.7%) | 840 (25.3%) | 3,275 (26.4%) | 2,905 (23.4%) | 0 (0.0%) | 0 (0.0%) | 4,294 (17.2%) | 3,745 (15.0%) | 0.06 |
| 55 -64; n (%) | 1,697 (51.2%) | 2,003 (60.4%) | 7,958 (64.1%) | 8,622 (69.4%) | 106 (1.2%) | 78 (0.9%) | 9,761 (39.2%) | 10,703 (43.0%) | -0.08 |
| 65 -74; n (%) | 475 (14.3%) | 388 (11.7%) | 942 (7.6%) | 733 (5.9%) | 7,436 (81.1%) | 7,495 (81.8%) | 8,853 (35.6%) | 8,616 (34.6%) | 0.02 |
| >=75; n (%) | 125 (3.8%) | 85 (2.6%) | 240 (1.9%) | 155 (1.2%) | 1,622 (17.7%) | 1,591 (17.4%) | 1,987 (8.0%) | 1,831 (7.4%) | 0.02 |
| Gender without zero category-United | | | | | | | | | |
| Maies; n (%) | 2,032 (61.3%) | 2,082 (62.8%) | 7,531 (60.7%) | 7,552 (60.8%) | 4,783 (52.2%) | 4,759 (51.9%) | 14,346 (57.6%) | 14,393 (57.8%) | 0.00 |
| Females; n (%) | 1,284 (38.7%) | 1,234 (37.2%) | 4,884 (39.3%) | 4,863 (39.2%) | 4,381 (47.8%) | 4,405 (48.1%) | 10,549 (42.4%) | 10,502 (42.2%) | 0.00 |
| Race | | | | | | | | | |
| White; n (%) | N/A | N/A | N/A | N/A | 7,401 (80.8%) | 7,387 (80.6%) | 7,401 (80.8%) | 7,387 (80.6%) | 0.01 |
| Black; n (%) | N/A | N/A | N/A | N/A | 799 (8.7%) | 756 (8.2%) | 799 (8.7%) | 756 (8.2%) | 0.02 |
| Asian; n (%) | N/A | N/A | N/A | N/A | 280 (3.1%) | 301 (3.3%) | 280 (3.1%) | 301 (3.3%) | -0.01 |
| Hispanic; n (%) | N/A | N/A | N/A | N/A | 283 (3.1%) | 298 (3.3%) | 283 (3.1%) | 298 (3.3%) | -0.01 |
| North American Native; n (%) | N/A | N/A | N/A | N/A | 29 (0.3%) | 25 (0.3%) | 29 (0.3%) | 25 (0.3%) | 0.00 |
| Other/Unknown; n (%)<br>Region without zero category-United v3 (lumping | N/A | N/A | N/A | N/A | 372 (4.1%) | 397 (4.3%) | 372 (4.1%) | 397 (4.3%) | -0.01 |
| missing&other category with West) | | | | | | | | | |
| Northeast; n (%) | 214 (6.5%) | 217 (6.5%) | 1,671 (13.5%) | 1,687 (13.6%) | 1,564 (17.1%) | 1,528 (16.7%) | 3,449 (13.9%) | 3,432 (13.8%) | 0.00 |
| South; n (%) | 1,859 (56.1%) | 1,874 (56.5%) | 2,045 (16.5%) | 2,095 (16.9%) | 4,342 (47.4%) | 4,257 (46.5%) | 8,246 (33.1%) | 8,226 (33.0%) | 0.00 |
| Midwest; n (%) | 832 (25.1%) | 795 (24.0%) | 7,690 (61.9%) | 7,595 (61.2%) | 1,780 (19.4%) | 1,822 (19.9%) | 10,302 (41.4%) | 10,212 (41.0%) | 0.01 |
| West; n (%) | 411 (12.4%) | 430 (13.0%) | 943 (7.6%) | 974 (7.8%) | 1,478 (16.1%) | 1,557 (17.0%) | 2,832 (11.4%) | 2,961 (11.9%) | -0.02 |
| Unknown+missing; n (%) | N/A | N/A | 66 (0.5%) | 64 (0.5%) | N/A | N/A | 66 (0.5%) | 64 (0.5%) | 0.00 |
| CV Covariates | | | | | | | | | |
| Ischemic heart disease; n (%) | 611 (18.4%) | 644 (19.4%) | 2,081 (16.8%) | 2,091 (16.8%) | 2,043 (22.3%) | 2,032 (22.2%) | 4,735 (19.0%) | 4,767 (19.1%) | 0.00 |
| Acute MI; n (%) | 31 (0.9%) | 32 (1.0%) | 68 (0.5%) | 68 (0.5%) | 45 (0.5%) | 45 (0.5%) | 144 (0.6%) | 145 (0.6%) | 0.00 |
| ACS/unstable angina; n (%) | 39 (1.2%) | 37 (1.1%) | 100 (0.8%) | 96 (0.8%) | 49 (0.5%) | 52 (0.6%) | 188 (0.8%) | 185 (0.7%) | 0.01 |
| Old MI; n (%) | 82 (2.5%) | 79 (2.4%) | 148 (1.2%) | 140 (1.1%) | 179 (2.0%) | 190 (2.1%) | 409 (1.6%) | 409 (1.6%) | 0.00 |
| Stable angina; n (%) | 99 (3.0%) | 107 (3.2%) | 296 (2.4%) | 320 (2.6%) | 292 (3.2%) | 283 (3.1%) | 687 (2.8%) | 710 (2.9%) | -0.01 |
| Coronary atherosclerosis and other forms of chronic | | | | | | | | | |
| ischemic heart disease; n (%) | 564 (17.0%) | 602 (18.2%) | 1,946 (15.7%) | 1,919 (15.5%) | 1,945 (21.2%) | 1,948 (21.3%) | 4,455 (17.9%) | 4,469 (18.0%) | 0.00 |
| Other atherosclerosis with ICD10 v2 Copy; n (%) | 27 (0.8%) | 21 (0.6%) | 55 (0.4%) | 53 (0.4%) | 82 (0.9%) | 80 (0.9%) | 164 (0.7%) | 154 (0.6%) | 0.01 |
| Previous cardiac procedure (CABG or PTCA or Stent) | 44 (0.781) | au to chi | 44 (0.4%) | 20 (0.281) | ac in niki | 17 (0.2%) | era (e rik) | 077 (0.7k) | 0.00 |
| v4; n (%) | 11 (0.3%)<br>147 (4.4%) | 21 (0.6%)<br>143 (4.4%) | 265 (2.1%) | 39 (0.3%)<br>270 (2.2%) | 16 (0.2%)<br>526 (5.7%) | 491 (5.4%) | 071 (0.3%)<br>938 (3.8%) | 077 (0.3%)<br>906 (3.6%) | 0.00 |
| History of CABG or PTCA; n (%) Any stroke; n (%) | 105 (3.2%) | 118 (3.6%) | 408 (3.3%) | 415 (3.3%) | | 543 (5.9%) | 1,038 (4.2%) | 1,076 (4.3%) | 0.00 |
| Ischemic stroke (w and w/o mention of cerebral | 103 (3.2%) | 118 (3.6%) | 400 (3.376) | 413 [3.376] | 525 (5.7%) | 343 (3.976) | 1,038 (4.276) | 1,076 [4.376] | 0.00 |
| infarction); n (%) | 105 (3.2%) | 115 (3.5%) | 407 (3.3%) | 415 (3.3%) | 519 (5.7%) | 542 (5.9%) | 1,031 (4.1%) | 1,072 (4.3%) | -0.01 |
| Hemorrhagic stroke; n (%) | 1 (0.0%) | 3 (0.1%) | 7 (0.1%) | 3 (0.0%) | 222 (2.774) | 2.2.0 | 2,002 (4.274) | 2,012 (3.374) | |
| ΠA; n (%) | 17 (0.5%) | 19 (0.6%) | 53 (0.4%) | 66 (0.5%) | 84 (0.9%) | 75 (0.8%) | 134 (0.6%) | 160 (0.6%) | 0.00 |
| Other cerebrovascular disease; n (%) | 26 (0.8%) | 22 (0.7%) | 75 (0.6%) | 75 (0.6%) | 101 (1.1%) | 113 (1.2%) | 202 (0.8%) | 210 (0.8%) | 0.00 |
| Late effects of cerebrovascular disease; n (%) | 12 (0.4%) | 14 (0.4%) | 50 (0.4%) | 51 (0.4%) | 63 (0.7%) | 79 (0.9%) | 125 (0.5%) | 144 (0.6%) | -0.01 |
| Cerebrovascular procedure; n (%) | 3 (0.1%) | 4 (0.1%) | 4 (0.0%) | 5 (0.0%) | | | | | |
| Heart failure (CHF); n (%) | 149 (4.5%) | 142 (4.3%) | 255 (2.1%) | 275 (2.2%) | 538 (5.9%) | 510 (5.6%) | 942 (3.8%) | 927 (3.7%) | 0.01 |
| Peripheral Vascular Disease (PVD) or PVD Surgery v2; | | | | | | | | | |
| n (%) | 122 (3.7%) | 127 (3.8%) | 376 (3.0%) | 382 (3.1%) | 632 (6.9%) | 641 (7.0%) | 1,130 (4.5%) | 1,150 (4.6%) | 0.00 |
| Atrial fibrillation; n (%) | 120 (3.6%) | 117 (3.5%) | 329 (2.7%) | 363 (2.9%) | 667 (7.3%) | 682 (7.4%) | 1,116 (4.5%) | 1,162 (4.7%) | -0.01 |
| Other cardiac dysrhythmia; n (%) | 165 (5.0%) | 175 (5.3%) | 472 (3.8%) | 483 (3.9%) | 849 (9.3%) | 842 (9.2%) | 1,486 (6.0%) | 1,500 (6.0%) | 0.00 |
| Cardiac conduction disorders; n (%) | 53 (1.6%) | 52 (1.6%) | 131 (1.1%) | 148 (1.2%) | 244 (2.7%) | 233 (2.5%) | 428 (1.7%) | 433 (1.7%) | 0.00 |
| Other CVD; n (%) | 231 (7.0%) | 223 (6.7%) | 650 (5.2%) | 629 (5.1%) | 947 (10.3%) | 927 (10.1%) | 1,828 (7.3%) | 1,779 (7.1%) | 0.01 |
| Diabetes related complications | | | | | | | | | |
| Diabetic retinopathy; n (%) | 124 (3.7%) | 142 (4.3%) | 367 (3.0%) | 373 (3.0%) | 590 (6.4%) | 615 (6.7%) | 1,081 (4.3%) | 1,130 (4.5%) | -0.01 |
| | | | | 2026-21 | and but-1 | 193 (2.1%) | 371 (1.5%) | 399 (1.6%) | -0.01 |
| Diabetes with other ophthalmic manifestations; n | n in all t | The second of the second of th | | | | | 371 (1 1%) | 399 (1 6%) | -0.01 |
| (%) | 2 (0.1%) | 3 (0.1%) | 173 (1.4%) | 203 (1.6%) | 196 (2.1%) | 255 (2.254) | 372(2.374) | 333 (2.0%) | |
| (%) Retinal detachment, vitreous hemorrhage, | | | | | | | | | |
| (%) Retinal detachment, vitreous hemorrhage, vitrectomy; n (%) | 5 (0.2%) | 9 (0.3%) | 36 (0.3%) | 30 (0.2%) | 46 (0.5%) | 31 (0.3%) | 087 (0.3%) | 070 (0.3%) | 0.00 |
| (%) Retinal detachment, vitreous hemorrhage, | | | | | | | | | |

| Occurrence of diabetic nephropathy V3 with ICD10 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Copy; n (%) | 183 (5.5%) | 172 (5.2%) | 455 (3.7%) | 479 (3.9%) | 481 (5.2%) | 495 (5.4%) | 1,119 (4.5%) | 1,146 (4.6%) | 0.00 |
| Hypoglycemia v2; n (%) | 73 (2.2%) | 71 (2.1%) | 191 (1.5%) | 200 (1.6%) | 128 (1.4%) | 116 (1.3%) | 392 (1.6%) | 387 (1.6%) | 0.00 |
| Hyperglycemia; n (%) | 112 (3.4%) | 107 (3.2%) | 449 (3.6%) | 437 (3.5%) | 348 (3.8%) | 345 (3.8%) | 909 (3.7%) | 889 (3.6%) | 0.01 |
| Disorders of fluid electrolyte and acid-base balance; n | | | | | | | | | |
| (%) | 91 (2.7%) | 94 (2.8%) | 343 (2.8%) | 332 (2.7%) | 271 (3.0%) | 288 (3.1%) | 705 (2.8%) | 714 (2.9%) | -0.01 |
| Diabetic ketoacidosis; n (%) | 10 (0.3%) | 7 (0.2%) | 13 (0.1%) | 12 (0.1%) | | | | | |
| Hyperosmolar hyperglycemic nonketotic syndrome | | | | | | | | | |
| (HONK); n (%) | 9 (0.3%) | 9 (0.3%) | 47 (0.4%) | 47 (0.4%) | 43 (0.5%) | 50 (0.5%) | 099 (0.4%) | 106 (0.4%) | 0.00 |
| Diabetes with peripheral circulatory disorders with | | | | | | | | | |
| ICD-10 v2 Copy; n (%) | 112 (3.4%) | 117 (3.5%) | 289 (2.3%) | 275 (2.2%) | 548 (6.0%) | 522 (5.7%) | 949 (3.8%) | 914 (3.7%) | 0.01 |
| Diabetic Foot; n (%) | 65 (2.0%) | 64 (1.9%) | 181 (1.5%) | 172 (1.4%) | 178 (1.9%) | 168 (1.8%) | 424 (1.7%) | 404 (1.6%) | 0.01 |
| Gangrenev2; n (%) | 5 (0.2%) | 5 (0.2%) | 15 (0.1%) | 18 (0.1%) | | | | | |
| Lower extremity amputation; n (%) | 21 (0.6%) | 20 (0.6%) | 48 (0.4%) | 38 (0.3%) | 35 (0.4%) | 29 (0.3%) | 104 (0.4%) | 087 (0.3%) | 0.02 |
| Osteomyelitis; n (%) | 21 (0.6%) | 19 (0.6%) | 46 (0.4%) | 51 (0.4%) | 34 (0.4%) | 27 (0.3%) | 101 (0.4%) | 097 (0.4%) | 0.00 |
| Skin infections v2; n (%) | 186 (5.6%) | 189 (5.7%) | 606 (4.9%) | 603 (4.9%) | 533 (5.8%) | 518 (5.7%) | 1,325 (5.3%) | 1,310 (5.3%) | 0.00<br>0.01 |
| Brectile dysfunction; n (%) | 147 (4.4%) | 136 (4.1%) | 385 (3.1%) | 387 (3.1%) | 295 (3.2%) | 268 (2.9%) | 827 (3.3%) | 791 (3.2%) | -0.01 |
| Diabetes with unspecified complication; n (%) Diabetes mellitus without mention of complications; | 131 (4.0%) | 131 (4.0%) | 638 (5.1%) | 669 (5.4%) | 509 (5.6%) | 515 (5.6%) | 1,278 (5.1%) | 1,315 (5.3%) | -0.01 |
| n (%) | 2,897 (87.4%) | 2,934 (88.5%) | 10,922 (88.0%) | 10,899 (87.8%) | 8,127 (88.7%) | 8,148 (88.9%) | 21,946 (88.2%) | 21,981 (88.3%) | 0.00 |
| Hypertension: 1 inpetient or 2 outpetient claims | 2,037 (07.470) | 2,554 (00.579) | 10,522 (00.074) | 10,035 (07.076) | 0,227 (00.770) | 0,240 (00.374) | 21,540 (00.274) | 21,301 (00.3/4) | 0.00 |
| within 365 days; n (%) | 2,554 (77.0%) | 2,578 (77.7%) | 9,099 (73.3%) | 9,066 (73.0%) | 7,910 (86.3%) | 7,933 (86.6%) | 19,563 (78.6%) | 19,577 (78.6%) | 0.00 |
| Hyperlipidemia v2; n (%) | 2,478 (74.7%) | 2,491 (75.1%) | 8,830 (71.1%) | 8,863 (71.4%) | 7,044 (76.9%) | 7,056 (77.0%) | 18,352 (73.7%) | 18,410 (74.0%) | -0.01 |
| Edema; n (%) | 158 (4.8%) | 146 (4.4%) | 358 (2.9%) | 343 (2.8%) | 540 (5.9%) | 557 (6.1%) | 1,056 (4.2%) | 1,046 (4.2%) | 0.00 |
| Renal Dysfunction (non-diabetic) v2; n (%) | 136 (4.1%) | 143 (4.3%) | 373 (3.0%) | 394 (3.2%) | 534 (5.8%) | 525 (5.7%) | 1,043 (4.2%) | 1,062 (4.3%) | 0.00 |
| Occurrence of acute renal disease v2; n (%) | 16 (0.5%) | 15 (0.5%) | 49 (0.4%) | 50 (0.4%) | 43 (0.5%) | 51 (0.6%) | 108 (0.4%) | 116 (0.5%) | -0.01 |
| Occurrence of chronic renal insufficiency; n (%) | 82 (2.5%) | 91 (2.7%) | 195 (1.6%) | 212 (1.7%) | 309 (3.4%) | 330 (3.6%) | 586 (2.4%) | 633 (2.5%) | -0.01 |
| Chronic kidney disease v2; n (%) | 63 (1.9%) | 76 (2.3%) | 169 (1.4%) | 173 (1.4%) | 276 (3.0%) | 285 (3.1%) | 508 (2.0%) | 534 (2.1%) | -0.01 |
| CKD Stage 3-4; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Occurrence of hypertensive nephropathy; n (%) | 41 (1.2%) | 39 (1.2%) | 92 (0.7%) | 93 (0.7%) | 137 (1.5%) | 134 (1.5%) | 270 (1.1%) | 266 (1.1%) | 0.00 |
| Occurrence of miscellaneous renal insufficiency v2; n | | | | | | | | | |
| (%) | 50 (1.5%) | 55 (1.7%) | 126 (1.0%) | 143 (1.2%) | 255 (2.8%) | 238 (2.6%) | 431 (1.7%) | 436 (1.8%) | -0.01 |
| Glaucoma or cataracts v2; n (%) | 410 (12.4%) | 403 (12.2%) | 1,445 (11.6%) | 1,423 (11.5%) | 2,357 (25.7%) | 2,332 (25.4%) | 4,212 (16.9%) | 4,158 (16.7%) | 0.01 |
| Cellulitis or abscess of toe; n (%) | 47 (1.4%) | 32 (1.0%) | 118 (1.0%) | 119 (1.0%) | 97 (1.1%) | 117 (1.3%) | 262 (1.1%) | 268 (1.1%) | 0.00 |
| Footulcer; n (%) | 61 (1.8%) | 59 (1.8%) | 175 (1.4%) | 173 (1.4%) | 169 (1.8%) | 163 (1.8%) | 405 (1.6%) | 395 (1.6%) | 0.00 |
| Bladder stones; n (%) | 3 (0.1%) | 0 (0.0%)<br>49 (1.5%) | 4 (0.0%)<br>141 (1.1%) | 6 (0.0%)<br>150 (1.2%) | 152 (1.7%) | 135 (1.5%) | 333 (1.3%) | 334 (1.3%) | 0.00 |
| Kidney stones; n (%) | 40 (1.2%) | | · · | | | | | , , , | 0.00 |
| Uninary tract infections (UTIs); n (%) | 7 (0.2%)<br>911 (27.5%) | 6 (0.2%)<br>853 (25.7%) | 57 (0.5%)<br>3,737 (30.1%) | 56 (0.5%)<br>3,629 (29.2%) | 60 (0.7%)<br>2,677 (29.2%) | 63 (0.7%)<br>2,690 (29.4%) | 124 (0.5%)<br>7,325 (29.4%) | 125 (0.5%)<br>7,172 (28.8%) | 0.00 |
| Dipstick urinalysis; n (%)<br>Non-dipstick urinalysis; n (%) | 1,387 (41.8%) | 1,371 (41.3%) | 5,150 (41.5%) | 5,074 (40.9%) | 3,897 (42.5%) | 3,816 (41.6%) | 10,434 (41.9%) | 10,261 (41.2%) | 0.01 |
| Urine function test; n (%) | 22 (0.7%) | 24 (0.7%) | 124 (1.0%) | 108 (0.9%) | 196 (2.1%) | 168 (1.8%) | 342 (1.4%) | 300 (1.2%) | 0.02 |
| Cytology; n (%) | 8 (0.2%) | 6 (0.2%) | 23 (0.2%) | 19 (0.2%) | 23 (0.3%) | 30 (0.3%) | 054 (0.2%) | 055 (0.2%) | 0.00 |
| Cystoscopy; n (%) | 7 (0.2%) | 8 (0.2%) | 37 (0.3%) | 36 (0.3%) | 48 (0.5%) | 34 (0.4%) | 092 (0.4%) | 078 (0.3%) | 0.02 |
| Other Covariates | () | -() | ( | | () | ( | ( | () | |
| Liver disease; n (%) | 68 (2.1%) | 73 (2.2%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 068 (0.3%) | 073 (0.3%) | 0.00 |
| Osteparthritis; n (%) | 324 (9.8%) | 358 (10.8%) | 1,189 (9.6%) | 1,184 (9.5%) | 1,832 (20.0%) | 1,811 (19.8%) | 3,345 (13.4%) | 3,353 (13.5%) | 0.00 |
| Other arthritis, arthropathies and musculoskeletal | | | | | | | | | |
| pain; n (%) | 1,072 (32.3%) | 1,027 (31.0%) | 3,446 (27.8%) | 3,493 (28.1%) | 3,560 (38.8%) | 3,511 (38.3%) | 8,078 (32.4%) | 8,031 (32.3%) | 0.00 |
| Dorsopathies; n (%) | 678 (20.4%) | 678 (20.4%) | 2,251 (18.1%) | 2,230 (18.0%) | 2,285 (24.9%) | 2,283 (24.9%) | 5,214 (20.9%) | 5,191 (20.9%) | 0.00 |
| Fractures; n (%) | 46 (1.4%) | 58 (1.7%) | 176 (1.4%) | 163 (1.3%) | 200 (2.2%) | 204 (2.2%) | 422 (1.7%) | 425 (1.7%) | 0.00 |
| Fallsv2; n (%) | 35 (1.1%) | 41 (1.2%) | 64 (0.5%) | 62 (0.5%) | 198 (2.2%) | 202 (2.2%) | 297 (1.2%) | 305 (1.2%) | 0.00 |
| Osteoporosis; n (%) | 54 (1.6%) | 55 (1.7%) | 136 (1.1%) | 136 (1.1%) | 480 (5.2%) | 482 (5.3%) | 670 (2.7%) | 673 (2.7%) | 0.00 |
| Hyperthyroidism; n (%) | 20 (0.6%) | 20 (0.6%) | 63 (0.5%) | 68 (0.5%) | 78 (0.9%) | 71 (0.8%) | 161 (0.6%) | 159 (0.6%) | 0.00 |
| Hypothyroidism v2; n (%) | 467 (14.1%) | 462 (13.9%) | 1,539 (12.4%) | 1,494 (12.0%) | 952 (10.4%) | 955 (10.4%) | 2,958 (11.9%) | 2,911 (11.7%) | 0.01<br>0.01 |
| Other disorders of thyroid gland V2; n (%) | 144 (4.3%) | 134 (4.0%)<br>237 (7.1%) | 453 (3.6%) | 463 (3.7%) | 462 (5.0%) | 415 (4.5%) | 1,059 (4.3%) | 1,012 (4.1%) | 0.01 |
| Depression; n (%) | 252 (7.6%)<br>227 (6.8%) | 220 (6.6%) | 792 (6.4%)<br>732 (5.9%) | 788 (6.3%)<br>724 (5.8%) | 734 (8.0%)<br>698 (7.6%) | 699 (7.6%)<br>652 (7.1%) | 1,778 (7.1%)<br>1,657 (6.7%) | 1,724 (6.9%)<br>1,596 (6.4%) | 0.01 |
| Anxiety; n (%)<br>Sleep Disorder; n (%) | 303 (9.1%) | 328 (9.9%) | 1,020 (8.2%) | 1,001 (8.1%) | 529 (5.8%) | 530 (5.8%) | 1,852 (7.4%) | 1,859 (7.5%) | 0.00 |
| Dementia; n (%) | 31 (0.9%) | 24 (0.7%) | 40 (0.3%) | 57 (0.5%) | 223 (2.4%) | 216 (2.4%) | 294 (1.2%) | 297 (1.2%) | 0.00 |
| Delirium; n (%) | 16 (0.5%) | 12 (0.4%) | 19 (0.2%) | 24 (0.2%) | 40 (0.4%) | 38 (0.4%) | 075 (0.3%) | 074 (0.3%) | 0.00 |
| Psychosis; n (%) | 19 (0.6%) | 12 (0.4%) | 32 (0.3%) | 35 (0.3%) | 67 (0.7%) | 62 (0.7%) | 118 (0.5%) | 109 (0.4%) | 0.01 |
| Obesity; n (%) | 841 (25.4%) | 845 (25.5%) | 2,353 (19.0%) | 2,343 (18.9%) | 1,566 (17.1%) | 1,517 (16.6%) | 4,760 (19.1%) | 4,705 (18.9%) | 0.01 |
| Overweight; n (%) | 144 (4.3%) | 146 (4.4%) | 354 (2.9%) | 344 (2.8%) | 371 (4.0%) | 368 (4.0%) | 869 (3.5%) | 858 (3.4%) | 0.01 |
| Smoking; n (%) | 285 (8.6%) | 314 (9.5%) | 649 (5.2%) | 680 (5.5%) | 981 (10.7%) | 974 (10.6%) | 1,915 (7.7%) | 1,968 (7.9%) | -0.01 |
| Alcohol abuse or dependence; n (%) | 15 (0.5%) | 26 (0.8%) | 44 (0.4%) | 44 (0.4%) | 46 (0.5%) | 41 (0.4%) | 105 (0.4%) | 111 (0.4%) | 0.00 |
| Drug abuse or dependence; n (%) | 42 (1.3%) | 31 (0.9%) | 65 (0.5%) | 71 (0.6%) | 92 (1.0%) | 78 (0.9%) | 199 (0.8%) | 180 (0.7%) | 0.01 |
| COPD; n (%) | 119 (3.6%) | 134 (4.0%) | 363 (2.9%) | 369 (3.0%) | 744 (8.1%) | 747 (8.2%) | 1,226 (4.9%) | 1,250 (5.0%) | 0.00 |

| *** 19:1 | (9·) | 4 = 2 (4 = 2) | and to add | 444 (2.494) | man (m mile) | ann in alti | a page (a alk) | a nen (a alki) | |
|---|---|---|---|---|---|---|---|---|---|
| Asthma; n (%) | 151 (4.6%) | 158 (4.8%) | 435 (3.5%) | 441 (3.6%) | 300 (5.5%) | 493 (5.4%) | 1,086 (4.4%) | 1,092 (4.4%) | 0.00 |
| Obstructive sleep apnea; n (%) | 375 (11.3%) | 387 (11.7%) | 1,490 (12.0%) | 1,464 (11.8%) | 820 (8.9%) | 841 (9.2%) | 2,685 (10.8%) | 2,692 (10.8%) | 0.00 |
| Pneumonia; n (%) | 53 (1.6%) | 43 (1.3%) | 108 (0.9%) | 110 (0.9%) | 130 (1.4%) | 134 (1.5%) | 291 (1.2%) | 287 (1.2%) | 0.00 |
| Imaging; n (%) | 2 (0.1%) | 1 (0.0%) | 5 (0.0%) | 3 (0.0%) | | | | - | |
| Diabetes Medications DM Medications - AGIs; n (%) | 10 (0.3%) | 7 (0.2%) | 31 (0.2%) | 32 (0.3%) | 77 (0.8%) | 36 (0.6%) | 118 (0.5%) | 095 (0.4%) | 0.01 |
| DM Medications - Glitazones; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| DM Medications - GLP-1 RA; n (%) | 598 (18.0%) | 599 (18.1%) | 1,777 (14.3%) | 1,937 (15.6%) | 1,480 (16.2%) | 1,463 (16.0%) | 3,855 (15.5%) | 3,999 (16.1%) | -0.02 |
| DM Medications - Insulin; n (%) | 797 (24.0%) | 830 (25.0%) | 2,835 (22.8%) | 2,944 (23.7%) | 2,495 (27.2%) | 2,509 (27.4%) | 6,127 (24.6%) | 6,283 (25.2%) | -0.01 |
| DM Medications - Meglitinides; n (%) | 18 (0.5%) | 20 (0.6%) | 106 (0.9%) | 113 (0.9%) | 147 (1.6%) | 153 (1.7%) | 271 (1.1%) | 286 (1.1%) | 0.01 |
| DM Medications - Metformin; n (%) | 2,488 (75.0%) | 2,517 (75.9%) | 9,948 (80.1%) | 9,865 (79.5%) | 6,908 (75.4%) | 6,834 (74.8%) | 19,344 (77.7%) | 19,236 (77.3%) | 0.01 |
| Concomitant initiation or current use of 2nd | 2,400 (75.070) | 2,327 (73.374) | 3,540 [00:279] | 5,005 (15.574) | 0,500 (75.474) | 0,034 (74.074) | 25,244 (77.774) | 25,250 (77.574) | |
| Generation SUs; n (%) | 885 (26.7%) | 882 (26.6%) | 3,002 (24.2%) | 3,012 (24.3%) | 2,916 (31.8%) | 2,966 (32.4%) | 6,803 (27.3%) | 6,860 (27.6%) | -0.01 |
| Concomitant initiation or current use of AGIs; n (%) | 6 (0.2%) | 3 (0.1%) | 20 (0.2%) | 21 (0.2%) | 49 (0.5%) | 40 (0.4%) | 075 (0.3%) | 064 (0.3%) | 0.00 |
| Concomitant initiation or current use of Glitazones; | . , | ` ' | | | | | | | |
| n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Concomitant initiation or current use of GLP-1 RA; n | | | | | | | | | |
| (%) | 395 (11.9%) | 402 (12.1%) | 1,158 (9.3%) | 1,271 (10.2%) | 1,033 (11.3%) | 1,075 (11.7%) | 2,586 (10.4%) | 2,748 (11.0%) | -0.02 |
| Concomitant initiation or current use of Insulin; n | | | | | | | | | |
| (%) | 594 (17.9%) | 609 (18.4%) | 2,180 (17.6%) | 2,233 (18.0%) | 2,018 (22.0%) | 2,002 (21.8%) | 4,792 (19.2%) | 4,844 (19.5%) | -0.01 |
| Concomitant initiation or current use of | | | | | | | | | |
| Meglitinides; n (%) | 15 (0.5%) | 13 (0.4%) | 87 (0.7%) | 64 (0.5%) | 100 (1.1%) | 107 (1.2%) | 202 (0.8%) | 184 (0.7%) | 0.01 |
| Concomitant initiation or current use of Metformin; | | | | | | | | | |
| n (%) | 2,021 (60.9%) | 2,049 (61.8%) | 8,574 (69.1%) | 8,537 (68.8%) | 5,896 (64.3%) | 5,902 (64.4%) | 16,491 (66.2%) | 16,488 (66.2%) | 0.00 |
| Past use of 2nd Generation SUs Copy; n (%) | 279 (8.4%) | 267 (8.1%) | 803 (6.5%) | 810 (6.5%) | 687 (7.5%) | 631 (6.9%) | 1,769 (7.1%) | 1,708 (6.9%) | 0.01 |
| Past use of AGIs Copy; n (%) | 4 (0.1%) | 4 (0.1%) | 11 (0.1%) | 11 (0.1%) | 28 (0.3%) | 16 (0.2%) | 043 (0.2%) | 031 (0.1%) | 0.03<br>#DIV/0! |
| Past use of Glitazones Copy; n (%) | 0 (0.0%)<br>230 (6.9%) | 0 (0.0%)<br>223 (6.7%) | 0 (0.0%)<br>675 (5.4%) | 0 (0.0%)<br>712 (5.7%) | 0 (0.0%)<br>447 (4.9%) | 0 (0.0%)<br>388 (4.2%) | 000 (0.0%)<br>1,352 (5.4%) | 000 (0.0%)<br>1,323 (5.3%) | 0.00 |
| Past use of GLP-1 RACopy; n (%) Past use of Insulin Copy; n (%) | 203 (6.1%) | 221 (6.7%) | 656 (5.3%) | 711 (5.7%) | 477 (5.2%) | 507 (5.5%) | 1,336 (5.4%) | 1,439 (5.8%) | -0.02 |
| Past use of Megitinides Copy; n (%) | 3 (0.1%) | 7 (0.2%) | 19 (0.2%) | 49 (0.4%) | 47 (0.5%) | 46 (0.5%) | 069 (0.3%) | 102 (0.4%) | -0.02 |
| Past use of metformin (final) Copy; n (%) | 467 (14.1%) | 468 (14.1%) | 1,374 (11.1%) | 1,328 (10.7%) | 1,012 (11.0%) | 952 (10.4%) | 2,853 (11.5%) | 2,748 (11.0%) | 0.02 |
| Other Medications | 407 [14.170] | 400 [14.1/0] | 1,3/4 [11.1/9] | 1,520 [10.7/9] | 1,012 [11.0/6] | 552 (10.4/6) | 2,035 [11.376] | 2,740 [11.0/9] | 0.02 |
| Use of ACE inhibitors; n (%) | 1,452 (43.8%) | 1,471 (44,4%) | 5,393 (43,4%) | 5,453 (43.9%) | 3.888 (42.4%) | 3.912 (42.7%) | 10.733 (43.1%) | 10.836 (43.5%) | -0.01 |
| Use of ARBs; n (%) | 922 (27.8%) | 939 (28.3%) | 3,785 (30.5%) | 3,740 (30.1%) | 3,074 (33.5%) | 3,092 (33.7%) | 7,781 (31.3%) | 7,771 (31.2%) | 0.00 |
| Use of Loop Diuretics - United; n (%) | 225 (6.8%) | 237 (7.1%) | 828 (6.7%) | 829 (6.7%) | 1,147 (12.5%) | 1,113 (12.1%) | 2,200 (8.8%) | 2,179 (8.8%) | 0.00 |
| Use of other diuretics- United; n (%) | 81 (2.4%) | 72 (2.2%) | 299 (2.4%) | 281 (2.3%) | 273 (3.0%) | 277 (3.0%) | 653 (2.6%) | 630 (2.5%) | 0.01 |
| Use of nitrates-United; n (%) | 135 (4.1%) | 130 (3.9%) | 441 (3.6%) | 453 (3.6%) | 454 (5.0%) | 471 (5.1%) | 1,030 (4.1%) | 1,054 (4.2%) | -0.01 |
| Use of other hypertension drugs; n (%) | 126 (3.8%) | 128 (3.9%) | 445 (3.6%) | 458 (3.7%) | 530 (5.8%) | 550 (6.0%) | 1,101 (4.4%) | 1,136 (4.6%) | -0.01 |
| Use of digoxin-United; n (%) | 23 (0.7%) | 30 (0.9%) | 84 (0.7%) | 87 (0.7%) | 189 (2.1%) | 197 (2.1%) | 296 (1.2%) | 314 (1.3%) | -0.01 |
| Use of Anti-arrhythmics; n (%) | 24 (0.7%) | 28 (0.8%) | 102 (0.8%) | 106 (0.9%) | 132 (1.4%) | 122 (1.3%) | 258 (1.0%) | 256 (1.0%) | 0.00 |
| Use of COPD/asthma meds- United; n (%) | 415 (12.5%) | 401 (12.1%) | 1,700 (13.7%) | 1,678 (13.5%) | 1,468 (16.0%) | 1,490 (16.3%) | 3,583 (14.4%) | 3,569 (14.3%) | 0.00 |
| Use of statins; n (%) | 2,212 (66.7%) | 2,214 (66.8%) | 8,213 (66.2%) | 8,228 (66.3%) | 6,530 (71.3%) | 6,605 (72.1%) | 16,955 (68.1%) | 17,047 (68.5%) | -0.01 |
| Use of other lipid-lowering drugs; n (%) | 402 (12.1%) | 436 (13.1%) | 1,714 (13.8%) | 1,755 (14.1%) | 1,196 (13.1%) | 1,176 (12.8%) | 3,312 (13.3%) | 3,367 (13.5%) | -0.01 |
| Use of antiplatelet agents; n (%) | 395 (11.9%) | 386 (11.6%) | 1,527 (12.3%) | 1,529 (12.3%) | 1,184 (12.9%) | 1,168 (12.7%) | 3,106 (12.5%) | 3,083 (12.4%) | 0.00 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, | | | | | | | | | |
| Apixaban, Warfarin); n (%) | 153 (4.6%) | 143 (4.3%) | 397 (3.2%) | 415 (3.3%) | 677 (7.4%) | 668 (7.3%) | 1,227 (4.9%) | 1,226 (4.9%) | 0.00 |
| Use of heparin and other low-molecular weight | | | | | | | | | |
| heparins; n (%) | 8 (0.2%) | 5 (0.2%) | 0 (0.0%) | 1 (0.0%) | 20 (0.2%) | 19 (0.2%) | 028 (0.1%) | 025 (0.1%) | 0.00 |
| Use of NSAIDs; n (%) | 540 (16.3%) | 353 (16.7%) | 2,347 (18.9%) | 2,306 (18.6%) | 1,677 (18.3%) | 1,600 (17.5%) | 4,564 (18.3%) | 4,461 (17.9%) | 0.01 |
| Use of oral corticosteroids; n (%) | 365 (11.0%) | 359 (10.8%) | 1,459 (11.8%) | 1,469 (11.8%) | 1,213 (13.2%) | 1,205 (13.1%) | 3,037 (12.2%) | 3,033 (12.2%) | 0.00 |
| Use of bisphosphonate (United); n (%) | 16 (0.5%)<br>749 (22.6%) | 20 (0.6%)<br>782 (23.6%) | 67 (0.5%)<br>2,822 (22.7%) | 66 (0.5%)<br>2,776 (22.4%) | 192 (2.1%)<br>1,931 (21.1%) | 185 (2.0%)<br>1,891 (20.6%) | 275 (1.1%)<br>5,502 (22.1%) | 271 (1.1%)<br>5,449 (21.9%) | 0.00 |
| Use of opioids-United; n (%) | 698 (21.0%) | 782 (23.6%)<br>732 (22.1%) | | 2,958 (23.8%) | | | 5,842 (23.5%) | | -0.01 |
| Use of antidepressants; n (%) | 58 (1.7%) | 732 (22.1%)<br>31 (1.3%) | 2,889 (23.3%)<br>176 (1.4%) | 198 (1.6%) | 2,255 (24.6%)<br>183 (2.0%) | 2,267 (24.7%)<br>187 (2.0%) | 417 (1.7%) | 5,957 (23.9%)<br>436 (1.8%) | -0.01 |
| Use of antipsychotics; n (%) | 478 (14.4%) | 462 (13.9%) | 1,471 (11.8%) | 1,488 (12.0%) | 1,448 (15.8%) | 1,463 (16.0%) | 3,397 (13.6%) | 3,413 (13.7%) | 0.00 |
| Use of anticonvulsants; n (%)<br>Use of lithium-United; n (%) | 6 (0.2%) | 2 (0.1%) | 17 (0.1%) | 16 (0.1%) | 2,773 (23.079) | 2,703 (20.079) | 2,227 (23,079) | 2,723(23.779) | 0.00 |
| Use of Benzos-United; n (%) | 336 (10.1%) | 327 (9.9%) | 1,239 (10.0%) | 1,241 (10.0%) | 926 (10.1%) | 914 (10.0%) | 2,501 (10.0%) | 2,482 (10.0%) | 0.00 |
| Use of anxiolytics/hypnotics-United; n (%) | 201 (6.1%) | 211 (6.4%) | 791 (6.4%) | 786 (6.3%) | 530 (5.8%) | 314 (3.6%) | 1,522 (6.1%) | 1,511 (6.1%) | 0.00 |
| Use of dementia meds-United; n (%) | 13 (0.4%) | 13 (0.4%) | 20 (0.2%) | 30 (0.2%) | 159 (1.7%) | 160 (1.7%) | 192 (0.8%) | 203 (0.8%) | 0.00 |
| Use of antiparkinsonian meds- United; n (%) | 48 (1.4%) | 48 (1.4%) | 221 (1.8%) | 220 (1.8%) | 289 (3.2%) | 265 (2.9%) | 558 (2.2%) | 533 (2.1%) | 0.01 |
| Any use of pramiintide; n (%) | 0 (0.0%) | 1 (0.0%) | 3 (0.0%) | 10 (0.1%) | | | | | |
| Any use of 1st generation sulfonyluress; n (%) | 0 (0.0%) | 0 (0.0%) | 1 (0.0%) | 0 (0.0%) | | | | | |
| Entresto (sacubitril/valsartan); n (%) | 4 (0.1%) | 3 (0.1%) | 8 (0.1%) | 1 (0.0%) | | | | | |
| Initiation as monotherapy v4 Copy; n (%) | 2,967 (89.5%) | 2,990 (90.2%) | 10,986 (88.5%) | 10,913 (87.9%) | 9,164 (100.0%) | 9,164 (100.0%) | 23,117 (92.9%) | 23,067 (92.7%) | 0.01 |
| Labs | | , , | | | | | 15,731 | 15,731 | |
| Lab values- HbA1.c (%) v3; n (%) | 1,334 (40.2%) | 1,332 (40.2%) | 941 (7.6%) | 798 (6.4%) | N/A | N/A | 2,275 (14.5%) | 2,130 (13.5%) | 0.03 |
| Lab values- HbA1c (%) (within 3 months) v3; n (%) | 1,092 (32.9%) | 1,085 (32.7%) | 788 (6.3%) | 646 (5.2%) | N/A | N/A | 1,880 (12.0%) | 1,731 (11.0%) | 0.03 |

| Lab values- HbA1c (%) (within 6 months) v3; n (%) | 1,334 (40.2%) | 1,332 (40.2%) | 941 (7.6%) | 798 (6.4%) | N/A | N/A | 2,275 (14.5%) | 2,130 (13.5%) | 0.03 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values- BNP; n (%) | 14 (0.4%) | 8 (0.2%) | 5 (0.0%) | 4 (0.0%) | N/A | N/A | 019 (0.1%) | 012 (0.1%) | 0.00 |
| Lab values- BNP (within 3 months); n (%) | 8 (0.2%) | 7 (0.2%) | 3 (0.0%) | 4(0.0%) | N/A | N/A | 011 (0.1%) | 011 (0.1%) | 0.00 |
| Lab values-BNP (within 6 months); n (%) | 14 (0.4%) | 8 (0.2%) | 5 (0.0%) | 4 (0.0%) | N/A | N/A | 019 (0.1%) | 012 (0.1%) | 0.00 |
| Lab values-BUN (mg/di); n (%) | 1,336 (40.3%) | 1,345 (40.6%) | 889 (7.2%) | 743 (6.0%) | N/A | N/A | 2,225 (14.1%) | 2,088 (13.3%) | 0.02 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 1,055 (31.8%) | 1,066 (32.1%) | 707 (5.7%) | 575 (4.6%) | N/A | N/A | 1,762 (11.2%) | 1,641 (10.4%) | 0.03 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 1,336 (40.3%) | 1,345 (40.6%) | 889 (7.2%) | 743 (6.0%) | N/A | N/A | 2,225 (14.1%) | 2,088 (13.3%) | 0.02 |
| Lab values- Creatinine (mg/dl) v2; n (%) | 1,381 (41.6%) | 1,381 (41.6%) | 970 (7.8%) | 792 (6.4%) | N/A | N/A | 2,351 (14.9%) | 2,173 (13.8%) | 0.03 |
| Lab values- Creatinine (mg/dl) (within 3 months) v2; | | | | . , | | | | | |
| n (%) | 1,095 (33.0%) | 1,098 (33.1%) | 775 (6.2%) | 616 (5.0%) | N/A | N/A | 1,870 (11.9%) | 1,714 (10.9%) | 0.03 |
| Lab values- Creatinine (mg/dl) (within 6 months) v2; | -, | 4 | ( | () | | | -,,, | 4.2.(2) | |
| | 1,381 (41.6%) | 4 204 (44 591) | 970 (7.8%) | 202 (5.4%) | N/A | N/A | 2,351 (14.9%) | 2,173 (13.8%) | 0.03 |
| n (%) | | 1,381 (41.6%) | \ <i>\</i> | 792 (6.4%) | | | | | |
| Lab values-HDL level (mg/dl); n (%) | 1,219 (36.8%) | 1,180 (35.6%) | 869 (7.0%) | 761 (6.1%) | N/A | N/A | 2,088 (13.3%) | 1,941 (12.3%) | 0.03 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 925 (27.9%) | 890 (26.8%) | 664 (5.3%) | 364 (4.5%) | N/A | N/A | 1,589 (10.1%) | 1,454 (9.2%) | 0.03 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 1,219 (36.8%) | 1,180 (35.6%) | 869 (7.0%) | 761 (6.1%) | N/A | N/A | 2,088 (13.3%) | 1,941 (12.3%) | 0.03 |
| Lab values-LDL level (mg/dl) v2; n (%) | 1,241 (37.4%) | 1,203 (36.3%) | 879 (7.1%) | 738 (5.9%) | N/A | N/A | 2,120 (13.5%) | 1,941 (12.3%) | 0.04 |
| Lab values-LDL level (mg/dl) (within 3 months) v2; n | | | | | | | | | |
| (%) | 944 (28.5%) | 907 (27.4%) | 671 (5.4%) | 550 (4.4%) | N/A | N/A | 1,615 (10.3%) | 1,457 (9.3%) | 0.03 |
| Lab values- LDL level (mg/dl) (within 6 months) v2; n | () | () | | () | | | -,,, | 2,101 (0.014) | |
| | 1,241 (37.4%) | 1,203 (36.3%) | 879 (7.1%) | 738 (5.9%) | N/A | N/A | 2,120 (13.5%) | 1,941 (12.3%) | 0.04 |
| (%) | | | | | N/A | | | | 0.04 |
| Lab values-NT-proBNP; n (%) | 3 (0.1%) | 5 (0.2%) | 1 (0.0%) | 1 (0.0%) | | N/A | 04 (0.0%) | 0 (0.0%) | - |
| Lab values- NT-proBNP (within 3 months); n (%) | 1 (0.0%) | 3 (0.1%) | 1 (0.0%) | 0 (0.0%) | N/A | N/A | 02 (0.0%) | 0 (0.0%) | - |
| Lab values- NT-proBNP (within 6 months); n (%) | 3 (0.1%) | 5 (0.2%) | 1 (0.0%) | 1 (0.0%) | N/A | N/A | 04 (0.0%) | 6 (0.0%) | - |
| Lab values-Total cholesterol (mg/dl) v2; n (%) | 1,249 (37.7%) | 1,212 (36.6%) | 875 (7.0%) | 766 (6.2%) | N/A | N/A | 2,124 (13.5%) | 1,978 (12.6%) | 0.03 |
| Lab values-Total cholesterol (mg/dl) (within 3 | | | | | | | | | |
| months) v2; n (%) | 950 (28.6%) | 913 (27.5%) | 668 (5.4%) | 568 (4.6%) | N/A | N/A | 1,618 (10.3%) | 1,481 (9.4%) | 0.03 |
| Lab values-Total cholesterol (mg/dl) (within 6 | (/ | () | | () | - | - | -,,, | -, | |
| months) v2; n (%) | 1,249 (37.7%) | 1,212 (36.6%) | 875 (7.0%) | 766 (6.2%) | N/A | N/A | 2,124 (13.5%) | 1,978 (12.6%) | 0.03 |
| | 1,237 (37.3%) | 1,211 (36.5%) | 868 (7.0%) | 752 (6.1%) | N/A | N/A | 2,105 (13.4%) | 1,963 (12.5%) | 0.03 |
| Lab values-Triglyceride level (mg/dl); n (%) | 1,237 (37.370) | 1,211 (50.5/6) | 868 (7.074) | 732(8.176) | NA. | N/A | 2,103 (13,4/6) | 1,563 (12.3/6) | 0.03 |
| Lab values-Triglyceride level (mg/dl) (within 3 | | | | | | | ( | | |
| months); n (%) | 941 (28.4%) | 914 (27.6%) | 662 (5.3%) | 559 (4.5%) | N/A | N/A | 1,603 (10.2%) | 1,473 (9.4%) | 0.03 |
| Lab values-Triglyceride level (mg/dl) (within 6 | | | | | | | | | |
| months); n (%) | 1,237 (37.3%) | 1,211 (36.5%) | 868 (7.0%) | 752 (6.1%) | N/A | N/A | 2,105 (13.4%) | 1,963 (12.5%) | 0.03 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | | | | | | | | | |
| included) v4 | 1,326 | 1,325 | 930 | 791 | N/A | N/A | 2,256 | 2,116 | |
| mean (sd) | 8.62 (1.81) | 8.59 (1.74) | 8.57 (1.88) | 8.51 (1.81) | N/A | N/A | 8.60 (1.84) | 8.56 (1.77) | 0.02 |
| median (IQR) | 8.25 [7.30, 9.60] | 8.20 [7.40, 9.50] | 8.10 [7.30, 9.60] | 8.00 [7.20, 9.50] | N/A | N/A | 8.19 (1.84) | 8.13 (1.77) | 0.03 |
| Missing n (%) | 1,990 (60.0%) | 1,991 (60.0%) | 11,485 (92.5%) | 11,624 (93.6%) | N/A | N/A | 13,475 (85.7%) | 13,615 (86.5%) | -0.02 |
| Lab result number- BNP mean v2 | 1,550 (60.0/6) | 1,331 (00.0%) | 11,463 (32.3/6) | 11,024 (33.070) | N/A | N/A | 13,473 (03.776) | 13,013 (00.3/6) | -0.02 |
| mean (sd) | 116.35 (114.30) | 62.94 (82.60) | 234.87 (258.20) | 25.75 (28.92) | N/A | N/A | 147.54 (165.17) | 50.54 (74.74) | 0.76 |
| median [IQR] | 56.45 [47.44, 207.60] | 13.10 [1.23, 159.75] | 147.00 [33.00, 460.67] | 20.00 [1.50, 55.75] | N/A | N/A | #VALUE! | 15.40 (74.74) | #VALUE! |
| Missing; n (%) | 3,302 (99.6%) | 3,308 (99.8%) | 12,410 (100.0%) | 12,411 (100.0%) | N/A | N/A | 15,712 (99.9%) | 15,719 (99.9%) | 0.00 |
| Lab result number- BUN (mg/di) mean v2 | 1,336 | 1,345 | 889 | 743 | N/A | N/A | 2,225 | 2,088 | |
| mean (sd) | 15.77 (5.28) | 15.66 (4.62) | 1,028.37 (11,952.55) | 237.83 (6,052.69) | N/A | N/A | 420.35 (7556.05) | 94.72 (3610.75) | 0.05 |
| median [IQR] | 15.00 [12.00, 18.00] | 15.00 [12.50, 18.00] | 15.33 [13.00, 18.50] | 15.00 [12.67, 18.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing n (%) | 1,980 (59.7%) | 1,971 (59.4%) | 11,526 (92.8%) | 11,672 (94.0%) | N/A | N/A | 13,506 (85.9%) | 13,643 (86.7%) | -0.02 |
| | 2,500 (55.776) | 2,372 (33.470) | 22,520 (52.0/9) | 22,072 (34.079) | 144 | N/A | 23,500 (05.576) | 22,043 [00.776] | 20.02 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 | 1,365 | 1,375 | 833 | 671 | N/A | N/A | 2.198 | 2,046 | |
| to 15 included) v3 | | | | | | | -, | | |
| mean (sd) | 0.91 (0.24) | 0.88 (0.19) | 0.94 (0.25) | 0.90 (0.19) | N/A | N/A | 0.92 (0.24) | 0.89 (0.19) | 0.14 |
| median [IQR] | 0.88 [0.76, 1.02] | 0.88 [0.74, 1.00] | 0.92 [0.77, 1.05] | 0.89 [0.76, 1.00] | N/A | N/A | 0.90 (0.24) | 0.88 (0.19) | 0.09 |
| Missing; n (%) | 1,951 (58.8%) | 1,941 (58.5%) | 11,582 (93.3%) | 11,744 (94.6%) | N/A | N/A | 13,533 (86.0%) | 13,685 (87.0%) | -0.03 |
| Lab result number- HDL level (mg/dl) mean (only | | | | | | | | | |
| =5000 included)v2 | 1,219 | 1,180 | 862 | 761 | N/A | N/A | 2,081 | 1,941 | |
| mean (sd) | 44.13 (12.67) | 43.43 (12.38) | 44.38 (13.55) | 44.06 (12.72) | N/A | N/A | 44.23 (13.04) | 43.68 (12.52) | 0.04 |
| median (IQR) | 42.00 [36.00, 51.00] | 42.00 [35.00, 51.00] | 42.58 [36.00, 52.12] | 42.50 [36.00, 51.00] | N/A | N/A | 42.24 (13.04) | 42.20(12.52) | 0.00 |
| | 2,097 (63.2%) | 2,136 (64.4%) | 11,553 (93.1%) | | N/A | N/A | 13,650 (86.8%) | 13,790 (87.7%) | -0.03 |
| Missing; n (%) | 2,057 (03.276) | 2,130 (44.4/6) | 11,333 [33.176] | 11,654 (93.9%) | nya. | NyA | 13,030 (00.078) | 13,730 07.776 | -0.05 |
| Lab result number-LDL level (mg/di) mean (only | | | | | aut- | | | | |
| =5000 included) v2 | 1,214 | 1,193 | 783 | 658 | N/A | N/A | 1,997 | 1,851 | |
| mean (sd) | 87.83 (43.08) | 82.21 (39.52) | 89.06 (43.42) | 89.56 (43.82) | N/A | N/A | 88.31 (43.22) | 84.82 (41.11) | 0.08 |
| median [IQR] | 88.00 [62.88, 112.50] | 83.00 [61.00, 105.75] | 88.00 [64.00, 116.00] | 88.00 [63.00, 114.00] | N/A | N/A | 88.00 (43.22) | 84.78 (41.11) | 0.08 |
| Missing n (%) | 2,102 (63.4%) | 2,123 (64.0%) | 11,632 (93.7%) | 11,757 (94.7%) | N/A | N/A | 13,734 (87.3%) | 13,880 (88.2%) | -0.03 |
| Lab result number-Total cholesterol (mg/dl) mean | . , | . , | | . , | | | . , | . , | |
| (only =:5000 included) v2 | 1,249 | 1,212 | 868 | 766 | N/A | N/A | 2,117 | 1,978 | |
| mean (sd) | 179.01 (47.89) | 173.61 (44.15) | 180.73 (52.25) | 177.64 (49.97) | N/A | N/A | 179.72 (49.74) | 175.17 (46.50) | 0.09 |
| median (IQR) | 173.00 [149.00, 203.75] | | 176.00 [150.00, 206.75] | | N/A | N/A | 174.23 (49.74) | 169.39 (46.50) | 0.10 |
| | | | | | N/A | N/A | · · · | | -0.03 |
| Missing; n (%) | 2,067 (62.3%) | 2,104 (63.4%) | 11,547 (93.0%) | 11,649 (93.8%) | NγA | N/A | 13,614 (86.5%) | 13,753 (87.4%) | -0.03 |

| Lab result number-Triglyceride level (mg/dl) mean | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| (only =: 5000 included) v2 | 1,237 | 1,211 | 860 | 752 | N/A | N/A | 2,097 | 1,963 | |
| mean (sd) | 212.55 (198.62) | 210.19 (184.38) | 214.38 (222.01) | 204.46 (193.38) | N/A | N/A | 213.30 (208.58) | 207.99 (187.93) | 0.03 |
| median [IQR] | 162.00 [114.25, 239.00] | 164.00 [118.00, 237.00] | 159.00 [110.00, 239.00] | 162.00 [110.21, 238.75] | N/A | N/A | 160.77 (208.58) | 163.23 (187.93) | -0.01 |
| Missing n (%) | 2,079 (62.7%) | 2,105 (63.5%) | 11,555 (93.1%) | 11,663 (93.9%) | N/A | N/A | 13,634 (86.7%) | 13,768 (87.5%) | -0.02 |
| Lab result number- Hemoglobin mean (only >0 | | | | | | | | | |
| included) | 897 | 876 | 629 | 508 | N/A | N/A | 1,526 | 1,384 | |
| mean (sd) | 14.17 (1.61) | 14.23 (1.56) | 1,097.16 (12,155.32) | 13.93 (1.54) | N/A | N/A | 460.57 (7805.42) | 14.12 (1.55) | 0.08 |
| median [IQR] | 14.20 [13.10, 15.30] | 14.30 [13.20, 15.26] | 13.95 [12.80, 15.00] | 14.00 [13.00, 15.00] | N/A | N/A | #VALUE! | 14.19 (1.55) | #WALUE! |
| Missing n (%) | 2,419 (72.9%) | 2,440 (73.6%) | 11,786 (94.9%) | 11,907 (95.9%) | N/A | N/A | 14,205 (90.3%) | 14,347 (91.2%) | -0.03 |
| Lab result number- Serum sodium mean (only > 90 | 1.350 | 1,348 | 929 | 787 | N/A | N/A | 2.279 | 2.135 | |
| and < 190 included)mean (sd) | 139.04 (2.65) | 139.22 (2.47) | 138.78(2.67) | 138.83 (2.36) | N/A | N/A<br>N/A | 138.93 (2.66) | 139.08 (2.43) | -0.06 |
| median [IQR] | 139.00 [137.00, 141.00] | 139.00 [138.00, 141.00] | 139.00 [137.00, 140.50] | 139.00 [137.00, 140.25] | N/A | N/A | 139.00 (2.66) | 139.00 (2.43) | 0.00 |
| Missing; n (%) | 1,966 (59.3%) | 1,968 (59.3%) | 11,486 (92.5%) | 11,628 (93.7%) | N/A | N/A | 13,452 (85.5%) | 13,596 (86.4%) | -0.03 |
| Lab result number- Albumin mean (only >0 and <=10 | -,, | 4,000 | | ,, | | | | ,() | |
| included) | 1,299 | 1,279 | 786 | 678 | N/A | N/A | 2,085 | 1,957 | |
| mean (sd) | 4.33 (0.30) | 4.34 (0.30) | 4.18 (0.44) | 4.20 (0.40) | N/A | N/A | 4.27 (0.36) | 4.29 (0.34) | -0.06 |
| median [IQR] | 4.30 [4.15, 4.50] | 4.35 [4.20, 4.55] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.45] | N/A | N/A | 4.26 (0.36) | 4.30 (0.34) | -0.11 |
| Missing; n (%) | 2,017 (60.8%) | 2,037 (61.4%) | 11,629 (93.7%) | 11,737 (94.5%) | N/A | N/A | 13,646 (86.7%) | 13,774 (87.6%) | -0.03 |
| Lab result number- Glucose (fasting or random) mean | | | | | | | | | |
| (only 10-1000 included) | 1,348 | 1,350 | 938 | 790 | N/A | N/A | 2,286 | 2,140 | |
| mean (sd) | 184.77 (72.64) | 176.69 (65.63) | 184.89 (75.51) | 178.63 (66.52) | N/A | N/A | 184.82 (73.85) | 177.41 (65.98) | 0.11 |
| median (IQR) | 168.75 [131.00, 221.00] | 160.58 [132.00, 209.00] | 167.00 [134.00, 218.00] | 164.00 [133.88, 212.00] | N/A | N/A | 168.03 (73.85) | 161.84 (65.98) | 0.09 |
| Missing n (%) | 1,968 (59.3%) | 1,966 (59.3%) | 11,477 (92.4%) | 11,625 (93.6%) | N/A | N/A | 13,445 (85.5%) | 13,591 (86.4%) | -0.03 |
| Lab result number- Potassium mean (only 1-7<br>included) | 1,368 | 1,369 | 886 | 720 | N/A | N/A | 2,254 | 2,089 | |
| mean (sd) | 4.44 (0.39) | 4.42 (0.39) | 4.33 (0.43) | 4.29 (0.42) | N/A | N/A | 4.40 (0.41) | 4.38 (0.40) | 0.05 |
| median (IQR) | 4.40 [4.20, 4.70] | 4.40 [4.20, 4.65] | 4.30 [4.00, 4.60] | 4.30 [4.00, 4.50] | N/A | N/A | 4.36 (0.41) | 4.37 (0.40) | -0.02 |
| Missing n (%) | 1,948 (58.7%) | 1,947 (58.7%) | 11,529 (92.9%) | 11,695 (94.2%) | N/A | N/A | 13,477 (85.7%) | 13,642 (86.7%) | -0.03 |
| Comorbidity Scores | | | | | | | | | |
| CCI (180 days)-ICD9 and ICD10 v2 | | | | | | | | | |
| mean (sd) | 1.69 (1.30) | 1.71 (1.29) | 1.49 (1.10) | 1.51 (1.10) | 2.11 (1.41) | 2.10 (1.41) | 1.74 (1.25) | 1.75 (1.25) | -0.01 |
| median [IQR] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 1.37 (1.25) | 1.37 (1.25) | 0.00 |
| Frailty Score: Qualitative Version 365 days as | | | | | | | | | |
| Categories, v1 | (0-) | | | | | | | | 0.02 |
| 0; n (%) | 1,875 (56.5%) | 1,788 (53.9%) | 7,443 (60.0%) | 7,280 (58.6%) | 5,602 (61.1%) | 5,623 (61.4%) | 14,920 (59.9%) | 14,691 (59.0%) | |
| 1 to 2; n (%) | 1,063 (32.1%)<br>378 (11.4%) | 1,151 (34.7%)<br>377 (11.4%) | 3,907 (31.5%)<br>1,063 (8.6%) | 4,036 (32.5%)<br>1,099 (8.9%) | 2,368 (25.8%)<br>1,194 (13.0%) | 2,382 (26.0%)<br>1,159 (12.6%) | 7,338 (29.5%)<br>2,637 (10.6%) | 7,569 (30.4%)<br>2,635 (10.6%) | -0.02<br>0.00 |
| 3 or more; n (%)<br>Frailty Score: Empirical Version 365 days as | 3/0 (11.4/0) | 3//(11.4/0) | 1,000 (0.0/0) | 1,055 (0.5/6) | 1,154(15.0/0) | 1,139 (12.0/9) | 2,037 (10.079) | 2,033 (10.0/6) | 0.00 |
| Categories, v3 | | | | | | | | | |
| <0.12908; n (%) | 1,208 (36.4%) | 1,152 (34.7%) | 4,498 (36.2%) | 4,477 (36.1%) | 1,848 (20.2%) | 1,794 (19.6%) | 7,554 (30.3%) | 7,423 (29.8%) | 0.01 |
| 0.12908 -0.1631167; n (%) | 1,121 (33.8%) | 1,199 (36.2%) | 4,449 (35.8%) | 4,461 (35.9%) | 2,986 (32.6%) | 3,028 (33.0%) | 8,556 (34.4%) | 8,688 (34.9%) | -0.01 |
| >=0.1631167; n (%) | 987 (29.8%) | 965 (29.1%) | 3,468 (27.9%) | 3,477 (28.0%) | 4,330 (47.3%) | 4,342 (47.4%) | 8,785 (35.3%) | 8,784 (35.3%) | 0.00 |
| Non-Frailty; n (%) | 1,787 (53.9%) | 1,739 (52.4%) | 6,483 (52.2%) | 6,469 (52.1%) | 514 (5.6%) | 381 (4.2%) | 8,784 (35.3%) | 8,589 (34.5%) | 0.02 |
| Frailty Score (mean): Qualitative Version 365 days, v1 | | | | | | | | | |
| mean (sd) | 0.88 (1.38) | 0.92 (1.38) | 0.74(1.17) | 0.77 (1.20) | 0.88 (1.49) | 0.87 (1.45) | 0.81 (1.32) | 0.83 (1.32) | -0.02 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (1.32) | 0.00 (1.32) | 0.00 |
| Prailty Score (mean): Empirical Version 365 days, v2 | 0.47 (0.04) | 0.45 (0.04) | 0.44/0.04 | 0.44(0.04) | 0.47 (0.08) | 0.47 (0.08) | 0.15 (0.04) | 0.15 (0.04) | 0.00 |
| mean (sd)<br>median (IQR) | 0.15 (0.04)<br>0.14 [0.12, 0.17] | 0.15 (0.04)<br>0.14 (0.12, 0.17) | 0.14 (0.04)<br>0.14 (0.12, 0.16) | 0.14 (0.04)<br>0.14 (0.12, 0.16) | 0.17 (0.05)<br>0.16 (0.13, 0.19) | 0.17 (0.05)<br>0.16 (0.14, 0.19) | 0.15 (0.04) | 0.15 (0.04) | 0.00 |
| Healthcare Utilization | 0.14[0.12, 0.17] | 0.14(0.12, 0.17) | 0.14(0.12, 0.10) | 0.14(0.12, 0.10) | 0.10 [0.13, 0.15] | 0.10 [0.14, 0.15] | 0.13 (0.04) | 0.13 (0.04) | 0.00 |
| Any hospitalization; n (%) | 120 (3.6%) | 132 (4.0%) | 362 (2.9%) | 380 (3.1%) | 322 (3.5%) | 313 (3.4%) | 804 (3.2%) | 825 (3.3%) | -0.01 |
| Any hospitalization within prior 30 days; n (%) | 27 (0.8%) | 23 (0.7%) | 38 (0.3%) | 52 (0.4%) | 44 (0.5%) | 48 (0.5%) | 109 (0.4%) | 123 (0.5%) | -0.01 |
| Any hospitalization during prior 31-180 days; n (%) | 95 (2.9%) | 111 (3.3%) | 325 (2.6%) | 334 (2.7%) | 281 (3.1%) | 273 (3.0%) | 701 (2.8%) | 718 (2.9%) | -0.01 |
| Endocrinologist Visit; n (%) | 586 (17.7%) | 605 (18.2%) | 1,792 (14.4%) | 1,866 (15.0%) | 1,429 (15.6%) | 1,435 (15.7%) | 3,807 (15.3%) | 3,906 (15.7%) | -0.01 |
| Endocrinologist Visit (30 days prior); n (%) | 433 (13.1%) | 449 (13.5%) | 1,363 (11.0%) | 1,398 (11.3%) | 943 (10.3%) | 951 (10.4%) | 2,739 (11.0%) | 2,798 (11.2%) | -0.01 |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 413 (12.5%) | 416 (12.5%) | 1,163 (9.4%) | 1,207 (9.7%) | 1,107 (12.1%) | 1,100 (12.0%) | 2,683 (10.8%) | 2,723 (10.9%) | 0.00 |
| Internal medicine/family medicine visits; n (%) | 1,971 (59.4%) | 1,968 (59.3%) | 10,936 (88.1%) | 10,932 (88.1%) | 7,411 (80.9%) | 7,303 (79.7%) | 20,318 (81.6%) | 20,203 (81.2%) | 0.01 |
| Internal medicine/family medicine visits (30 days | | | | | | | | | |
| prior) v2; n (%) | 1,303 (39.3%) | 1,325 (40.0%) | 8,395 (67.6%) | 8,318 (67.0%) | 5,254 (57.3%) | 5,160 (56.3%) | 14,952 (60.1%) | 14,803 (59.5%) | 0.01 |
| Internal medicine/family medicine visits (31 to 180 | 4 540 (40 00) | 4 543 (45 =61 | 0.000/73 491 | 0.007/77.781 | C 447/70 491 | c 20c/co ch1 | 47 055 (cg = 2·1 | 47 00c/co 381 | 0.00 |
| days prior) v2; n (%)<br>Cardiologist visit; n (%) | 1,618 (48.8%)<br>722 (21.8%) | 1,643 (49.5%)<br>707 (21.3%) | 8,990 (72.4%)<br>2,377 (19.1%) | 8,967 (72.2%)<br>2,316 (18.7%) | 6,447 (70.4%)<br>2,283 (24.9%) | 6,396 (69.8%)<br>2,279 (24.9%) | 17,055 (68.5%)<br>5,382 (21.6%) | 17,006 (68.3%)<br>5,302 (21.3%) | 0.00 |
| Number of Cardiologist visits (30 days prior); n (%) | 268 (8.1%) | 243 (7.3%) | 708 (5.7%) | 698 (5.6%) | 680 (7.4%) | 687 (7.5%) | 1,656 (6.7%) | 1,628 (6.5%) | 0.01 |
| manage of cardiologic visits (so only prior ), it (re) | 200 (0.270) | 242 (7.3/0) | 700 (3.779) | 050[5.0/6] | 000 [7.470] | 007 [7.376] | 2,030 [0.776] | 2,020 [0.3/6] | 3.01 |

| Number of Cardiologist visits (31 to 180 days prior); | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| n (%) | 593 (17.9%) | 591 (17.8%) | 2,013 (16.2%) | 1,958 (15.8%) | 1,972 (21.5%) | 1,989 (21.7%) | 4,578 (18.4%) | 4,538 (18.2%) | 0.01 |
| Bectrocardiogram v2; n (%) | 792 (23.9%) | 780 (23.5%) | 3,120 (25.1%) | 3,010 (24.2%) | 2,420 (26.4%) | 2,441 (26.6%) | 6,332 (25.4%) | 6,231 (25.0%) | 0.01 |
| Use of glucose test strips; n (%) | 134 (4.0%) | 128 (3.9%) | 476 (3.8%) | 472 (3.8%) | 214 (2.3%) | 227 (2.5%) | 824 (3.3%) | 827 (3.3%) | 0.00 |
| Dialysis; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Naive new user v8 Copy; n (%) | 396 (11.9%) | 368 (11.1%) | 1,573 (12.7%) | 1,609 (13.0%) | 864 (9.4%) | 877 (9.6%) | 2,833 (11.4%) | 2,854 (11.5%) | 0.00 |
| Nantidiabetic drugs at index date v3 Copy | | | | | | | | | |
| mean (sd) | 2.19 (0.83) | 2.20 (0.87) | 2.21 (0.79) | 2.22 (0.83) | 2.31 (0.77) | 2.32 (0.86) | 2.24 (0.79) | 2.25 (0.85) | -0.01 |
| median [IQR] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | 2.00 (0.79) | 2.00 (0.85) | 0.00 |
| number of different/distinct medication | | | | | | | | | |
| prescriptions | | | | | | | | | |
| mean (sd) | 9.40 (4.76) | 9.51 (4.66) | 9.50 (4.58) | 9.50 (4.46) | 9.75 (4.27) | 9.75 (4.29) | 9.58 (4.49) | 9.59 (4.43) | 0.00 |
| median (IQR) Number of Hospitalizations | 9.00 [6.00, 12.00] | 9.00 [6.00, 12.00] | 9.00 [6.00, 12.00] | 9.00 [6.00, 12.00] | 9.00 [7.00, 12.00] | 9.00 [7.00, 12.00] | 9.00 (4.49) | 9.00 (4.43) | 0.00 |
| | 0.04/0.74 | 0.04 (0.33) | 0.07 (0.40) | 0.02 (0.20) | 0.04 (0.22) | 0.04(0.77) | 0.04/0.741 | 0.04/0.741 | |
| mean (sd) | 0.04 (0.21) | 0.04 (0.22)<br>0.00 (0.00, 0.00) | 0.03 (0.19)<br>0.00 (0.00, 0.00) | 0.03 (0.20)<br>0.00 (0.00, 0.00) | 0.04 (0.23)<br>0.00 (0.00, 0.00) | 0.04 (0.23)<br>0.00 (0.00, 0.00) | 0.04 (0.21) | 0.04 (0.21) | 0.00 |
| median (ICR) | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 (0.21) | 0.00 (0.21) | 0.00 |
| Number of hospital days<br>mean (sd) | 0.18 (1.23) | 0.19 (1.14) | 0.16(1.37) | 0.15 (1.15) | 0.23 (1.63) | 0.21(1.63) | 0.19 (1.45) | 0.18 (1.35) | 0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (1.45) | 0.00 (1.35) | 0.00 |
| Number of Emergency Department (ED) visits v3 | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (2.45) | 0.00 (2.33) | 0.00 |
| mean (sd) | 0.20 (0.68) | 0.20 (0.73) | 0.05 (0.57) | 0.06 (0.67) | 0.28 (0.87) | 0.28 (0.94) | 0.15 (0.71) | 0.16 (0.79) | -0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.71) | 0.00 (0.79) | 0.00 |
| Number of Office visits | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.72] | 0.00 (0.75) | 0.00 |
| mean (sd) | 4.33 (3.62) | 4.31 (3.24) | 4.27 (3.24) | 4.27 (3.21) | 4.98 (3.66) | 4.96 (3.55) | 4.54 (3.45) | 4.53 (3.34) | 0.00 |
| median (IQR) | 3.00 [2.00, 6.00] | 3.00 [2.00, 6.00] | 3.00 [2.00, 6.00] | 3.00 [2.00, 6.00] | 4.00 [2.00, 7.00] | 4.00 [2.00, 7.00] | 3.37 (3.45) | 3.37 (3.34) | 0.00 |
| Number of Endocrinologist visits | | | | | | | | | |
| mean (sd) | 0.92 (3.08) | 1.02 (3.47) | 0.67 (2.55) | 0.79 (3.02) | 0.90 (3.58) | 1.02 (4.01) | 0.79 (3.04) | 0.91 (3.47) | -0.04 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (3.04) | 0.00 (3.47) | 0.00 |
| Number of internal medicine/family medicine visits | | | | | | | | | |
| mean (sd) | 5.03 (9.27) | 4.85 (8.11) | 6.75 (7.93) | 6.68 (7.61) | 7.04 (9.32) | 7.19 (10.03) | 6.63 (8.65) | 6.62 (8.64) | 0.00 |
| median [IQR] | 2.00 [0.00, 7.00] | 2.00 [0.00, 7.00] | 5.00 [2.00, 9.00] | 5.00 [2.00, 9.00] | 4.00 [1.00, 9.00] | 4.00 [1.00, 10.00] | 4.23 (8.65) | 4.23 (8.64) | 0.00 |
| Number of Cardiologist visits | | | | | | | | | |
| mean (sd) | 0.96 (2.96) | 0.97 (2.94) | 0.75 (2.40) | 0.71 (2.17) | 1.13 (3.38) | 1.14 (3.20) | 0.92 (2.87) | 0.90 (2.70) | 0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (2.87) | 0.00 (2.70) | 0.00 |
| Number electrocardiograms received v2 | | | | | | | | | |
| mean (sd) | 0.37 (0.87) | 0.37 (0.94) | 0.40 (0.94) | 0.38 (0.90) | 0.45 (0.98) | 0.46 (1.03) | 0.41 (0.95) | 0.41 (0.96) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.95) | 0.00 (0.96) | 0.00 |
| Number of HbA1c tests ordered | | | | | | | | | |
| mean (sd) | 1.27 (0.86) | 1.27 (0.85) | 1.31 (0.86) | 1.30 (0.80) | 1.48 (0.85) | 1.48 (0.81) | 1.37 (0.86) | 1.36 (0.81) | 0.01 |
| median [IQR] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 (0.86) | 1.00 (0.81) | 0.00 |
| Number of glucose tests ordered | 0.37 (0.91) | 0.77 (0.05) | 0.44/4.75 | 0.40 (4.07) | 0.44 (0.04) | 0.43 (0.00) | 0.40 (4.40) | 0.40 (1.02) | 0.00 |
| mean (sd)<br>median (IQR) | 0.00 [0.00, 0.00] | 0.37 (0.96)<br>0.00 (0.00, 0.00) | 0.41 (1.25)<br>0.00 (0.00, 0.00) | 0.40 (1.07)<br>0.00 (0.00, 0.00) | 0.41 (0.94)<br>0.00 (0.00, 0.00) | 0.42 (0.98)<br>0.00 (0.00, 0.00) | 0.40 (1.10)<br>0.00 (1.10) | 0.40 (1.02) | 0.00 |
| Number of lipid tests ordered | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 (1.10) | 0.00 (2.02) | 0.00 |
| mean (sd) | 1.05 (0.95) | 1.05 (0.96) | 1.10(1.39) | 1.09 (1.12) | 1.08 (0.83) | 1.07 (0.83) | 1.09 (1.16) | 1.08 (1.00) | 0.01 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 (1.16) | 1.00 (1.00) | 0.00 |
| Number of creatinine tests ordered | 2.00 (0.00, 2.00) | 2.00 (0.00, 2.00) | 2.00 [0.00, 2.00] | 2.00 [0.00, 2.00] | 2.00 [2.00, 2.00] | 2.00 [2.00, 2.00] | 2.00 [2.20] | 2.00 (2.00) | 2.00 |
| mean (sd) | 0.04 (0.25) | 0.04 (0.28) | 0.03 (0.23) | 0.03 (0.22) | 0.06 (0.30) | 0.06 (0.32) | 0.04 (0.26) | 0.04 (0.27) | 0.00 |
| median (IQR) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.26) | 0.00 (0.27) | 0.00 |
| Number of BUN tests ordered | | | | | | | | · / | |
| mean (sd) | 0.02 (0.19) | 0.02 (0.17) | 0.02 (0.18) | 0.02 (0.16) | 0.04 (0.24) | 0.04 (0.24) | 0.03 (0.21) | 0.03 (0.19) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.21) | 0.00 (0.19) | 0.00 |
| Number of tests for microal burninuma | | | | | | | | | |
| mean (sd) | 0.73 (1.06) | 0.74 (1.11) | 0.73 (1.08) | 0.71 (1.08) | 0.47 (0.68) | 0.47 (0.68) | 0.63 (0.95) | 0.63 (0.96) | 0.00 |
| median (IQR) | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.95) | 0.00 (0.96) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd | | | | | | | | | |
| digit level Copy | | | | | | | | | |
| mean (sd) | 4.05 (5.92) | 4.03 (6.10) | 2.84 (3.82) | 2.79 (3.90) | 6.52 (6.78) | 6.53 (6.84) | 4.36 (5.37) | 4.33 (5.46) | 0.01 |
| median (IQR) | 0.00 [0.00, 7.00] | 0.00 [0.00, 6.00] | 1.00 [0.00, 5.00] | 0.00 [0.00, 5.00] | 5.00 [0.00, 10.00] | 5.00 [0.00, 10.00] | 2.34 (5.37) | 1.84 (5.46) | 0.09 |
| Use of this rider of RC) | ana in nich | 274/40 481 | a page in oils! | a paralo ella | 4 483 (43 49) | a and the obt | 3 702 (40 00) | 2 202 (40 00) | |
| Use of thiszide; n (%)<br>Use of beta blockers; n (%) | 322 (9.7%)<br>1,034 (31.2%) | 334 (10.1%)<br>1,051 (31.7%) | 1,229 (9.9%)<br>4,049 (32.6%) | 1,212 (9.8%)<br>4,037 (32.5%) | 1,152 (12.6%)<br>3,834 (41.8%) | 1,156 (12.6%)<br>3,838 (41.9%) | 2,703 (10.9%)<br>8,917 (35.8%) | 2,702 (10.9%)<br>8,926 (35.9%) | 0.00 |
| Use of calcium channel blockers; n (%) | 706 (21.3%) | 721 (21.7%) | 2,893 (23.3%) | 2,917 (23.5%) | 2,728 (29.8%) | 2,685 (29.3%) | 6,327 (25.4%) | 6,323 (25.4%) | 0.00 |
| | - 30 [22.379] | | 2,223 (23.374) | 2,227 (22374) | 2,.20 (23.014) | 2,525 (25.574) | 2,22. (23.4.4) | 2,222 (23.4.4) | |